# CLINICAL RESEARCH IN INFECTIOUS DISEASES

# STATISTICAL ANALYSIS PLAN FOR

**DMID PROTOCOL: 21-0002 (COHORT 1)** 

### STUDY TITLE:

PHASE I, OPEN-LABEL, RANDOMIZED STUDY OF THE SAFETY AND IMMUNOGENICITY OF A SARS-CoV-2 VARIANT VACCINE (mRNA-1273.351) IN NAÏVE AND PREVIOUSLY VACCINATED ADULTS

NCT04785144

**VERSION 2.0** 

**DATE: 23 MAY 2023** 

THIS COMMUNICATION IS PRIVILEGED AND CONFIDENTIAL

### **STUDY TITLE**

| <b>Protocol Number Code:</b> | DMID Protocol: 21-0002 Cohort 1 |
|---|---|
| <b>Development Phase:</b> | Phase 1 |
| Products: | mRNA-1273/mRNA-1273.351 |
| Form/Route: | Injection |
| Indication Studied: | COVID-19 |
| Sponsor: | Division of Microbiology and Infectious Diseases<br>National Institute of Allergy and Infectious Diseases<br>National Institutes of Health |
| Clinical Trial Initiation Date: | 30MAR2021 |
| <b>Clinical Trial Completion Date:</b> | Ongoing |
| Date of the Analysis Plan: | 23 May 2023 |
| Version Number: | 2.0 |

This study was performed in compliance with Good Clinical Practice.

Information contained in this publication is the property of Division of Microbiology and Infectious Diseases and is confidential. This information may not be disclosed to third parties without written authorization from Division of Microbiology and Infectious Diseases. This report may not be reproduced, stored in a retrieval system or transmitted in any form or by any means - electronic, mechanical, recording or otherwise - without the prior authorization from Division of Microbiology and Infectious Diseases. This document must be returned to Division of Microbiology and Infectious Diseases upon request.

# TABLE OF CONTENTS

# **TABLE OF CONTENTS**

| STUDY TI | ITLE | I |
|---|---|---|
| TABLE OF | F CONTENTS | II |
| LIST OF A | ABBREVIATIONS | V |
| 1. | PREFACE. | 7 |
| 2. | INTRODUCTION | 8 |
| 2.1. | Purpose of the Analyses | 9 |
| 3. | STUDY OBJECTIVES AND ENDPOINTS | 10 |
| 3.1. | Study Objectives and Endpoints | 10 |
| 3.2. | Study Definitions and Derived Variables | 11 |
| 4. | INVESTIGATIONAL PLAN | 12 |
| 4.1. | Overall Study Design and Plan | 12 |
| 4.2. | Discussion of Study Design, Including the Choice of Control Groups | 13 |
| 4.3. | Selection of Study Population | 14 |
| 4.4. | Treatments | 18 |
| 4.4.1. | Treatments Administered. | 18 |
| 4.4.2. | Identity of Investigational Product(s) | 18 |
| 4.4.3. | Method of Assigning Subjects to Treatment Groups (Randomization) | 18 |
| 4.4.4. | Selection of Dose in the Study | 18 |
| 4.4.5. | Prior and Concomitant Therapy | 18 |
| 4.4.6. | Treatment Compliance | 18 |
| 5. | SAMPLE SIZE CONSIDERATIONS | 19 |
| 6. | GENERAL STATISTICAL CONSIDERATIONS | 20 |
| 6.1. | General Principles | 20 |
| 6.2. | Analysis Populations | 20 |
| 6.2.1. | Safety Population | 20 |
| 6.2.2. | Modified Intent-to Treat Population | 20 |
| 6.2.3. | Per Protocol Population | 20 |
| 6.3. | Covariates and Subgroups | 20 |
| 6.4. | Missing Data | 20 |

# **Table of Contents** (continued)

| 6.5. | Interim Analyses and Data Monitoring | 21 |
|---|---|---|
| 6.6. | Multicenter Studies | 21 |
| 6.7. | Multiple Comparisons/Multiplicity | 21 |
| 7. | STUDY SUBJECTS | 22 |
| 7.1. | Disposition of Subjects | 22 |
| 7.2. | Protocol Deviations | 22 |
| 8. | IMMUNOGENICITY EVALUATION | 23 |
| 8.1. | Primary Immunogenicity Analysis | 23 |
| 8.2. | Secondary Immunogenicity Analyses | 23 |
| 8.3. | Exploratory Immunogenicity Analyses | 24 |
| 9. | SAFETY EVALUATION | 25 |
| 9.1. | Demographic and Other Baseline Characteristics | 25 |
| 9.1.1. | Prior and Concurrent Medical Conditions | 25 |
| 9.1.2. | Prior and Concomitant Medications | 25 |
| 9.2. | Measurements of Treatment Compliance | 26 |
| 9.3. | Adverse Events | 26 |
| 9.3.1. | Solicited Events and Symptoms | 26 |
| 9.3.2. | Unsolicited Adverse Events | 26 |
| 9.4. | Deaths, Serious Adverse Events and other Significant Adverse Events | 27 |
| 9.5. | Pregnancies | 27 |
| 9.6. | Clinical Laboratory Evaluations | 27 |
| 9.7. | Vital Signs and Physical Evaluations | 27 |
| 9.8. | Concomitant Medications | 28 |
| 9.9. | Other Safety Measures | 28 |
| 10. | PHARMACOKINETICS | 29 |
| 11. | IMMUNOGENICITY | 30 |
| 12. | OTHER ANALYSES | 31 |
| 13. | REPORTING CONVENTIONS | 32 |
| 14. | TECHNICAL DETAILS | 33 |
| 15. | SUMMARY OF CHANGES IN THE CONDUCT OF THE STUDY OR PLANNED ANALYSES | 34 |
| 16. | REFERENCES | 35 |

| V | <sup>7</sup> ersic | n | 2.0 |
|----|--------------------|---|---------------|
| 23 | May | 2 | $02^{\prime}$ |

| | | 23 May 202 |
|-----------------------|--------------------|------------|
| <b>Table of Conte</b> | nts (continued) | |
| APPENDIX 1. | TABLE MOCK-UPS | 37 |
| APPENDIX 2. | FIGURE MOCK-UPS | 139 |
| APPENDIX 3 | LISTINGS MOCK-LIPS | 191 |

# LIST OF ABBREVIATIONS

| AE | Adverse Event |
|--------|--------------------------------------------------|
| ALT | Alanine Aminotransferase |
| AST | Aspartate Aminotransferase |
| AUC | Area Under the Curve |
| BP | Blood Pressure |
| С | Celsius |
| CI | Confidence Interval |
| CRF | Case Report Form |
| DMID | Division of Microbiology and Infectious Diseases |
| EDC | Electronic Data Capture |
| ECLIA | Electro-chemiluminescence |
| ELISA | Enzyme-linked Immunosorbent Assay |
| F | Fahrenheit |
| FRNT | Focus Reduction Neutralization Test |
| GMT | Geometric Mean Titer |
| GMFR | Geometric Mean Fold Rise |
| ICH | International Council on Harmonisation |
| IRB | Institutional Review Board |
| LLN | Lower Limit of Normal |
| μg | Microgram |
| MedDRA | Medical Dictionary for Regulatory Activities |
| N | Number (typically refers to subjects) |
| NIH | National Institutes of Health |
| PI | Principal Investigator |
| PP | Per Protocol |
| PT | Preferred Term |
| RBC | Red Blood Cell |
| S-2P | S Protein in its Prefusion Conformation |
| SAE | Serious Adverse Event |
| SD | Standard Deviation |
| SDCC | Statistical and Data Coordinating Center |

| SMC | Safety Monitoring Committee |
|-----|-------------------------------|
| SOC | System Organ Class |
| SOP | Standard Operating Procedures |
| ULN | Upper Limit of Normal |
| WBC | White Blood Cell |
| WHO | World Health Organization |

### 1. PREFACE

The Statistical Analysis Plan (SAP) for "Phase 1, Open-Label, Randomized Study of the Safety and Immunogenicity of a SARS-CoV-2 Variant Vaccine (mRNA-1273.351) in Naïve and Previously Vaccinated Adults" (DMID Protocol 21-0002) describes and expands upon the statistical information presented in the protocol for cohort 1 only. A separate SAP will be written for cohort 2. This document describes all planned analyses and provides reasons and justifications for these analyses. It also includes sample tables, listings, and figures planned for the final analyses. Regarding the final analyses and Clinical Study Report (CSR), this SAP follows the International Conference on Harmonisation of Technical Requirements for Registration of Pharmaceuticals for Human Use (ICH) Guidelines, as indicated in Topic E3 (Structure and Content of Clinical Study Reports), and more generally is consistent with Topic E8 (General Considerations for Clinical Trials) and Topic E9 (Statistical Principles for Clinical Trials). The structure and content of the SAP provides sufficient detail to meet the requirements identified by the FDA and ICH, while all work planned and reported for this SAP will follow internationally accepted guidelines published by the American Statistical Association and the Royal Statistical Society for statistical practice.

This document contains a review of the study design, general statistical considerations, comprehensive statistical analysis methods for immunogenicity and safety outcomes, and a list of proposed tables, figures and listings. Within the table, figure, and listing mock-ups (Appendix 1, Appendix 2, and Appendix 3), references to CSR sections are included. The reader of this SAP is encouraged to also review the study protocol for details on conduct of the study and the operational aspects of clinical assessments.

### 2. INTRODUCTION

An outbreak of COVID-19 caused by a novel SARS-CoV-2 began in Wuhan, Hubei Province, China in December 2019, and the disease has since spread globally [10]. The World Health Organization (WHO) declared COVID-19 a pandemic on 11 Mar 2020; however, widespread community transmission was already occurring in many locations. As of 14 Jan 2021, more than 92 million cases and 1.9 million deaths worldwide have been attributed to the COVID-19 pandemic [2,10].

ModernaTX, Inc has developed a vaccine platform based on the principle and observations that cells *in vivo* can take up mRNA, translate it, and then express protein viral antigen(s) on the cell surface. mRNA is highly precise in its translation into proteins that match viral antigens. The delivered mRNA does not enter the cell nucleus or interact with the genome, is nonreplicating, and is expressed transiently. The estimated half-life for mRNA after injection is approximately 8 to 10 hours, before degradation by native RNases in the body, but the duration of effect also depends on the half-life of the expressed protein, which persists in the body for several days. mRNA vaccines have been used to induce immune responses against infectious viral pathogens such as cytomegalovirus, human metapneumovirus, parainfluenza virus type 3, Zika, and influenza.

The mRNA-1273 encodes for the full-length spike (S) protein of SARS-CoV-2, modified to introduce 2 proline residues to stabilize the S protein (S-2P) in a prefusion conformation, derived from the Wuhan-Hu-1 strain [5]. The mRNA-1273 vaccine is currently being evaluated for safety and immunogenicity in a dose-ranging Phase 1 study sponsored by DMID (NCT04283461), for safety and immunogenicity in a Moderna-sponsored Phase 2a study (NCT04405076), and for safety, efficacy, and immunogenicity in a Moderna-sponsored Phase 3 study (NCT04470427). All three of these studies are ongoing and conducted in the US.

The primary efficacy objective of the Phase 3 study was met, with the vaccine efficacy of mRNA-1273 to prevent symptomatic COVID-19 disease observed to be 94.1%. The vaccine was also observed to be efficacious in preventing severe COVID-19. In December 2020 the FDA issued Emergency Use Authorization of mRNA-1273 (Moderna COVID-19 Vaccine) for active immunization to prevent COVID-19 in individuals 18 years of age and older.

Recently, SARS-CoV-2 variants with mutations in the S protein have emerged. A variant first identified in South Africa (B.1.351) is associated with increased transmission, higher viral burden, and possibly increased mortality in infected persons [8]. To date, four vaccines, all based on the Wuhan-sequence of the S protein, have shown reduced activity against the B.1.351 variant. Sera from individuals vaccinated with mRNA-based vaccines had a 6-to-9-fold reduction in neutralizing activity against a B.1.351-matched pseudovirion relative to a Wuhan-matched pseudovirion [9,11]. More recently, pivotal studies testing both viral vector and adjuvanted protein technologies had lower efficacy in regions where B.1.351 was known to be circulating [2]. Hence, the development and testing of vaccines targeting this SARS-CoV-2 variant is urgently needed.

mRNA-1273.351, like mRNA-1273, encodes the prefusion stabilized S protein of SARS-CoV-2. However, the mRNA of mRNA-1273.351 incorporates the key mutations present in the B.1.351 strain of the virus. This phase 1 clinical trial will evaluate the immunological benefit of boosting subjects previously vaccinated with mRNA-1273 (DMID 20-0003) with the B.1.351

strain-specific S protein, as well as the breadth of response induced by vaccinating with mRNA-1273 and mRNA-1273.351 in naïve persons, who have not previously received a SARS-CoV-2 vaccine and are not known to have been previously infected with SARS-CoV-2.

## 2.1. Purpose of the Analyses

These analyses will assess the immunogenicity and safety of monovalent mRNA-1273.351 vaccine at a dose 50  $\mu g$  and bivalent mRNA-1273/mRNA-1273.351 at a dose of 25  $\mu g$  each (50  $\mu g$  total) in subjects opting to terminate DMID 20-0003 early and enrolling in 21-0002 Cohort 1.

# 3. STUDY OBJECTIVES AND ENDPOINTS

# 3.1. Study Objectives and Endpoints

| OBJECTIVES | ENDPOINTS |
|---|---|
| | (OUTCOME MEASURES) |
| To evaluate the safety and reactogenicity of mRNA-1273 and mRNA-1273.351 vaccines, in previously vaccinated individuals. | Frequency and grade of each solicited local and systemic reactogenicity AE during a 7-day follow-up period post each vaccination. |
| | Frequency and grade of any unsolicited AEs during the 28-day follow-up period post each vaccination. |
| | <ul> <li>Frequency of any SAEs, Protocol<br/>Specified AESIs, NOCMCs, and<br/>MAAEs from the first vaccination<br/>through 12 months after the last<br/>vaccination.</li> </ul> |
| Secondary | |
| To assess humoral immunogenicity of mRNA-1273 and mRNA-1273.351 vaccines, in previously vaccinated individuals. | <ul> <li>Response rate, and magnitude of<br/>SARS-CoV-2-specific antibody<br/>binding and neutralization titers in<br/>serum samples as assessed via a<br/>range of assays at all timepoints.</li> </ul> |
| Exploratory | |
| To assess, in at least a subset of samples the innate immune response and B cell response following vaccination. | Magnitude, phenotype, and percentage of innate immune cells and SARS-CoV-2 specific B cells, as measured by flow cytometry, and targeted B cell repertoire analysis at different timepoints post vaccination relative to baseline. |
| To assess, in at least a subset of samples, the SARS-CoV-2 S protein-specific T cell responses. | Magnitude, phenotype, and percentage of cytokine producing S protein-specific T cells, as measured by flow cytometry at different timepoints post vaccination relative to baseline. |

# 3.2. Study Definitions and Derived Variables

For calculations using the baseline value, the value obtained pre-third vaccination (Day 1) will be used. For samples with an AUC of zero at baseline, fold-rise will be calculated by dividing post-vaccination result by the lowest reported value. AUC is calculated using the trapezoidal method applied to a serial dilution curve. 20-0003 Cohort will be used to refer to the 20-0003 cohort that the subjects were originally assigned.

The Williams mean is a variation of the geometric mean using log(1+x) transformation of the data, where x is each data point. The Williams mean is used in cases where 0 is a possible and/or reported value of the data.

### 4. INVESTIGATIONAL PLAN

## 4.1. Overall Study Design and Plan

This is a phase 1, open-label, randomized clinical trial in males and non-pregnant females, 18 years of age and older, who are in good health, have no known history of COVID-19 or SARS-CoV-2 infection, and meet all other eligibility criteria. This clinical trial is designed to assess the safety, reactogenicity and immunogenicity of mRNA-1273.351 manufactured by ModernaTX, Inc, given in vaccination schedules alone, sequentially, or coadministered with mRNA-1273. mRNA-1273.351 is a novel LNP-encapsulated mRNA-based vaccine that encodes for a full-length, prefusion stabilized S protein of the SARS-CoV-2 B.1.351 variant. Enrollment will occur at approximately five domestic clinical research sites.

This study includes two cohorts. Cohort 1 will provide rapid information about the immunogenicity of mRNA-1273.351 in a previously vaccinated group. This cohort can inform near term public health decisions if the variant virus becomes more widespread. Cohort 2 will evaluate different strategies for generation of cross protective immune responses in a naïve population. This cohort will take longer to provide information on the immunogenicity of mRNA-1273.351, but is important to inform future public health strategies. As Cohorts 1 and 2 are in different populations, they can be enrolled in parallel as determined by each site.

Cohort 1 will include subjects 18 years of age and older who received two vaccinations of mRNA-1273 at dosages of 50 mcg, 100 mcg, or 250 mcg in the Phase 1 clinical trial (DMID 20-0003). Those subjects will be offered enrollment into this study approximately 9 to 12 months after they received the second vaccination in DMID 20-0003. At enrollment in this study, their long-term follow-up in DMID 20-0003 will be terminated. Subjects will be randomized, within each of the DMID 20-0003 cohorts (age and dosage groups – 50 mcg, 100 mcg, and 250 mcg), 1:1 (as outlined in Table 7) to either:

- Arm 1A, vaccination with a 50-mcg dose of the mRNA-1273.351 variant, or
- Arm 1B, vaccination with a combination vaccination that includes 25 mcg of mRNA-1273 and 25 mcg of mRNA-1273.351.

The anticipated sample size to be drawn from the DMID 20-0003 study population is approximately 45 subjects 18 through 55 years of age and approximately 20 subjects 56 years of age and older.

Subjects in Cohort 1 will receive a single intramuscular (IM) injection of the designated vaccine and will be followed through 12 months after vaccination. Follow-up visits will occur on Days 8, 15, and 29, as well as 3, 6, and 12 months after the vaccination.

Cohort 2 will include approximately 150 participants 18 through 55 years of age who have not received a COVID-19 vaccine, have no known history of COVID-19 or SARS-CoV-2 infection, and do not have underlying conditions that are associated with an increased risk of severe illness from SARS-CoV-2 infection. Enrollment may close before the full 150 participants based on estimates on the timing of immunogenicity results and the need to inform public health decisions. They will be randomly assigned to one of 8 treatment arms and will receive 2 or 3 IM injections of the vaccine and followed through 12 months after the last vaccination. Follow-up

visits will occur 7, 14, and 28 days after each vaccination, as well as 3, 6, and 12 months post the last vaccination.

For both Cohorts 1 and 2, reactogenicity will be assessed and blood will be drawn for immunogenicity assays.

After the IND is in effect, IRB review and approval, and site activation, the participating sites will begin recruitment outreach efforts, which can include fliers, letters, telephone calls, etc. Information regarding this trial may be provided to potential subjects who have previously participated in other vaccine trials conducted at the participating site. Other forms and/or mechanisms of recruitment may also be used. The IRB will approve the recruitment process and all materials prior to use. Screening can occur up to 42 days prior to the first dose.

## 4.2. Discussion of Study Design, Including the Choice of Control Groups

This phase 1 clinical trial is designed as an open-label study, without administration of a placebo formulation. An open-label study will facilitate the need for rapid review and dissemination of study data for public health reasons.

In the Phase 1 clinical trial, DMID 20-0003, mRNA-1273, administered as two injections 28 days apart, was investigated at dosages of 25, 50, 100 and 250 mcg in subjects 18 through 55 years of age, and at dosages of 25, 50, and 100 mcg in older cohorts (56-70 years of age and >71 years of age) [1,7]. The 100-mcg dose induced higher antibody titers than the 25-mcg dose, whereas the 250-mcg dose did not lead to significant increases, which supported evaluation of the 100-mcg dose in Phase 2 and Phase 3 trials. Subsequent to the start of the Phase 3 trial, an interim analysis of immunogenicity data from the Phase 2 demonstrated that the 50 and 100-mcg doses in a two-dose series are similarly immunogenic [4] and warrants further evaluation. The primary efficacy analysis from the Phase 3 trial evaluating a two-dose schedule of a 100-mcg mRNA-1273 vaccine led to the issuance of the EUA and initiation of a vaccination campaign in the United States.

The Phase 2 trial of mRNA-1273 evaluated doses of 50 mcg and 100 mcg, administered as a two-vaccination series, in 600 adults ≥18 years of age. The safety profile of both formulations was acceptable [4]. Anti-SARS-CoV-2 S binding and neutralizing antibodies were induced by both dose levels of mRNA-1273 within 28 days after the first vaccination, and rose substantially to peak titers by 14 days after the second vaccination, exceeding levels of convalescent sera from COVID-19 patients. The antibodies remained elevated through the last timepoint assessed at 57 days. Neutralizing responses met criteria for seroconversion within 28 days after the first vaccination in the majority of participants, with rates of 100% observed at 14 and 28 days after the second vaccination. Binding and neutralizing antibody responses were generally comparable in participants who received the 100 mcg mRNA-1273 and the 50 mcg dose at all time points and across the age groups of ≥18 to <55 years and ≥55 years. These findings support the evaluation of mRNA-1273 and mRNA-1273.351 at total dosages of 50 or 100 mcg per vaccination.

# 4.3. Selection of Study Population

Two cohorts will be enrolled. For Cohort 1, approximately 60 males and non-pregnant female subjects 18 years of age and older, who are in good health and received two vaccinations of mRNA-1273 at dosages of 50 mcg, 100 mcg or 250 mcg in DMID 20-0003 will be invited to participate in this study.

For Cohort 2, approximately 150 males and non-pregnant females, 18 through 55 years of age, who have never been vaccinated against SARS-CoV-2 or are not known to have been infected with SARS-CoV-2, and are at low risk for severe disease, in good health, and meet all eligibility criteria will be enrolled. The target population should reflect the community at large.

The estimated time from initiation of enrollment to complete enrollment in this clinical trial is approximately 4 weeks (though could take up to 8 weeks). Information regarding this trial may be provided to potential subjects who have previously participated in other vaccine trials conducted at the participating site. Other forms and/or mechanisms of recruitment may also be used. The IRB will approve the recruitment process and all materials prior to use. Screening can occur up to 42 days prior to the first vaccination.

Subject Inclusion and Exclusion Criteria must be confirmed by a study clinician, licensed to make medical diagnoses and listed on the Form FDA 1572 as the participating site principal investigator (PI) or appropriate sub-investigator. No exemptions are granted on Subject Inclusion or Exclusion Criteria in DMID-sponsored studies.

#### **Inclusion Criteria**

A subject must meet all the following criteria to be eligible to participate in this substudy:

- 1. Provides written informed consent prior to initiation of any study procedures.
- 2. Be able to understand and agrees to comply with planned study procedures and be available for all study visits.
- 3. Agrees to the collection of venous blood per protocol.
- 4. Cohort 1: previously received 2 doses of mRNA-1273 IM as part of DMID 20-0003.
- 5. Cohort 1: Male or non-pregnant female, ≥18 years of age at time of enrollment.Cohort 2: Male or non-pregnant female, 18 through 55 years of age at time of enrollment.
- 6. Women of childbearing potential<sup>1</sup> must agree to practice abstinence or use at least one acceptable primary form of contraception.<sup>2,3</sup>
  - Note: These criteria are applicable to females in a heterosexual relationship and child-bearing potential (i.e., the criteria do not apply to subjects in a same sex relationship).
  - Not of childbearing potential post-menopausal females (defined as having a history of amenorrhea for at least one year) or a documented status as being surgically sterile (hysterectomy, bilateral oophorectomy, tubal ligation/salpingectomy, or Essure® placement).

• <sup>2</sup>Acceptable forms of primary contraception include monogamous relationship with a vasectomized partner who has been vasectomized for 180 days or more prior to the subject's first vaccination, intrauterine devices, birth control pills, and injectable/implantable/insertable hormonal birth control products.

<sup>3</sup>Must use at least one acceptable primary form of contraception for at least 30 days prior to the first vaccination and at least one acceptable primary form of contraception for 60 days after the last vaccination.

### 7. In good health.<sup>4</sup>

- <sup>4</sup>As determined by medical history and physical examination to evaluate acute or ongoing chronic medical diagnoses/conditions that have been present for at least 90 days, which would affect the assessment of safety of subjects. Chronic medical diagnoses/conditions should be stable for the last 60 days (no hospitalizations, ER, or urgent care for condition or need for supplemental oxygen). This includes no change in chronic prescription medication, dose, or frequency as a result of deterioration of the chronic medical diagnosis/condition in the 60 days before enrollment. Any prescription change that is due to change of health care provider, insurance company, etc., or done for financial reasons, and in the same class of medication, will not be considered a deviation of this inclusion criterion. Any change in prescription medication due to improvement of a disease outcome or for dose optimization, as determined by the participating site PI or appropriate sub-investigator, will not be considered a deviation of this inclusion criterion. Subjects may be on chronic or as needed (prn) medications if, in the opinion of the participating site PI or appropriate sub-investigator, they pose no additional risk to subject safety or assessment of reactogenicity and immunogenicity, and do not indicate a worsening of medical diagnosis/condition. Similarly, medication changes subsequent to enrollment and study vaccination are acceptable provided the change was not precipitated by deterioration in the chronic medical condition, and there is no anticipated additional risk to the subject or interference with the evaluation of responses to study vaccination.
- 8. Oral temperature is less than 100.0°F (37.8°C).
- 9. Must agree to have samples stored for secondary research.
- 10. Agrees to adhere to Lifestyle Considerations (defined in Section 5.4 of the Protocol) throughout study duration.
- 11. Must agree to refrain from donating blood or plasma during the study (outside of this study).

#### **Exclusion Criteria**

A subject who meets any of the following criteria will be excluded from participation in this study:

- 1. Positive pregnancy test prior to each vaccine administration.
- 2. BMI  $>40.0 \text{ kg/m}^2$ .

- 3. Female subject who is breastfeeding.
- 4. Has any medical disease or condition that, in the opinion of the participating site PI or appropriate sub-investigator, precludes study participation.<sup>5</sup>
  - <sup>5</sup>Including acute, subacute, intermittent or chronic medical disease or condition that would place the subject at an unacceptable risk of injury, render the subject unable to meet the requirements of the protocol, or may interfere with the evaluation of responses or the subject's successful completion of this trial.
- 5. Presence of self-reported or medically documented significant medical or psychiatric condition(s).<sup>6</sup>

<sup>6</sup>Significant medical or psychiatric conditions include but are not limited to:

- Respiratory disease (e.g., chronic obstructive pulmonary disease [COPD], asthma) requiring daily medications currently or any treatment of respiratory disease exacerbations (e.g., asthma exacerbation) in the last 5 years. Asthma medications: inhaled, oral, or intravenous (IV) corticosteroids, leukotriene modifiers, long and short acting beta agonists, theophylline, ipratropium, biologics.
- Significant cardiovascular disease (e.g., congestive heart failure, cardiomyopathy, ischemic heart disease), history of myocarditis or pericarditis as an adult, myocardial infarction (MI) within past 6 months, coronary artery bypass surgery or stent placement, or uncontrolled cardiac arrhythmia.
- Neurological or neurodevelopmental conditions (e.g., history of migraines in the past 5 years, epilepsy, stroke, seizures in the last 3 years, encephalopathy, focal neurologic deficits, Guillain-Barré syndrome, encephalomyelitis, transverse myelitis, stroke or transient ischemic attack, multiple sclerosis, Parkinson's disease, amyotrophic lateral sclerosis, Creutzfeldt-Jakob disease, or Alzheimer's disease).
- Ongoing malignancy or recent diagnosis of malignancy in the last five years excluding basal cell and squamous cell carcinoma of the skin, which are allowed.
- An autoimmune disease, including hypothyroidism without a defined non-autoimmune cause, localized or history of psoriasis.
- An immunodeficiency of any cause.
- Chronic kidney disease, estimated glomerular filtration rate (eGFR) <60 mL/min/1.73m<sup>2</sup>.
- Type 2 diabetes mellitus, not including prediabetes.
- 6. Has an acute illness<sup>7</sup>, as determined by the participating site PI or appropriate sub-investigator, with or without fever [oral temperature ≥38.0°C (100.4°F)] within 72 hours prior to each vaccination.

<sup>7</sup>An acute illness which is nearly resolved with only minor residual symptoms remaining is allowable if, in the opinion of the participating site PI or appropriate sub-investigator, the residual symptoms will not interfere with the ability to assess safety parameters as required by the protocol.

- 7. Has participated in another investigational study involving any investigational product<sup>8</sup> within 5 half-lives before the first vaccine administration.
  - <sup>8</sup>study drug, biologic or device
- 8. Currently enrolled in or plans to participate in another clinical trial with an investigational agent<sup>9</sup> that will be received during the study-reporting period.<sup>10</sup>
  - <sup>9</sup>Including licensed or unlicensed vaccine, drug, biologic, device, blood product, or medication.
  - <sup>10</sup>Up to 15 months after the first vaccination.
- 9. Has a history of hypersensitivity or severe allergic reaction (e.g., anaphylaxis, generalized urticaria, angioedema, other significant reaction) to drugs or any previous licensed or unlicensed vaccines or to polyethylene glycol (PEG) or a PEG-containing product.
- 10. Chronic use (more than 14 continuous days) of any medications that may be associated with impaired immune responsiveness.<sup>11</sup>
  - <sup>11</sup>Including, but not limited to, systemic corticosteroids exceeding 10 mg/day of prednisone equivalent, allergy injections, immunoglobulin, interferon, immunomodulators, cytotoxic drugs, or other similar or toxic drugs during the preceding 6-month period prior to vaccine administration (Day 1). The use of low dose topical, ophthalmic, inhaled and intranasal steroid preparations will be permitted.
- 11. Anticipating the need for immunosuppressive treatment within the next 6 months.
- 12. Received immunoglobulins and/or any blood or blood products within the 4 months before the first vaccine administration or at any time during the study.
- 13. Has any blood dyscrasias or significant disorder of coagulation.
- 14. Received or plans to receive a licensed, live vaccine within 4 weeks before or after each vaccination.
- 15. Received or plans to receive a licensed, inactivated vaccine within 2 weeks before or after each vaccination.
- 16. Receipt of any other SARS-CoV-2 vaccine or any experimental coronavirus vaccine at any time prior to or during the study, except Cohort 1 subjects who received mRNA-1273 in DMID 20-0003.
- 17. Close contact of anyone known to have SARS-CoV-2 infection within 14 days prior to vaccine administration.
- 18. History of COVID-19 diagnosis, positive SARS-CoV-2 PCR test, or, for Cohort 2 only, a known positive SARS-CoV-2 serologic test.
- 19. On current treatment with investigational agents for prophylaxis of COVID-19.

### 4.4. Treatments

#### 4.4.1. Treatments Administered

A booster dose of monovalent mRNA-1273.351 will be administered at 50mcg or a booster dose of bivalent mRNA-1273.351/ mRNA-1273 will be administered at 50mcg (25mcg of each).

#### 4.4.2. Identity of Investigational Product(s)

# <u>Product: There are two clinical presentations of mRNA-1273 — mRNA-1273 and mRNA-1273.351</u>

mRNA-1273 (0.2 mg/mL) is an LNP dispersion containing an mRNA that encodes for the pre fusion stabilized S protein of the Wuhan-Hu-1 strain of SARS-CoV-2. mRNA-1273 consists of an mRNA Drug Substance that is manufactured into LNPs composed of the proprietary ionizable lipid, SM-102, and 3 commercially available lipids, cholesterol, 1,2-distearoyl-sn-glycero-3-phosphocholine (DSPC), and PEG2000 DMG.

mRNA-1273.351 (0.5 mg/mL) is formulated in the same way but contains mRNA that encodes for the prefusion stabilized S protein of the B.1.351 variant SARS-CoV-2 strain.

### 4.4.3. Method of Assigning Subjects to Treatment Groups (Randomization)

Subjects in Cohort 1 will be stratified by DMID 20-0003 cohort (age and dosage group) and randomized 1:1 to Arm 1A or 1B. Randomization will be done in the SDCC's Advantage eClinical<sup>SM</sup> (Electronic Data Capture System).

#### 4.4.4. Selection of Dose in the Study

See Section 4.2 for a discussion of dose selection for this study.

### 4.4.5. Prior and Concomitant Therapy

Concomitant medications include only prescription medications and vaccines received outside of the study taken by the subject at the time of enrollment through 28 days after the last vaccination. At each study visit, if there are new SAEs, Protocol Specified AESIs, MAAEs, or NOCMCs, concomitant medications should be recorded on the appropriate DCF.

#### 4.4.6. Treatment Compliance

All subjects are to receive 1 additional dose of study product administered in the clinic.

### 5. SAMPLE SIZE CONSIDERATIONS

Rare AEs are not demonstrable in a clinical study of this size; however, the probabilities of observing one or more AEs given various true event rates are presented in Table 3. With the assumption that all enrolled subjects will likely complete immunizations and safety visits in this relatively short duration study, the following statistical considerations apply. With approximately 30 subjects in each arm (Arms 1A and 1B), the chance of observing at least one AE of probability 10% or more is approximately 96%. Therefore, if no AEs of a given type occur in a Cohort 1 Arm, we can be relatively confident that they will occur in fewer than 10% of people once the vaccine is implemented. With approximately 60 subjects across these two Arms (1A and 1B), the chance of observing at least one AE of probability 5% or more is at least 95%. Therefore, if no AEs of a given type occur across Cohort 1, we can be very confident that any combination independent event will occur in fewer than 5% of people once the vaccine is implemented as a boost.

### 6. GENERAL STATISTICAL CONSIDERATIONS

## **6.1.** General Principles

In general continuous variables will be summarized using the following descriptive statistics: n (non-missing sample size), mean, standard deviation, median, maximum, and minimum. The frequency and percentages (based on the non-missing sample size) of observed levels will be reported for all categorical measures. In general, all data will be listed, sorted by site, treatment, and subject, and when appropriate by visit number within subject. All summary tables will be structured with a column for each treatment and will be annotated with the total population size relevant to that table/cohort, including any missing observations.

### **6.2.** Analysis Populations

#### **6.2.1.** Safety Population

The Safety Analysis population includes all subjects who received the third vaccination.

### **6.2.2. Modified Intent-to Treat Population**

The modified intent-to-treat (mITT) population includes all subjects who received the third vaccination and contributed both pre- and at least one post-third vaccination venous blood samples for immunogenicity testing for which valid results were reported.

### **6.2.3.** Per Protocol Population

In the final analysis, protocol deviations will be reviewed to determine which protocol deviations may affect the analysis. The per protocol (PP) population will then be defined – and this includes all subjects in the mITT subset with the following exclusions:

- Data from all available visits for subjects found to be ineligible at baseline.
- Data from all visits subsequent for the protocol deviations that are considered to affect the science.
- Data from any visit that occurs substantially out of window.

# 6.3. Covariates and Subgroups

The protocol does not define any formal subgroup analyses, and the study is not adequately powered to perform subgroup analyses.

# 6.4. Missing Data

There are no imputations planned for missing data.

For immunogenicity assays, any values below zero may be imputed as zero (or slightly above zero) for analysis purposes. Any such imputations will be noted in the corresponding analysis.

### 6.5. Interim Analyses and Data Monitoring

Cumulative safety information, study status, and primary endpoint results may be published, presented at a public forum, or presented as summaries aggregated by study arm at the discretion of the sponsor while the study is ongoing. Any ad-hoc analyses, jointly developed by the SDCC and/or the Vaccine Research Center (VRC), other participating laboratories and ModernaTX, Inc., will be executed by the SDCC as needed. None of the interim analyses will include any formal statistical hypothesis testing; therefore, p value adjustment will not be made to any analyses.

The SMC will not need to meet (unless halting rules are met), and materials will be provided electronically. Documentation of review and any concerns noted will be solicited electronically. The SMC will review cumulative AE data after all subjects in Cohort 1 have been dosed and completed Day 8.

• Interim data review of immunogenicity may be performed to inform public health decisions.

Statistical analyses of secondary immunogenicity endpoints, by vaccine schedule group, may be performed when subjects have completed key immunogenicity visits. Immunogenicity reviews may be shared with the SMC, as determined by DMID.

Data may be disseminated to public health officials and partners as needed and included in publications and presentations to inform the global scientific community.

Interim analyses of safety, reactogenicity, and immunologic response data may be done, as needed.

#### 6.6. Multicenter Studies

Data will be pooled across all clinical sites. Center effects are not anticipated because the sites are using standardized procedures for vaccination and assessment of solicited and unsolicited adverse events, and the study relies on central laboratories for the assessment of immunogenicity endpoints.

# 6.7. Multiple Comparisons/Multiplicity

There are no adjustments planned for multiple comparisons.

### 7. STUDY SUBJECTS

## 7.1. Disposition of Subjects

Table 8 will present a summary of the reasons that subjects were screened but not enrolled.

The composition of analysis populations, including reasons for subject exclusion, by treatment arm, is presented in Table 7.

The disposition of subjects in the study will be tabulated by treatment group (Table 6). The table shows the total number of subjects screened, enrolled, receiving first vaccination, discontinuing treatment, receiving second vaccination, study ongoing or terminated from study follow-up and the number completing the study.

A flowchart showing the disposition of study subjects, adapted from the Consort Statement [5] will be included (Figure 1). This figure will present the number of subjects screened, enrolled, lost to follow-up, and analyzed, by treatment group.

A listing of subjects who discontinued dosing or terminated from study follow-up and the reason will be included in Listing 2.

### 7.2. Protocol Deviations

A summary of subject-specific protocol deviations will be presented by the reason for the deviation, the deviation category, and treatment group for all subjects (Table 4) as well as similar summaries for major subject-specific protocol deviations (Table 5). All subject-specific protocol deviations and non-subject specific protocol deviations will be included in Appendix 3 as data listings (Listing 3 and Listing 4, respectively).

### 8. IMMUNOGENICITY EVALUATION

## 8.1. Primary Immunogenicity Analysis

See Section 9 for safety analyses which are the primary endpoints of this study.

# 8.2. Secondary Immunogenicity Analyses

Summaries and analysis of immunogenicity data will be presented for the mITT population. If there are protocol deviations which may affect the analysis, a per-protocol (PP) analysis may also be performed.

Seroconversion is defined as a 4-fold increase in result over baseline.

Binding will be measured three types of ECLIA assays. The first is a single-plex (ECLIA) that produces arbitrary units/mL that is a validated assay and can be converted to binding antibody units for Wa-1 S-2P binding. The second is a 4-plex (ECLIAv2) assay that is also validated and produces arbitrary units/mL to measure variant specific binding. The final assay is a 10-plex (ECLIAv2) that is a fit for purpose assay that produces area under the curve and is used to assess binding for variants of concern.

Seroconversion rates, geometric mean fold rise (GMFR) and geometric mean (GM) or Williams mean of arbitrary units per mL (AU/mL), binding antibody unit/mL (BAU, only for Wa-1 [S2-P] variant), and AUC for SARS-CoV-2 will be calculated at Study Days 1 (GM only), 15, 29, 91, 181 and 366 post third vaccination by treatment group and will include both tabular and graphical summaries. Seroconversion rates, GMFR and GM will be presented with their corresponding 95% confidence interval (CI) estimates (using Student's t-distribution for GM and GMFR and the Clopper-Pearson binomial method for seroconversion) at each post vaccination timepoint and overall peak GM. Summaries of GM are included starting with Table 12 and ending with Table 33 and summaries of GMFR and seroconversion are included starting with Table 78 and ending with Table 99. Graphical displays will include reverse cumulative distribution plots (starting with Figure 2 and ending with Figure 23), individual values over time (starting with Figure 24 and ending with Figure 45), geometric mean over time (starting with Figure 46 and ending with Figure 67), and distribution of responses over time (starting with Figure 108 and ending with Figure 129).

Neutralization assays using SARS-CoV-2 pseudovirus neutralization assay (PsVNA) and focus reduction neutralization test (FRNT) will be run using serial dilutions against available variants (e.g., Beta, Delta). ID<sub>50</sub> and ID<sub>80</sub> will be calculated using a 5-parameter logistic regression model. ID<sub>50</sub> and ID<sub>80</sub> will be summarized by group using the geometric mean and 95% CI (using Student's t-distribution) at each post vaccination timepoint and overall peak GM (starting with Table 34 and ending with Table 73). Summaries of GMFR and seroconversion are included starting with Table 100 and ending with Table 139. The ratio of the result for each variant divided by the result of the D614G variant will be calculated and summarized as the geometric mean ratio (GMR) (Table 140, Table 141, Table 142, Table 143, Table 144, Table 145, Table 146, Table 147). Graphical displays for PsVNA and FRNT will include geometric mean over time (starting with Figure 68 and ending with Figure 107) and distributions of responses over time (starting with Figure 130 and ending with Figure 169).

Correlations between all assays will be displayed in a heatmap (Figure 170, Figure 171, Figure 173, Figure 174, Figure 175, Figure 176, Figure 177, Figure 178, Figure 179).

Individual immunogenicity responses are shown in Listing 8.

Any additional variants of concern not listed in the appendices that are of scientific interest may be analyzed in an analogous manner in the final report.

### 8.3. Exploratory Immunogenicity Analyses

The magnitude, phenotype and percentage of cytokine expressing S protein specific T cells will be summarized at each timepoint by Treatment Group. Mean percentages of CD4 and CD8 T cells expressing cytokines and proportions of responders with 95% CI along with median, minimum, and maximum will be presented by peptide pool stimulation (Table 74, Table 75, Table 76, Table 77). Distributions of T cell percentages will be graphically displayed (starting with Figure 180 and ending with Figure 299).

Individual T-cell responses are shown in Listing 9.

### 9. SAFETY EVALUATION

Summaries and analysis of safety data will be presented for the Safety Analysis Population.

Solicited AEs will be summarized by severity for each day post third vaccination (Study Days 1-8) and as the maximum severity over all 8 days. Additionally, solicited AEs will be analyzed by taking the most severe response over the follow-up period and using standard techniques, such as exact confidence intervals (CI), to summarize the proportion of subjects reporting each symptom, any local symptom, and any systemic symptom.

Unsolicited non-serious AEs will be collected from the time of the third vaccination through 28 days after the third vaccination. Unsolicited AEs will be coded by MedDRA for preferred term and system organ class (SOC). SAEs, Protocol Specified AESIs, MAAEs, and NOCMCs will be collected from the time of third vaccination through 12 months after the third vaccination. The numbers of SAEs and MAAEs will be reported by detailed listings showing the event description, MedDRA preferred term and SOC, relevant dates (vaccinations and AEs), severity, relatedness, and outcome for each event. Non-serious unsolicited AEs will be summarized as number and percentage of subjects reporting at least one event in each MedDRA preferred term and SOC, cross tabulated by severity and relationship to study product. Additionally, the proportion of subjects and exact 95% CIs of AEs in aggregate and by MedDRA categories will be computed.

# 9.1. Demographic and Other Baseline Characteristics

Summaries of age, sex, ethnicity, time since second dose, and race will be presented by Treatment Group (Table 9 and Table 10). Ethnicity is categorized as Hispanic or Latino, or not Hispanic and not Latino. In accordance with NIH reporting policy, subjects may self-designate as belonging to more than one race or may refuse to identify a race, the latter reflected in the CRF as "No" to each racial option.

Individual subject listings will be presented for all demographics (Listing 6).

#### 9.1.1. Prior and Concurrent Medical Conditions

All current illnesses and past pre-existing medical conditions will be MedDRA® coded using MedDRA dictionary version 23.0r higher.

Summaries of subjects' pre-existing medical conditions will be presented by Treatment Group (Table 11).

Individual subject listings will be presented for all medical conditions (Listing 7).

#### 9.1.2. Prior and Concomitant Medications

Summaries of medications that were started prior to dosing and continuing at the time of dosing will be presented by WHO Drug Terms 2 and 3 and Treatment Group (Table 165).

Individual subject listings will be presented for all concomitant medications (Listing 15).

### 9.2. Measurements of Treatment Compliance

All subjects are to receive 1 additional dose of study product administered in the clinic. The number of subjects receiving experimental (third) dose will be summarized as part of the subject disposition table (Table 6).

### 9.3. Adverse Events

When calculating the incidence of adverse events (i.e., on a per subject basis), each subject will only be counted once and any repetitions of adverse events within a subject will be ignored; the denominator will be the total population size. All adverse events reported will be included in the summaries and analyses.

### 9.3.1. Solicited Events and Symptoms

Systemic solicited adverse events were collected pre-third vaccination, and systemic and local solicited adverse events were collected 30 minutes post-third vaccination and then daily for 7 days after the third vaccination and graded on a scale of 0 (absent), 1 (mild), 2 (moderate) and 3 (severe). Systemic events include: fatigue, headache, myalgia, arthralgia, nausea, chills and fever. Local events include: pain at injection site, erythema, and induration.

The proportion of subjects reporting at least one solicited adverse event will be summarized for each solicited adverse event, any systemic symptom, any local symptom, and any symptoms. The 95% CI calculated using Clopper-Pearson methodology from a binomial distribution (SAS Proc Freq with a binomial option) will be presented (Table 149).

For each systemic and local event, any systemic event, any local event, and any solicited event, the maximum severity over 7 days after the third vaccination will be summarized for the Safety population. The number and percentage of subjects reporting each event will be summarized by the maximum severity and treatment group (Table 150). For each event the denominator is the number of subjects with non-missing data for the specific event.

The number of subjects reporting a solicited adverse event will be summarized for each day post-third vaccination both in a summary table (Table 151 and Table 152) and graphically in a bar chart (Figure 300 and Figure 301).

The mean, standard deviation, median, minimum and maximum duration of solicited events will be summarized (Table 153).

Day of solicited symptom onset will be summarized graphically (Figure 302 and Figure 303).

Solicited adverse events by subject will be presented in listings (Listing 10 and Listing 11) and graphically (starting with Figure 304 and ending with Figure 315).

### 9.3.2. Unsolicited Adverse Events

The proportion of subjects reporting at least one unsolicited adverse event will be summarized by MedDRA system organ class and preferred term for the third vaccination. Denominators for percentages are the number of subjects who received the vaccination.

Adverse events by subject will be presented in Listing 12.

The following summaries for unsolicited adverse events will be presented by MedDRA system organ class, preferred term, and Treatment Group:

- Subject incidence and total frequency of adverse events (Table 156);
- Summary of severity and relationship to study product (Table 154 and Table 155);
- Listing of Non-Serious, Unsolicited, Moderate or Severe Adverse Events (Table 158);
- Bar chart of frequency of adverse events by severity and MedDRA system organ class (Figure 316);
- Bar chart of incidence of adverse events by severity and MedDRA system organ class (Figure 317).

# 9.4. Deaths, Serious Adverse Events and other Significant Adverse Events

The following listings will be presented including Subject ID, Age (years) Adverse Event Description, Adverse Event Onset Date/End Date, Last Dose Received/Days Post Dose, Reason Reported as an SAE, Relationship to Treatment, Alternate Etiology if not Related, Outcome, and Duration of Event (days):

- Deaths and Serious Adverse Events (Table 157);
- New Onset Chronic Medical Conditions and Medically Attended Adverse Events (Table 159).

# 9.5. Pregnancies

For any subjects in the Safety population who became pregnant during the study, every attempt will be made to follow these subjects to completion of pregnancy to document the outcome, including information regarding any complications with pregnancy and/or delivery. A listing of pregnancies and outcomes will be presented (Listing 16, Listing 17, Listing 18, Listing 19, and Listing 20).

# 9.6. Clinical Laboratory Evaluations

Not applicable.

# 9.7. Vital Signs and Physical Evaluations

Vital sign measurements included systolic blood pressure, diastolic blood pressure, pulse, and oral temperature. Vital signs were assessed at Study Day 1, Study Day 15, Study Day 29, Study Day 91, Study Day 118, and Study Day 366. Vital signs will be tabulated by visit and Treatment Group in Table 160, Table 161, Table 162, Table 163, Table 164 (Listing 13).

Physical Examinations were only to be performed if clinically indicated at Study Day 1, Study Day 15, Study Day 29, Study Day 91, Study Day 118, and Study Day 366. The following body systems will be assessed: Abdomen, Cardiovascular/heart, Extremities, General Appearance, Hepatobiliary/spleen, HEENT, Lymph nodes, Musculoskeletal, Neck, Neurological, Pulmonary/Chest, and Skin (Listing 14).

## 9.8. Concomitant Medications

Concomitant medications will be coded to the Anatomical Therapeutic Classification using the WHO Drug Dictionary. The use of prior and concomitant medications taken during the study will be recorded on the CRFs. A by-subject listing of concomitant medication use will be presented (Listing 15). The use of concomitant medications during the study will be summarized by ATC1, ATC2 code and Treatment Group for the Safety population (Table 165).

## 9.9. Other Safety Measures

Not applicable.

# 10. PHARMACOKINETICS

Not applicable.

# 11. IMMUNOGENICITY

See Section 8.

# 12. OTHER ANALYSES

Not Applicable.

## 13. REPORTING CONVENTIONS

The mean, standard deviation, and other statistics will be reported to 1 decimal place greater than the original data. The minimum and maximum will use the same number of decimal places as the original data. Proportions will be presented as 2 decimal places; values greater than zero but <0.01 will be presented as "<0.01". Percentages will be reported to the nearest whole number; values greater than zero but < 1% will be presented as "<1"; values greater than 99% but less than 100% will be reported as >99%. Estimated parameters, not on the same scale as raw observations (e.g., regression coefficients) will be reported to 3 significant figures.

# 14. TECHNICAL DETAILS

SAS version 9.4 and R 3.6.2 or above will be used to generate all tables, figures and listings.

# 15. SUMMARY OF CHANGES IN THE CONDUCT OF THE STUDY OR PLANNED ANALYSES

Not Applicable.

## 16. REFERENCES

- Anderson, E. J., Rouphael, N. G., Widge, A. T., Jackson, L. A., Roberts, P. C., Makhene, M., Chappell, J. D., Denison, M. R., Stevens, L. J., Pruijssers, A. J., McDermott, A. B., Flach, B., Lin, B. C., Doria-Rose, N. A., O'Dell, S., Schmidt, S. D., Corbett, K. S., Swanson, P. A., 2nd, Padilla, M., Neuzil, K. M., ... mRNA-1273 Study Group (2020). Safety and Immunogenicity of SARS-CoV-2 mRNA-1273 Vaccine in Older Adults. The New England Journal of Medicine, 383(25), 2427–2438. https://doi.org/10.1056/NEJMoa2028436.
- 2. Callaway, E. & Mallapaty, S. (2021). Novavax offers first evidence that COVID vaccines protect people against variants. Nature, 10.1038/d41586-021-00268-9. Advance online publication. https://doi.org/10.1038/d41586-021-00268-9.
- 3. Center for Systems Science and Engineering (CCSE) at Johns Hopkins University (JHU). COVID-19 Dashboard. 2020. https://coronavirus.jhu.edu/map.html. Accessed 04 Feb 2021.
- 4. Chu L., McPhee R., Huang W., Bennett H., Pajon R., Nestorova B., Leav B., ... mRNA-1273 Study Group (2021). A Preliminary Report of a Randomized Controlled Phase 2 Trial of the Safety and Immunogenicity of mRNA-1273 SARS-CoV-2 Vaccine. Vaccine. Advance online publication. https://doi.org/10.1016/j.vaccine.2021.02.007.
- 5. Corbett, K. S., Edwards, D. K., Leist, S. R., Abiona, O. M., Boyoglu-Barnum, S., Gillespie, R. A., Himansu, S., Schäfer, A., Ziwawo, C. T., DiPiazza, A. T., Dinnon, K. H., Elbashir, S. M., Shaw, C. A., Woods, A., Fritch, E. J., Martinez, D. R., Bock, K. W., Minai, M., Nagata, B. M., Hutchinson, G. B., ... Graham, B. S. (2020). SARS-CoV-2 mRNA vaccine design enabled by prototype pathogen preparedness. Nature, 586(7830), 567–571. https://doi.org/10.1038/s41586-020-2622-0
- 6. Drummond R. CONSORT Revised: Improving the Reporting of Randomized Clinical Trials. JAMA. 2001; 285(15): 2006-2007.
- Jackson, L. A., Anderson, E. J., Rouphael, N. G., Roberts, P. C., Makhene, M., Coler, R. N., McCullough, M. P., Chappell, J. D., Denison, M. R., Stevens, L. J., Pruijssers, A. J., McDermott, A., Flach, B., Doria-Rose, N. A., Corbett, K. S., Morabito, K. M., O'Dell, S., Schmidt, S. D., Swanson, P. A., 2nd, Padilla, M., ... mRNA-1273 Study Group (2020). An mRNA Vaccine against SARS-CoV-2 Preliminary Report. The New England Journal of Medicine, 383(20), 1920–1931. https://doi.org/10.1056/NEJMoa2022483.
- 8. Tegally H, Wilkinson E, Giovanetti M, Iranzadeh A, Fonseca V, Giandhari J, Doolabh D, Pillay S, San EJ, Msomi N, et al. Emergence and rapid spread of a new severe acute respiratory syndrome-related coronavus 2 (SARS-CoV-2) lineage with multiple spike mutations in South Africa. MedRxiv 2020.12.21.20248640.
- 9. Wang P, Liu L, Iketani S, et al. Increased resistance of SARS-CoV-2 variants B.1.351 and B.1.1.7 to antibody neutralization. bioRxiv: the preprint server for biology, 2021.01.428137. https://doi.org/10.1101/2021.01.25.428137.
- 10. World Health Organization (WHO). (Data reported as of 13 Nov 2020). Weekly Operational Update on COVID-19. 2020a.
- https://www.who.int/publications/m/item/weekly-operational-update-on-covid-19---13-november-2020. Accessed 04 Feb 2021.
- 11. Wu, K., Werner, A. P., Moliva, J. I., Koch, M., Choi, A., Stewart-Jones, G., Bennett, H., Boyoglu-Barnum, S., Shi, W., Graham, B. S., Carfi, A., Corbett, K. S., Seder, R. A., & Edwards, D. K. (2021). mRNA-1273 vaccine induces neutralizing antibodies against spike mutants from global SARS-CoV-2 variants. bioRxiv: the preprint server for biology, 2021.01.25.427948. https://doi.org/10.1101/2021.01.25.427948.

## APPENDIX 1. TABLE MOCK-UPS

## LIST OF TABLES

| Table 1: | Study Design | 50 |
|---|---|---|
| Table 2: | Schedule of Study Procedures | 51 |
| Table 3: | Sample Size/Probability Estimates | 52 |
| Table 4: | Distribution of Protocol Deviations by Category, Type, and Treatment<br>Group | 53 |
| Table 5: | Distribution of Major Protocol Deviations by Category, Type, and Treatment Group | 53 |
| Table 6: | Subject Disposition by Treatment Group | 54 |
| Table 7: | Analysis Populations by Treatment Group - All Subjects | 55 |
| Table 8: | Ineligibility Summary of Screen Failures | 56 |
| Table 9: | Summary of Categorical Demographic and Baseline Characteristics by Treatment Group | 57 |
| Table 10: | Summary of Continuous Demographic and Baseline Characteristics by Treatment Group | 58 |
| Table 11: | Summary of Subjects with Pre-Existing Medical Conditions by MedDRA System Organ Class and Treatment Group | 59 |
| Table 12: | Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIA Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P–Wa-1 – mITT Population | 60 |
| Table 13: | Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIA Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P–Wa-1 – Per Protocol Population | 61 |
| Table 14: | Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIA<br>Geometric Mean Results with 95% Confidence Intervals by Time Point and<br>Treatment Group, RBD–Wa-1 – mITT Population | 61 |
| Table 15: | Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIA<br>Geometric Mean Results with 95% Confidence Intervals by Time Point and<br>Treatment Group, RBD–Wa-1 – Per Protocol Population | 61 |
| Table 16: | Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIAv2 (4-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P–Wa-1 – mITT Population | 61 |
| Table 17: | Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIAv2 (4-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P–Wa-1 – Per Protocol Population | 61 |

| Table 18: | Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIAv2 (4-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P–B.1.351 – mITT Population |
|---|---|
| Table 19: | Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIAv2 (4-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P–B.1.351 – Per Protocol Population |
| Table 20: | Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIAv2 (4-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, RBD–B.1.351 – mITT Population |
| Table 21: | Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIAv2 (4-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, RBD–B.1.351 – Per Protocol Population |
| Table 22: | Serum IgG Binding Assay Binding Antibody Units/mL Measured by ECLIAv2 (4-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P–Wa-1 – mITT Population62 |
| Table 23: | Serum IgG Binding Assay Binding Antibody Units/mL Measured by ECLIAv2 (4-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P–Wa-1 – Per Protocol Population62 |
| Table 24: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P–Wa-1 – mITT Population |
| Table 25: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P–Wa-1 – Per Protocol Population |
| Table 26: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P–B.1.351 – mITT Population |
| Table 27: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P–B.1.351 – Per Protocol Population |
| Table 28: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P–B.1.617.2 – mITT Population |
| Table 29: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P–B.1.617.2 – Per Protocol Population |
| Table 30: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P–P.1 – mITT Population |

| Table 31: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P–P.1 – Per Protocol Population | 63 |
|---|---|---|
| Table 32: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P–B.1.1.7 – mITT Population | 63 |
| Table 33: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P–B.1.1.7 – Per Protocol Population | 63 |
| Table 34: | Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G – mITT Population | 64 |
| Table 35: | Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G – Per Protocol Population | 65 |
| Table 36: | Pseudovirus Neutralization Assay ID <sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G – mITT Population | 65 |
| Table 37: | Pseudovirus Neutralization Assay ID <sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G – Per Protocol Population | 65 |
| Table 38: | Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 – mITT Population | 65 |
| Table 39: | Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 – Per Protocol Population | 65 |
| Table 40: | Pseudovirus Neutralization Assay ID <sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 – mITT Population | 66 |
| Table 41: | Pseudovirus Neutralization Assay ID <sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 – Per Protocol Population | 66 |
| Table 42: | Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.617.2 – mITT Population | |
| Table 43: | Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.617.2 – Per Protocol Population | |

| Table 44: | Pseudovirus Neutralization Assay ID <sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.617.2 – mITT Population | 66 |
|---|---|---|
| Table 45: | Pseudovirus Neutralization Assay ID <sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.617.2 – Per Protocol Population | 66 |
| Table 46: | Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, P.1 – mITT Population | 66 |
| Table 47: | Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, P.1 – Per Protocol Population | 66 |
| Table 48: | Pseudovirus Neutralization Assay ID <sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, P.1 – mITT Population | 66 |
| Table 49: | Pseudovirus Neutralization Assay ID <sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, P.1 – Per Protocol Population | 66 |
| Table 50: | Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.7 – mITT Population | 66 |
| Table 51: | Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.7 – Per Protocol Population | 66 |
| Table 52: | Pseudovirus Neutralization Assay ID <sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.7 – mITT Population | 66 |
| Table 53: | Pseudovirus Neutralization Assay ID <sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.7 – Per Protocol Population | 67 |
| Table 54: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G – mITT Population | 68 |
| Table 55: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G – Per Protocol Population | |
| Table 56: | Focus Reduction Neutralization Test ID <sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G – mITT Population | |

| Table 57: | Focus Reduction Neutralization Test ID <sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G – Per Protocol Population | 69 |
|---|---|---|
| Table 58: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 – mITT Population | 69 |
| Table 59: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 – Per Protocol Population | 70 |
| Table 60: | Focus Reduction Neutralization Test ID <sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 – mITT Population | 70 |
| Table 61: | Focus Reduction Neutralization Test ID <sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 – Per Protocol Population | 70 |
| Table 62: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.617.2 – mITT Population | 70 |
| Table 63: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.617.2 – Per Protocol Population | 70 |
| Table 64: | Focus Reduction Neutralization Test ID <sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.617.2 – mITT Population | 70 |
| Table 65: | Focus Reduction Neutralization Test ID <sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.617.2 – Per Protocol Population | 70 |
| Table 66: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, P.1 – mITT Population | |
| Table 67: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, P.1 – Per Protocol Population | |
| Table 68: | Focus Reduction Neutralization Test ID <sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, P.1 – mITT Population | |
| Table 69: | Focus Reduction Neutralization Test ID <sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, P.1 – Per Protocol Population | |

| Table 70: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.7 – mITT Population | 70 |
|---|---|---|
| Table 71: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.7 – Per Protocol Population | 70 |
| Table 72: | Focus Reduction Neutralization Test ID <sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.7 – mITT Population | 71 |
| Table 73: | Focus Reduction Neutralization Test ID <sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.7 – Per Protocol Population | 71 |
| Table 74: | Mean Percentages of CD4 T Cells Expressing Cytokines with 95% CI – mITT Population. | 72 |
| Table 75: | Mean Percentages of CD4 T Cells Expressing Cytokines with 95% CI – Per Protocol Population | 80 |
| Table 76: | Mean Percentages of CD8 T Cells Expressing Cytokines with 95% CI – mITT Population | 81 |
| Table 77: | Mean Percentages of CD8 T Cells Expressing Cytokines with 95% CI – Per Protocol Population | 88 |
| Table 78: | Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIA<br>Geometric Mean Fold Rise and 4-Fold Rise Results by Time Point and<br>Treatment Group, S-2P–Wa-1 – mITT Population | 89 |
| Table 79: | Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIA<br>Geometric Mean Fold Rise and 4-Fold Rise Results with 95% Confidence<br>Intervals by Time Point and Treatment Group, S-2P–Wa-1 – Per Protocol<br>Population | 90 |
| Table 80: | Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIA<br>Geometric Mean Fold Rise and 4-Fold Rise Results with 95% Confidence<br>Intervals by Time Point and Treatment Group, RBD–Wa-1 – mITT<br>Population | 90 |
| Table 81: | Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIA<br>Geometric Mean Fold Rise and 4-Fold Rise Results with 95% Confidence<br>Intervals by Time Point and Treatment Group, RBD–Wa-1 – Per Protocol<br>Population | 90 |
| Table 82: | Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIAv2 (4-plex) Geometric Mean Fold Rise and 4-Fold Rise Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P–Wa-1 – mITT Population | 90 |

| Table 83: | Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIAv2 (4-plex) Geometric Mean Fold Rise and 4-Fold Rise Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-Wa-1 – Per Protocol Population | 90 |
|---|---|---|
| Table 84: | Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIAv2 (4-plex) Geometric Mean Fold Rise and 4-Fold Rise Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P–B.1.351 – mITT Population. | 90 |
| Table 85: | Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIAv2 (4-plex) Geometric Mean Fold Rise and 4-Fold Rise Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P–B.1.351 – Per Protocol Population | 90 |
| Table 86: | Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIAv2 (4-plex) Geometric Mean Fold Rise and 4-Fold Rise Results with 95% Confidence Intervals by Time Point and Treatment Group, RBD–B.1.351 – mITT Population | 90 |
| Table 87: | Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIAv2 (4-plex) Geometric Mean Fold Rise and 4-Fold Rise Results with 95% Confidence Intervals by Time Point and Treatment Group, RBD–B.1.351 – Per Protocol Population | 90 |
| Table 88: | Serum IgG Binding Assay Binding Antibody Units/mL Measured by ECLIAv2 (4-plex) Geometric Mean Fold Rise and 4-Fold Rise Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P–Wa-1 – mITT Population | 90 |
| Table 89: | Serum IgG Binding Assay Binding Antibody Units/mL Measured by ECLIAv2 (4-plex) Geometric Mean Fold Rise and 4-Fold Rise Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P–Wa-1 – Per Protocol Population | 91 |
| Table 90: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Fold Rise and 4-Fold Rise Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P–Wa-1 – mITT Population | 91 |
| Table 91: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Fold Rise and 4-Fold Rise Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P–Wa-1 – Per Protocol Population | 91 |
| Table 92: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Fold Rise and 4-Fold Rise Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P–B.1.351 – mITT Population | 91 |

| Table 93: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Fold Rise and 4-Fold Rise Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P–B.1.351 – Per Protocol Population | 91 |
|---|---|---|
| Table 94: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Fold Rise and 4-Fold Rise Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P–B.1.617.2 – mITT Population. | 91 |
| Table 95: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Fold Rise and 4-Fold Rise Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P–B.1.617.2 – Per Protocol Population | 91 |
| Table 96: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Fold Rise and 4-Fold Rise Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P–P.1 – mITT Population | 91 |
| Table 97: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Fold Rise and 4-Fold Rise Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P–P.1 – Per Protocol Population | 91 |
| Table 98: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Fold Rise and 4-Fold Rise Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P–B.1.1.7 – mITT Population. | 91 |
| Table 99: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Fold Rise and 4-Fold Rise Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P–B.1.1.7 – Per Protocol Population | 91 |
| Table 100: | Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean Fold Rise and 4-Fold Rise Results by Time Point and Treatment Group, S-2P–Wa-1, mITT Population | 92 |
| Table 101: | Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean Fold Rise and 4-Fold Rise Results by Time Point and Treatment Group, D614G – Per Protocol Population | 93 |
| Table 102: | Pseudovirus Neutralization Assay ID <sub>80</sub> Geometric Mean Fold Rise and 4-Fold Rise Results by Time Point and Treatment Group,1 D614G – mITT Population | 93 |
| Table 103: | Pseudovirus Neutralization Assay ID <sub>80</sub> Geometric Mean Fold Rise and 4-Fold Rise Results by Time Point and Treatment Group, D614G – Per Protocol Population | 93 |

| Table 104: | Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean Fold Rise and 4-Fold Rise Results by Time Point and Treatment Group, B.1.351 – mITT Population | 93 |
|---|---|---|
| Table 105: | Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean Fold Rise and 4-Fold Rise Results by Time Point and Treatment Group, B.1.351 – Per Protocol Population | 93 |
| Table 106: | Pseudovirus Neutralization Assay ID <sub>80</sub> Geometric Mean Fold Rise and 4-Fold Rise Results by Time Point and Treatment Group, B.1.351 – mITT Population | 93 |
| Table 107: | Pseudovirus Neutralization Assay ID <sub>80</sub> Geometric Mean Fold Rise and 4-Fold Rise Results by Time Point and Treatment Group, B.1.351 – Per Protocol Population | 93 |
| Table 108: | Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean Fold Rise and 4-Fold Rise Results by Time Point and Treatment Group, B.1.617.2 – mITT Population | 93 |
| Table 109: | Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean Fold Rise and 4-Fold Rise Results by Time Point and Treatment Group, B.1.617.2 – Per Protocol Population | 93 |
| Table 110: | Pseudovirus Neutralization Assay ID <sub>80</sub> Geometric Mean Fold Rise and 4-Fold Rise Results by Time Point and Treatment Group, B.1.617.2 – mITT Population | 93 |
| Table 111: | Pseudovirus Neutralization Assay ID <sub>80</sub> Geometric Mean Fold Rise and 4-Fold Rise Results by Time Point and Treatment Group, B.1.617.2 – Per Protocol Population | 93 |
| Table 112: | Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean Fold Rise and 4-Fold Rise Results by Time Point and Treatment Group, P.1 – mITT Population | 93 |
| Table 113: | Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean Fold Rise and 4-Fold Rise Results by Time Point and Treatment Group, P.1 – Per Protocol Population | 94 |
| Table 114: | Pseudovirus Neutralization Assay ID <sub>80</sub> Geometric Mean Fold Rise and 4-Fold Rise Results by Time Point and Treatment Group, P.1 – mITT Population | 94 |
| Table 115: | Pseudovirus Neutralization Assay ID <sub>80</sub> Geometric Mean Fold Rise and 4-Fold Rise Results by Time Point and Treatment Group, P.1 – Per Protocol Population | |
| Table 116: | Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean Fold Rise and 4-Fold Rise Results by Time Point and Treatment Group, B.1.1.7 – mITT Population | |

| Table 117: | Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean Fold Rise and 4-Fold Rise Results by Time Point and Treatment Group, B.1.1.7 – Per Protocol Population | 94 |
|---|---|---|
| Table 118: | Pseudovirus Neutralization Assay ID <sub>80</sub> Geometric Mean Fold Rise and 4-Fold Rise Results by Time Point and Treatment Group, B.1.1.7 – mITT Population | 94 |
| Table 119: | Pseudovirus Neutralization Assay ID <sub>80</sub> Geometric Mean Fold Rise and 4-Fold Rise Results by Time Point and Treatment Group, B.1.1.7 – Per Protocol Population | 94 |
| Table 120: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean Fold Rise and 4-Fold Rise Results by Time Point and Treatment Group, S-2P–Wa-1 – mITT Population | 95 |
| Table 121: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean Fold Rise and 4-Fold Rise Results by Time Point and Treatment Group, D614G – Per Protocol Population | 96 |
| Table 122: | Focus Reduction Neutralization Test ID <sub>80</sub> Geometric Mean Fold Rise and 4-Fold Rise Results by Time Point and Treatment Group, D614G – mITT Population | 96 |
| Table 123: | Focus Reduction Neutralization Test ID <sub>80</sub> Geometric Mean Fold Rise and 4-Fold Rise Results by Time Point and Treatment Group, D614G – Per Protocol Population | 96 |
| Table 124: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean Fold Rise and 4-Fold Rise Results by Time Point and Treatment Group, B.1.351 – mITT Population | 96 |
| Table 125: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean Fold Rise and 4-Fold Rise Results by Time Point and Treatment Group, B.1.351 – Per Protocol Population | 96 |
| Table 126: | Focus Reduction Neutralization Test ID <sub>80</sub> Geometric Mean Fold Rise and 4-Fold Rise Results by Time Point and Treatment Group, B.1.351 – mITT Population | 96 |
| Table 127: | Focus Reduction Neutralization Test ID <sub>80</sub> Geometric Mean Fold Rise and 4-Fold Rise Results by Time Point and Treatment Group, B.1.351 – Per Protocol Population | |
| Table 128: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean Fold Rise and 4-Fold Rise Results by Time Point and Treatment Group, B.1.617.2 – mITT Population | |
| Table 129: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean Fold Rise and 4-Fold Rise Results by Time Point and Treatment Group, B.1.617.2 – Per Protocol Population | |

| Table 130: | Focus Reduction Neutralization Test ID <sub>80</sub> Geometric Mean Fold Rise and 4-Fold Rise Results by Time Point and Treatment Group, B.1.617.2 – mITT Population | 96 |
|---|---|---|
| Table 131: | Focus Reduction Neutralization Test ID <sub>80</sub> Geometric Mean Fold Rise and 4-Fold Rise Results by Time Point and Treatment Group, B.1.617.2 – Per Protocol Population | 96 |
| Table 132: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean Fold Rise and 4-Fold Rise Results by Time Point and Treatment Group, P.1 – mITT Population | 96 |
| Table 133: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean Fold Rise and 4-Fold Rise Results by Time Point and Treatment Group, P.1 – Per Protocol Population | 97 |
| Table 134: | Focus Reduction Neutralization Test ID <sub>80</sub> Geometric Mean Fold Rise and 4-Fold Rise Results by Time Point and Treatment Group, P.1 – mITT Population | 97 |
| Table 135: | Focus Reduction Neutralization Test ID <sub>80</sub> Geometric Mean Fold Rise and 4-Fold Rise Results by Time Point and Treatment Group, P.1 – Per Protocol Population | 97 |
| Table 136: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean Fold Rise and 4-Fold Rise Results by Time Point and Treatment Group, B.1.1.7 – mITT Population | 97 |
| Table 137: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean Fold Rise and 4-Fold Rise Results by Time Point and Treatment Group, B.1.1.7 – Per Protocol Population | |
| Table 138: | Focus Reduction Neutralization Test ID <sub>80</sub> Geometric Mean Fold Rise and 4-Fold Rise Results by Time Point and Treatment Group, B.1.1.7 – mITT Population | 97 |
| Table 139: | Focus Reduction Neutralization Test ID <sub>80</sub> Geometric Mean Fold Rise and 4-Fold Rise Results by Time Point and Treatment Group, B.1.1.7 – Per Protocol Population | 97 |
| Table 140: | Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean Ratio to D614G Variant with 95% Confidence Intervals by Variant, Time Point, and Treatment Group – mITT Population | 98 |
| Table 141: | Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean Ratio to D614G Variant with 95% Confidence Intervals by Variant, Time Point, and Treatment Group – Per Protocol Population | 102 |
| Table 142: | Pseudovirus Neutralization Assay ID <sub>80</sub> Geometric Mean Ratio to D614G Variant with 95% Confidence Intervals by Variant, Time Point, and Treatment Group – mITT Population | |

| Table 143: | Pseudovirus Neutralization Assay ID <sub>80</sub> Geometric Mean Ratio to D614G Variant with 95% Confidence Intervals by Variant, Time Point, and Treatment Group – Per Protocol Population | 102 |
|---|---|---|
| Table 144: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean Ratio to D614G Variant with 95% Confidence Intervals by Variant, Time Point, and Treatment Group – mITT Population | 103 |
| Table 145: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean Ratio to D614G Variant with 95% Confidence Intervals by Variant, Time Point, and Treatment Group – Per Protocol Population | 107 |
| Table 146: | Focus Reduction Neutralization Test ID <sub>80</sub> Geometric Mean Ratio to D614G Variant with 95% Confidence Intervals by Variant, Time Point, and Treatment Group – mITT Population | 107 |
| Table 147: | Focus Reduction Neutralization Test ID <sub>80</sub> Geometric Mean Ratio to D614G Variant with 95% Confidence Intervals by Variant, Time Point, and Treatment Group – Per Protocol Population | 107 |
| Table 148: | Overall Summary of Adverse Events by Treatment Group - All Subjects | 108 |
| Table 149: | Serious Adverse Events and Non-Serious Adverse Events Occurring in 5% of Subjects in Any Treatment Group by MedDRA System Organ Class and Preferred Term, and Treatment Group - All Subjects | 110 |
| Table 150: | Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Maximum Severity, and Treatment Group | 111 |
| Table 151: | Summary of Solicited Events by Days Post Treatment, Symptom, and Treatment Group – 50 µg mRNA-1273.351 | 115 |
| Table 152: | Summary of Solicited Events by Days Post Treatment, Symptom, and Treatment Group $-25~\mu g$ mRNA-1273 $+25~\mu g$ mRNA-1273.351 | 118 |
| Table 153: | Summary of Duration of Solicited Symptoms by Treatment Group - All Subjects | 119 |
| Table 154: | All Adverse Events Cross-Classified by MedDRA System Organ Class,<br>Severity, Relationship to Study Treatment, and Treatment Group | 123 |
| Table 155: | Summary of All Unsolicited Adverse Events by MedDRA System Organ Class and Preferred Term, Severity, Relationship, and Treatment Group | 125 |
| Table 156: | Number and Percentage of Subjects Experiencing Unsolicited Adverse Events by MedDRA® System Organ Class and Preferred Term, Severity, Relationship, and Treatment Group | 126 |
| Table 157: | Listing of Serious Adverse Events | 127 |
| Table 158: | Listing of Non-Serious, Unsolicited, Moderate or Severe Adverse Events | 128 |
| Table 159: | Listing of MAAEs and NOCMCs | 129 |

| Table 160: | Vital Signs by Assessment, Maximum Severity, Time Point, and Treatment Group, Any Assessment – All Subjects | 131 |
|---|---|---|
| Table 161: | Vital Signs by Assessment, Maximum Severity, Time Point, and Treatment Group, Systolic Blood Pressure – All Subjects | 133 |
| Table 162: | Vital Signs by Assessment, Maximum Severity, Time Point, and Treatment Group, Diastolic Blood Pressure – All Subjects | 133 |
| Table 163: | Vital Signs by Assessment, Maximum Severity, Time Point, and Treatment Group, Pulse Rate – All Subjects | 133 |
| Table 164: | Vital Signs by Assessment, Maximum Severity, Time Point, and Treatment Group, Temperature – All Subjects | 133 |
| Table 165: | Number and Percentage of Subjects with Prior and Concurrent Medications by WHO Drug Classification and Treatment Group – All Subjects | 134 |

## 9.1 Overall Study Design and Plan Description

Table 1: Study Design

| Arm | Sample Size | Vaccination Product and Dose |
|-----|-------------|--------------------------------------------|
| 1A | ~30 | 50 mcg mRNA-1273.351 |
| 1B | ~30 | 25 mcg mRNA-1273<br>+ 25 mcg mRNA-1273.351 |

## 9.5.1 Efficacy/Immunogenicity and Safety Measurements Assessed and Flow Chart

**Table 2:** Schedule of Study Procedures

| Study Day | -42 to -1 | 1 | 8* | 15 | 29 | 91 | 181 | 366 | Unscheduled<br>Visit | Early Termination<br>Visit |
|---|---|---|---|---|---|---|---|---|---|---|
| Visit Window (±number of days) | | 0 | 1 | 2 | 2 | 7 | 7 | 14 | | |
| Study Visit | Screening<br>(optional)<br>00 | 01 | 02 | 03 | 04 | 05 | 06 | 07 | | |
| Informed Consent | X | Xa | | | | | | | | |
| Review Eligibility Criteria | X | X | | | | | | | | |
| Medical History | X | Xa | | | | | | | | |
| Vaccination | | X | | | | | | | | |
| Concomitant Medications | | X | X | X | X | | | | | |
| Interim History | | $X^{b}$ | | X | X | X | X | X | X | X |
| Symptom-Directed Physical Examination | X | X | | X | X | X | X | X | X | X |
| Vital Signs <sup>c</sup> | | X | | X | X | X | X | X | X | X |
| Height and Weight (for BMI) | X | Xa | | | | | | | | |
| Pregnancy Test <sup>d</sup> | | X | | | | | | | | |
| Memory Aid: Solicited AEs | | X | X | Xe | | | | | | |
| Unsolicited AEs | | X | X | X | X | | | | X | X |
| SAEs, Protocol Specified AESIs, MAAEs, and NOCMCs | | X | X | X | X | X | X | X | X | X |
| Serum for Serological Immunogenicity Assays | | X | | X | X | X | X | X | | X |
| Peripheral Blood Mononuclear Cells (PBMCs) for<br>Cellular Immunology Assays (and Plasma) | | X | | X | | | X | X | | X |

<sup>\*</sup> Telephone call.

- a) If not performed at Visit 00.
- b) If medical history performed at Visit 00, then interim history at Visit 01.
- c) Vital signs to be obtained pre and post vaccination. Otherwise, only as clinically indicated.
- d) For women of childbearing potential, a negative urine pregnancy test on Day 1 with results confirmed prior to enrollment.
- e) Collect Memory Aid and assess for delayed onset local reactions.

## 9.7.1 Sample Size

**Table 3:** Sample Size/Probability Estimates

| | Cohort 1 | | | | |
|---|---|---|---|---|---|
| N | "True" Event<br>Rate | Probability of Observation (%) | N | "True" Event<br>Rate | Probability of Observation (%) |
| | 0.1% | 3.0 | | 0.1% | 5.8 |
| | 0.5% | 14.0 | | 0.5% | 26.0 |
| | 1.0% | 26.0 | | 1.0% | 45.3 |
| | 2.0% | 45.5 | | 2.0% | 70.2 |
| 20 | 3.0% | 59.9 | 60 | 3.0% | 83.9 |
| 30 | 4.0% | 70.6 | 60 | 4.0% | 91.4 |
| | 5.0% | 78.5 | | 5.0% | 95.4 |
| | 10.0% | 95.8 | | 10.0% | 99.8 |
| | 15.0% | 99.2 | | 15.0% | >99.9 |
| | 20.0% | 99.9 | | 20.0% | >99.9 |

### **10.2** Protocol Deviations

## Table 4: Distribution of Protocol Deviations by Category, Type, and Treatment Group

[Implementation Note: Below are example categories and deviation types. All reported categories and deviations types will be presented.]

| | | 50 μg<br>mRNA-1273.351<br>(N=X) | | mRNA<br>25<br>mRNA - | μg<br>-1273 +<br>μg<br>1273.351<br>=X) | All Su<br>(N= | bjects<br>=X) |
|---|---|---|---|---|---|---|---|
| Category | Deviation Type | # of<br>Subj. | # of<br>Dev. | # of<br>Subj. | # of<br>Dev. | # of<br>Subj. | # of<br>Dev. |
| Follow-up visit schedule | Missed visit/visit not conducted | | | | | | |
| | Out of window visit | | | | | | |
| Protocol procedure/assessment | Other: breach of confidentiality | | | | | | |
| | Other: non-required lab tests performed | | | | | | |
| | Required procedure done incorrectly | | | | | | |
| | Required procedure not conducted | | | | | | |
| | Specimen result not obtained | | | | | | |
| | Too few aliquots obtained | | | | | | |
| Treatment administration schedule | Required procedure done incorrectly | | | | | | |

Table with Similar Format:

Table 5: Distribution of Major Protocol Deviations by Category, Type, and Treatment Group

#### 14.1 **Description of Study Subjects**

# 14.1.1 Disposition of Subjects

Table 6: **Subject Disposition by Treatment Group** 

| | 50 μg<br>mRNA-1273.351<br>(N=X) | | 25 μg<br>mRNA -1273 +<br>25 μg<br>mRNA -1273.351<br>(N=X) | | | Subjects<br>N=X) |
|---|---|---|---|---|---|---|
| Subject Disposition | n | % | n % | | n | % |
| Screened | | | | | | |
| Enrolled | | | | | | |
| Received the third vaccination | | | | | | |
| Early termination <sup>a</sup> | | | | | | |
| Completed study | | | | | | |
| <sup>a</sup> Refer to Listing 2 for reasons subjects discontinued | or terminated | early. | • | <u>'</u> | | |

**Table 7:** Analysis Populations by Treatment Group - All Subjects

| Analysis Populations | Reason Subjects Excluded | 50 μg<br>mRNA-1273.351<br>(N=X) | | mRNA<br>25<br>mRNA - | μg<br>-1273 +<br>μg<br>1273.351<br>=X) | | ıbjects<br>=X) |
|---|---|---|---|---|---|---|---|
| | | % | n | % | n | % | n |
| Safety | Any Reason | X | XX | X | XX | X | xx |
| Modified Intent-To-Treat | Any Reason | | | | | | |
| Per Protocol | Any Reason | | | | | | |
| | [Reason 1] | | | | | | |

Note: The subjects removed from the Per Protocol Population were in Cohorts X and on visits post Day 29 were removed.

**Table 8:** Ineligibility Summary of Screen Failures

| Inclusion/Exclusion Category | Inclusion/Exclusion Criterion | n <sup>a</sup> | % b |
|---|---|---|---|
| Inclusion and Exclusion | Number of subjects failing any eligibility criterion | X | 100 |
| Inclusion | Any inclusion criterion | X | XX |
| | [inclusion criterion 1] | X | XX |
| | [inclusion criterion 2] | X | XX |
| | [inclusion criterion 3] | X | XX |
| Exclusion | Any exclusion criterion | X | XX |
| | [exclusion criterion 1] | X | XX |
| | [exclusion criterion 2] | X | XX |
| | [exclusion criterion 3] | X | XX |

<sup>&</sup>lt;sup>a</sup> More than one criterion may be marked per subject.

<sup>&</sup>lt;sup>b</sup> Denominator for percentages is the total number of screen failures.

# 14.1.2 Demographic Data by Treatment Group

Table 9: Summary of Categorical Demographic and Baseline Characteristics by Treatment Group

| | | mRNA- | 50 μg<br>mRNA-1273.351<br>(N=X) | | 25 μg<br>mRNA -1273 +<br>25 μg<br>mRNA -1273.351<br>(N=X) | | bjects<br>=X) |
|---|---|---|---|---|---|---|---|
| Demographic Category | Characteristic | n | % | n | % | n | % |
| Sex | Male | | | | | | |
| | Female | | | | | | |
| Ethnicity | Not Hispanic or Latino | | | | | | |
| | Hispanic or Latino | | | | | | |
| | Not Reported | | | | | | |
| | Unknown | | | | | | |
| Race | American Indian or<br>Alaska Native | | | | | | |
| | Asian | | | | | | |
| | Native Hawaiian or other Pacific Islander | | | | | | |
| | Black | | | | | | |
| | White | | | | | | |
| | Multi Racial | | | | | | |
| | Unknown | | | | | | |

Table 10: Summary of Continuous Demographic and Baseline Characteristics by Treatment Group

| Variable | Statistic | 50 μg<br>mRNA-1273.351<br>(N=X) | 25 μg<br>mRNA -1273 +<br>25 μg<br>mRNA -1273.351<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|
| Age (Years) | Mean | | | |
| | Standard Deviation | | | |
| | Median | | | |
| | Minimum | | | |
| | Maximum | | | |
| Height (cm) | Mean | | | |
| | Standard Deviation | | | |
| | Median | | | |
| | Minimum | | | |
| | Maximum | | | |
| Weight (kg) | Mean | | | |
| | Standard Deviation | | | |
| | Median | | | |
| | Minimum | | | |
| | Maximum | | | |
| BMI (kg/m²) | Mean | | | |
| | Standard Deviation | | | |
| | Median | | | |
| | Minimum | | | |
| | Maximum | | | |
| Time Between Dose 2 and Dose 3 | Mean | | | |
| (Days) | Standard Deviation | | | |
| | Median | | | |
| | Minimum | | | |
| | Maximum | | | |

### 14.1.3 Prior and Concurrent Medical Conditions

Table 11: Summary of Subjects with Pre-Existing Medical Conditions by MedDRA System Organ Class and Treatment Group

| MedDRA System Organ Class | 50 μg<br>mRNA-1273.351<br>(N=X) | | 25 μg<br>mRNA -1273 +<br>25 μg<br>mRNA -1273.351<br>(N=X) | | | ıbjects<br>=X) |
|---|---|---|---|---|---|---|
| | n | % | n | % | n | % |
| Any SOC | х | XX | X | XX | X | XX |
| [SOC 1] | | | | | | |
| [SOC 2] | | | | | | |

Note: N = Number of subjects in the Safety Population; n = Number of subjects reporting medical history within the specified SOC. A subject is only counted once per SOC.

## 14.2 Immunogenicity Data

Table 12: Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIA Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-Wa-1 – mITT Population

| Planned Time Point | Statistic | 50 μg<br>mRNA-1273.351<br>(N=X) | 25 μg<br>mRNA -1273 +<br>25 μg<br>mRNA -1273.351<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|
| Day 1, Pre-Booster Dose | n | | | |
| | GM | | | |
| | 95% CI | | | |
| Day 8 | n | | | |
| | GM | | | |
| | 95% CI | | | |
| Day 15 | n | | | |
| | GM | | | |
| | 95% CI | | | |
| Day 29 | n | | | |
| | GM | | | |
| | 95% CI | | | |
| Day 91 | n | | | |
| | GM | | | |
| | 95% CI | | | |
| Day 181 | n | | | |
| | GM | | | |

| | 95% CI |
|---------|--------|
| Day 366 | n |
| | GM |
| | 95% CI |
| Peak GM | n |
| | GM |
| | 95% CI |

Notes: N=Number of subjects in the mITT population.

n=Number of subjects with results available at time point.

GM=Geometric Mean, NE=Not Estimable.

Confidence intervals of the geometric means were calculated with the Student's t distribution on log-transformed data.

#### Tables with Similar Format:

### Implementation notes:

For tables using the PP population, update footnote to read: "Notes: N=Number of subjects in the Per Protocol population."

For all AUC tables, add footnote reading: "Geometric Mean is calculated as the Williams mean using log(1+x)."

- Table 13: Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIA Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-Wa-1 Per Protocol Population
- Table 14: Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIA Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, RBD-Wa-1 mITT Population
- Table 15: Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIA Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, RBD-Wa-1 Per Protocol Population
- Table 16: Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIAv2 (4-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-Wa-1 mITT Population
- Table 17: Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIAv2 (4-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-Wa-1 Per Protocol Population

- Table 18: Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIAv2 (4-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-B.1.351 mITT Population
- Table 19: Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIAv2 (4-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-B.1.351 Per Protocol Population
- Table 20: Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIAv2 (4-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, RBD-B.1.351 mITT Population
- Table 21: Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIAv2 (4-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, RBD-B.1.351 Per Protocol Population
- Table 22: Serum IgG Binding Assay Binding Antibody Units/mL Measured by ECLIAv2 (4-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-Wa-1 mITT Population
- Table 23: Serum IgG Binding Assay Binding Antibody Units/mL Measured by ECLIAv2 (4-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-Wa-1 Per Protocol Population
- Table 24: Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-Wa-1 mITT Population
- Table 25: Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-Wa-1 Per Protocol Population
- Table 26: Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-B.1.351 mITT Population
- Table 27: Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-B.1.351 Per Protocol Population
- Table 28: Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-B.1.617.2 mITT Population
- Table 29: Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-B.1.617.2 Per Protocol Population
- Table 30: Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-P.1 mITT Population

- Table 31: Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P–P.1 Per Protocol Population
- Table 32: Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-B.1.1.7 mITT Population
- Table 33: Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-B.1.1.7 Per Protocol Population

Table 34: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G – mITT Population

| Planned Time Point | Statistic | 50 μg<br>mRNA-1273.351<br>(N=X) | 25 μg<br>mRNA -1273 +<br>25 μg<br>mRNA -1273.351<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|
| Day 1, Pre-Booster Dose | n<br>GM | | | |
| | 95% CI | | | |
| Day 8 | n<br>GM<br>95% CI | | | |
| Day 15 | n<br>GM<br>95% CI | | | |
| Day 29 | n<br>GM<br>95% CI | | | |
| Day 91 | n<br>GM<br>95% CI | | | |
| Day 181 | n<br>GM<br>95% CI | | | |
| Day 366 | n | | | |

| Planned Time Point | Statistic | 50 μg<br>mRNA-1273.351<br>(N=X) | 25 μg<br>mRNA -1273 +<br>25 μg<br>mRNA -1273.351<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|
| | GM | | | |
| | 95% CI | | | |
| Peak GM | n | | | |
| | GM | | | |
| | 95% CI | | | |

Notes: N=Number of subjects in the mITT population.

n=Number of subjects with results available at time point.

GM=Geometric Mean, NE=Not Estimable.

Confidence intervals of the geometric means were calculated with the Student's t distribution on log-transformed data.

### Tables with Similar Format:

Implementation note: For tables using the PP population, update footnote to read: "Notes: N=Number of subjects in the Per Protocol population."

- Table 35: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G Per Protocol Population
- Table 36: Pseudovirus Neutralization Assay ID<sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G mITT Population
- Table 37: Pseudovirus Neutralization Assay ID<sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G Per Protocol Population
- Table 38: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 mITT Population
- Table 39: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 Per Protocol Population

- Table 40: Pseudovirus Neutralization Assay ID<sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 mITT Population
- Table 41: Pseudovirus Neutralization Assay ID<sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 Per Protocol Population
- Table 42: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.617.2 mITT Population
- Table 43: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.617.2 Per Protocol Population
- Table 44: Pseudovirus Neutralization Assay ID<sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.617.2 mITT Population
- Table 45: Pseudovirus Neutralization Assay ID<sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.617.2 Per Protocol Population
- Table 46: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, P.1 mITT Population
- Table 47: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, P.1 Per Protocol Population
- Table 48: Pseudovirus Neutralization Assay ID<sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, P.1 mITT Population
- Table 49: Pseudovirus Neutralization Assay ID<sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, P.1 Per Protocol Population
- Table 50: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.7 mITT Population
- Table 51: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.7 Per Protocol Population
- Table 52: Pseudovirus Neutralization Assay ID<sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.7 mITT Population

Table 53: Pseudovirus Neutralization Assay ID<sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.7 – Per Protocol Population

Table 54: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G – mITT Population

| Planned Time Point | Statistic | 50 μg<br>mRNA-1273.351<br>(N=X) | 25 μg<br>mRNA -1273 +<br>25 μg<br>mRNA -1273.351<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|
| Day 1, Pre-Booster Dose | n | | | |
| | GM | | | |
| | 95% CI | | | |
| Day 8 | n | | | |
| | GM | | | |
| | 95% CI | | | |
| Day 15 | n | | | |
| | GM | | | |
| | 95% CI | | | |
| Day 29 | n | | | |
| | GM | | | |
| | 95% CI | | | |
| Day 91 | n | | | |
| | GM | | | |
| | 95% CI | | | |
| Day 181 | n | | | |
| | GM | | | |
| | 95% CI | | | |
| Day 366 | n | | | |

| Planned Time Point | Statistic | 50 μg<br>mRNA-1273.351<br>(N=X) | 25 μg<br>mRNA -1273 +<br>25 μg<br>mRNA -1273.351<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|
| | GM | | | |
| | 95% CI | | | |
| Peak GM | n | | | |
| | GM | | | |
| | 95% CI | | | |

Notes: N=Number of subjects in the mITT population.

n=Number of subjects with results available at time point.

GM=Geometric Mean, NE=Not Estimable.

Confidence intervals of the geometric means were calculated with the Student's t distribution on log-transformed data.

### Tables with Similar Format:

Implementation note: For tables using the PP population, update footnote to read: "Notes: N=Number of subjects in the Per Protocol population."

- Table 55: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G Per Protocol Population
- Table 56: Focus Reduction Neutralization Test ID<sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G mITT Population
- Table 57: Focus Reduction Neutralization Test ID<sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, D614G Per Protocol Population
- Table 58: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 mITT Population

- Table 59: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 Per Protocol Population
- Table 60: Focus Reduction Neutralization Test ID<sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 mITT Population
- Table 61: Focus Reduction Neutralization Test ID<sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.351 Per Protocol Population
- Table 62: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.617.2 mITT Population
- Table 63: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.617.2 Per Protocol Population
- Table 64: Focus Reduction Neutralization Test ID<sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.617.2 mITT Population
- Table 65: Focus Reduction Neutralization Test ID<sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.617.2 Per Protocol Population
- Table 66: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, P.1 mITT Population
- Table 67: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, P.1 Per Protocol Population
- Table 68: Focus Reduction Neutralization Test ID<sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, P.1 mITT Population
- Table 69: Focus Reduction Neutralization Test ID<sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, P.1 Per Protocol Population
- Table 70: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.7 mITT Population
- Table 71: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.7 Per Protocol Population

- Table 72: Focus Reduction Neutralization Test ID<sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.7 mITT Population
- Table 73: Focus Reduction Neutralization Test ID<sub>80</sub> Geometric Mean Results with 95% Confidence Intervals by Time Point and Treatment Group, B.1.1.7 Per Protocol Population
Table 74: Mean Percentages of CD4 T Cells Expressing Cytokines with 95% CI – mITT Population

[Implementation Note: Tables should include rows for median, min, max, GMFR and 95% CI of GMFR. Column order should be Peptide Pool, Cytokine and Time Point.]

| Time Point | Peptide Pool | Cytokine | Statistic | 50 μg<br>mRNA-1273.351<br>(N=X) | 25 μg<br>mRNA -1273 +<br>25 μg<br>mRNA -1273.351<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|---|---|
| Day 1, Pre-Booster Dose | Beta Mutations | IFNγ | n | | | |
| | | | Mean | | | |
| | | | 95% CI <sup>a</sup> | | | |
| | | | Response Rate | | | |
| | | | 95% CI <sup>b</sup> | | | |
| | | IFNγ or IL-2 | n | | | |
| | | | Mean | | | |
| | | | 95% CI <sup>a</sup> | | | |
| | | | Response Rate | | | |
| | | | 95% CI <sup>b</sup> | | | |
| | | IFNγ or IL-2/CM | n | | | |
| | | | Mean | | | |
| | | | 95% CI <sup>a</sup> | | | |
| | | | Response Rate | | | |
| | | | 95% CI <sup>b</sup> | | | |
| | | IFNγ or IL-2/EM | n | | | |
| | | | Mean | | | |
| | | | 95% CI <sup>a</sup> | | | |
| | | | Response Rate | | | |

| Time Point | Peptide Pool | Cytokine | Statistic | 50 μg<br>mRNA-1273.351<br>(N=X) | 25 μg<br>mRNA -1273 +<br>25 μg<br>mRNA -1273.351<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|---|---|
| | | | 95% CI <sup>b</sup> | | | |
| | | IFNγ or IL-2/N | n | | | |
| | | | Mean | | | |
| | | | 95% CI <sup>a</sup> | | | |
| | | | Response Rate | | | |
| | | | 95% CI <sup>b</sup> | | | |
| | | IFNγ or IL-2/TD | n | | | |
| | | | Mean | | | |
| | | | 95% CI <sup>a</sup> | | | |
| | | | Response Rate | | | |
| | | | 95% CI <sup>b</sup> | | | |
| | | IFNγ or IL-2 and 154 | n | | | |
| | | | Mean | | | |
| | | | 95% CI <sup>a</sup> | | | |
| | | | Response Rate | | | |
| | | | 95% CI <sup>b</sup> | | | |
| | | IFNγ or IL-2 or 154 | n | | | |
| | | | Mean | | | |
| | | | 95% CI <sup>a</sup> | | | |
| | | | Response Rate | | | |
| | | | 95% CI <sup>b</sup> | | | |
| | | IFNγ or IL-2 or 154/C | n | | | |
| | | | Mean | | | |

| Time Point | Peptide Pool | Cytokine | Statistic | 50 μg<br>mRNA-1273.351<br>(N=X) | 25 μg<br>mRNA -1273 +<br>25 μg<br>mRNA -1273.351<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|---|---|
| | | | 95% CI <sup>a</sup> | | | |
| | | | Response Rate | | | |
| | | | 95% CI <sup>b</sup> | | | |
| | | IFNγ or IL-2 or 154/E | n | | | |
| | | | Mean | | | |
| | | | 95% CI <sup>a</sup> | | | |
| | | | Response Rate | | | |
| | | | 95% CI <sup>b</sup> | | | |
| | | IFNγ or IL-2 or 154/N | n | | | |
| | | | Mean | | | |
| | | | 95% CI <sup>a</sup> | | | |
| | | | Response Rate | | | |
| | | | 95% CI <sup>b</sup> | | | |
| | | IFNγ or IL-2 or 154/T | n | | | |
| | | | Mean | | | |
| | | | 95% CI <sup>a</sup> | | | |
| | | | Response Rate | | | |
| | | | 95% CI <sup>b</sup> | | | |
| | | IL-17a | n | | | |
| | | | Mean | | | |
| | | | 95% CI <sup>a</sup> | | | |
| | | | Response Rate | | | |
| | | | 95% CI <sup>b</sup> | | | |

| Time Point | Peptide Pool | Cytokine | Statistic | 50 μg<br>mRNA-1273.351<br>(N=X) | 25 μg<br>mRNA -1273 +<br>25 μg<br>mRNA -1273.351<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|---|---|
| | | IL-2 | n | | | |
| | | | Mean | | | |
| | | | 95% CI <sup>a</sup> | | | |
| | | | Response Rate | | | |
| | | | 95% CI <sup>b</sup> | | | |
| | | IL-4 and 154 | n | | | |
| | | | Mean | | | |
| | | | 95% CI <sup>a</sup> | | | |
| | | | Response Rate | | | |
| | | | 95% CI <sup>b</sup> | | | |
| | | IL-4 IL-5 IL-13 and 154 | n | | | |
| | | | Mean | | | |
| | | | 95% CI <sup>a</sup> | | | |
| | | | Response Rate | | | |
| | | | 95% CI <sup>b</sup> | | | |
| | | TNFα | n | | | |
| | | | Mean | | | |
| | | | 95% CI <sup>a</sup> | | | |
| | | | Response Rate | | | |
| | | | 95% CI <sup>b</sup> | | | |
| | Beta S | ΙΕΝγ | n | | | |
| | | | Mean | | | |
| | | | 95% CI <sup>a</sup> | | | |

| Time Point | Peptide Pool | Cytokine | Statistic | 50 μg<br>mRNA-1273.351<br>(N=X) | 25 μg<br>mRNA -1273 +<br>25 μg<br>mRNA -1273.351<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|---|---|
| | | | Response Rate | | | |
| | | | 95% CI <sup>b</sup> | | | |
| | | IFNγ or IL-2 | n | | | |
| | | | Mean | | | |
| | | | 95% CI <sup>a</sup> | | | |
| | | | Response Rate | | | |
| | | | 95% CI <sup>b</sup> | | | |
| | | IFNγ or IL-2/CM | n | | | |
| | | | Mean | | | |
| | | | 95% CI <sup>a</sup> | | | |
| | | | Response Rate | | | |
| | | | 95% CI <sup>b</sup> | | | |
| | | IFNγ or IL-2/EM | n | | | |
| | | | Mean | | | |
| | | | 95% CI <sup>a</sup> | | | |
| | | | Response Rate | | | |
| | | | 95% CI <sup>b</sup> | | | |
| | | | | Repeat for all cytokines | | |
| | Conserved S1 | IFNγ | n | | | |
| | | | Mean | | | |
| | | | 95% CI <sup>a</sup> | | | |
| | | | Response Rate | | | |
| | | | 95% CI <sup>b</sup> | | | |

| Time Point | Peptide Pool | Cytokine | Statistic | 50 μg<br>mRNA-1273.351<br>(N=X) | 25 μg<br>mRNA -1273 +<br>25 μg<br>mRNA -1273.351<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|---|---|
| | | IFNγ or IL-2 | n | | | |
| | | | Mean | | | |
| | | | 95% CI <sup>a</sup> | | | |
| | | | Response Rate | | | |
| | | | 95% CI <sup>b</sup> | | | |
| | | IFNγ or IL-2/CM | n | | | |
| | | | Mean | | | |
| | | | 95% CI <sup>a</sup> | | | |
| | | | Response Rate | | | |
| | | | 95% CI <sup>b</sup> | | | |
| | | IFNγ or IL-2/EM | n | | | |
| | | | Mean | | | |
| | | | 95% CI <sup>a</sup> | | | |
| | | | Response Rate | | | |
| | | | 95% CI <sup>b</sup> | | | |
| | | | | Repeat for all cytokines | | |
| | Conserved S2 | IFNγ | n | | | |
| | | | Mean | | | |
| | | | 95% CI <sup>a</sup> | | | |
| | | | Response Rate | | | |
| | | | 95% CI <sup>b</sup> | | | |
| | | IFNγ or IL-2 | n | | | |
| | | | Mean | | | |

| Time Point | Peptide Pool | Cytokine | Statistic | 50 μg<br>mRNA-1273.351<br>(N=X) | 25 μg<br>mRNA -1273 +<br>25 μg<br>mRNA -1273.351<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|---|---|
| | | | 95% CI <sup>a</sup> | | | |
| | | | Response Rate | | | |
| | | | 95% CI <sup>b</sup> | | | |
| | | IFNγ or IL-2/CM | n | | | |
| | | | Mean | | | |
| | | | 95% CI <sup>a</sup> | | | |
| | | | Response Rate | | | |
| | | | 95% CI <sup>b</sup> | | | |
| | | IFNγ or IL-2/EM | n | | | |
| | | | Mean | | | |
| | | | 95% CI <sup>a</sup> | | | |
| | | | Response Rate | | | |
| | | | 95% CI <sup>b</sup> | | | |
| | | | | Repeat for all cytokines | | |
| | Original Matched | ΙΕΝγ | n | | | |
| | | | Mean | | | |
| | | | 95% CI <sup>a</sup> | | | |
| | | | Response Rate | | | |
| | | | 95% CI <sup>b</sup> | | | |
| | IFNγ or IL-2 | n | | | | |
| | | | Mean | | | |
| | | | 95% CI <sup>a</sup> | | | |
| | | | Response Rate | | | |

| Time Point | Peptide Pool | Cytokine | Statistic | 50 μg<br>mRNA-1273.351<br>(N=X) | 25 μg<br>mRNA -1273 +<br>25 μg<br>mRNA -1273.351<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|---|---|
| | | | 95% CI <sup>b</sup> | | | |
| | | IFNγ or IL-2/CM | n | | | |
| | | | Mean | | | |
| | | | 95% CI <sup>a</sup> | | | |
| | | | Response Rate | | | |
| | | | 95% CI <sup>b</sup> | | | |
| | | IFNγ or IL-2/EM | n | | | |
| | | | Mean | | | |
| | | | 95% CI <sup>a</sup> | | | |
| | | | Response Rate | | | |
| | | | 95% CI <sup>b</sup> | | | |
| | | Repeat for all cytokines | | | | |
| | Original S | IFNγ | n | | | |
| | | | Mean | | | |
| | | | 95% CI <sup>a</sup> | | | |
| | | | Response Rate | | | |
| | | | 95% CI <sup>b</sup> | | | |
| | | IFNγ or IL-2 | n | | | |
| | | | Mean | | | |
| | | | 95% CI <sup>a</sup> | | | |
| | | | Response Rate | | | |
| | | | 95% CI <sup>b</sup> | | | |
| | | IFNγ or IL-2/CM | n | | | |

| Time Point | Peptide Pool | Cytokine | Statistic | 50 μg<br>mRNA-1273.351<br>(N=X) | 25 μg<br>mRNA -1273 +<br>25 μg<br>mRNA -1273.351<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|---|---|
| | | | Mean | | | |
| | | | 95% CI <sup>a</sup> | | | |
| | | | Response Rate | | | |
| | | | 95% CI <sup>b</sup> | | | |
| | | IFNγ or IL-2/EM | n | | | |
| | | | Mean | | | |
| | | | 95% CI <sup>a</sup> | | | |
| | | | Response Rate | | | |
| | | | 95% CI <sup>b</sup> | | | |
| | | | • | Repeat for all cytokines | | |

Repeat for all study days

Note: N=Number of Subjects.

n=Number of subjects with results available at time point.

NE=Not Estimable

## Table with Similar Format:

Table 75: Mean Percentages of CD4 T Cells Expressing Cytokines with 95% CI – Per Protocol Population

<sup>&</sup>lt;sup>a</sup> Confidence interval calculated based on the Student's t-distribution

<sup>&</sup>lt;sup>b</sup> Exact binomial confidence interval calculated using the Clopper-Pearson methodology.

# Table 76: Mean Percentages of CD8 T Cells Expressing Cytokines with 95% CI – mITT Population

[Implementation Note: Tables should include rows for median, min, max, GMFR and 95% CI of GMFR. Column order should be Peptide Pool, Cytokine and Time Point.]

| Time Point | Peptide Pool | Cytokine | Statistic | 50 μg<br>mRNA-1273.351<br>(N=X) | 25 μg<br>mRNA -1273 +<br>25 μg<br>mRNA -1273.351<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|---|---|
| Day 1, Pre-Booster Dose | Beta Mutations | IFNγ or IL-2 | n | | | |
| | | | Mean | | | |
| | | | 95% CI <sup>a</sup> | | | |
| | | | Response Rate | | | |
| | | | 95% CI <sup>b</sup> | | | |
| | | IFNγ or IL-2/CM | n | | | |
| | | | Mean | | | |
| | | | 95% CI <sup>a</sup> | | | |
| | | | Response Rate | | | |
| | | | 95% CI <sup>b</sup> | | | |
| | | IFNγ or IL-2/EM | n | | | |
| | | | Mean | | | |
| | | | 95% CI <sup>a</sup> | | | |
| | | | Response Rate | | | |
| | | | 95% CI <sup>b</sup> | | | |
| | | IFNγ or IL-2/N | n | | | |
| | | | Mean | | | |
| | | | 95% CI <sup>a</sup> | | | |
| | | | Response Rate | | | |

| Time Point | Peptide Pool | Cytokine | Statistic | 50 μg<br>mRNA-1273.351<br>(N=X) | 25 μg<br>mRNA -1273 +<br>25 μg<br>mRNA -1273.351<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|---|---|
| | | | 95% CI <sup>b</sup> | | | |
| | | IFNγ or IL-2/TD | n | | | |
| | | | Mean | | | |
| | | | 95% CI <sup>a</sup> | | | |
| | | | Response Rate | | | |
| | | | 95% CI <sup>b</sup> | | | |
| | Beta S | IFNγ or IL-2 | n | | | |
| | | | Mean | | | |
| | | | 95% CI <sup>a</sup> | | | |
| | | | Response Rate | | | |
| | | | 95% CI <sup>b</sup> | | | |
| | | IFNγ or IL-2/CM | n | | | |
| | | | Mean | | | |
| | | | 95% CI <sup>a</sup> | | | |
| | | | Response Rate | | | |
| | | | 95% CI <sup>b</sup> | | | |
| | | IFNγ or IL-2/EM | n | | | |
| | | | Mean | | | |
| | | | 95% CI <sup>a</sup> | | | |
| | | | Response Rate | | | |
| | | | 95% CI <sup>b</sup> | | | |
| | | IFNγ or IL-2/N | n | | | |
| | | | Mean | | | |

PREPARED BY EMMES

| Time Point | Peptide Pool | Cytokine | Statistic | 50 μg<br>mRNA-1273.351<br>(N=X) | 25 μg<br>mRNA -1273 +<br>25 μg<br>mRNA -1273.351<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|---|---|
| | | | 95% CI <sup>a</sup> | | | |
| | | | Response Rate | | | |
| | | | 95% CI <sup>b</sup> | | | |
| | | IFNγ or IL-2/TD | n | | | |
| | | | Mean | | | |
| | | | 95% CI <sup>a</sup> | | | |
| | | | Response Rate | | | |
| | | | 95% CI <sup>b</sup> | | | |
| | Conserved S1 | IFNγ or IL-2 | n | | | |
| | | | Mean | | | |
| | | | 95% CI <sup>a</sup> | | | |
| | | | Response Rate | | | |
| | | | 95% CI <sup>b</sup> | | | |
| | | IFNγ or IL-2/CM | n | | | |
| | | | Mean | | | |
| | | | 95% CI <sup>a</sup> | | | |
| | | | Response Rate | | | |
| | | | 95% CI <sup>b</sup> | | | |
| | | IFNγ or IL-2/EM | n | | | |
| | | | Mean | | | |
| | | | 95% CI <sup>a</sup> | | | |
| | | | Response Rate | | | |
| | | | 95% CI <sup>b</sup> | | | |

| Time Point | Peptide Pool | Cytokine | Statistic | 50 μg<br>mRNA-1273.351<br>(N=X) | 25 μg<br>mRNA -1273 +<br>25 μg<br>mRNA -1273.351<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|---|---|
| | | IFNγ or IL-2/N | n | | | |
| | | | Mean | | | |
| | | | 95% CI <sup>a</sup> | | | |
| | | | Response Rate | | | |
| | | | 95% CI <sup>b</sup> | | | |
| | | IFNγ or IL-2/TD | n | | | |
| | | | Mean | | | |
| | | | 95% CI <sup>a</sup> | | | |
| | | | Response Rate | | | |
| | | | 95% CI <sup>b</sup> | | | |
| | Conserved S2 | IFNγ or IL-2 | n | | | |
| | | | Mean | | | |
| | | | 95% CI <sup>a</sup> | | | |
| | | | Response Rate | | | |
| | | | 95% CI <sup>b</sup> | | | |
| | | IFNγ or IL-2/CM | n | | | |
| | | | Mean | | | |
| | | | 95% CI <sup>a</sup> | | | |
| | | | Response Rate | | | |
| | | | 95% CI <sup>b</sup> | | | |
| | | IFNγ or IL-2/EM | n | | | |
| | | | Mean | | | |
| | | | 95% CI <sup>a</sup> | | | |

| Time Point | Peptide Pool | Cytokine | Statistic | 50 μg<br>mRNA-1273.351<br>(N=X) | 25 μg<br>mRNA -1273 +<br>25 μg<br>mRNA -1273.351<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|---|---|
| | | | Response Rate | | | |
| | | | 95% CI <sup>b</sup> | | | |
| | | IFNγ or IL-2/N | n | | | |
| | | | Mean | | | |
| | | | 95% CI <sup>a</sup> | | | |
| | | | Response Rate | | | |
| | | | 95% CI <sup>b</sup> | | | |
| | | IFNγ or IL-2/TD | n | | | |
| | | | Mean | | | |
| | | | 95% CI <sup>a</sup> | | | |
| | | | Response Rate | | | |
| | | | 95% CI <sup>b</sup> | | | |
| | Original Matched | IFNγ or IL-2 | n | | | |
| | | | Mean | | | |
| | | | 95% CI <sup>a</sup> | | | |
| | | | Response Rate | | | |
| | | | 95% CI <sup>b</sup> | | | |
| | | IFNγ or IL-2/CM | n | | | |
| | | | Mean | | | |
| | | | 95% CI <sup>a</sup> | | | |
| | | | Response Rate | | | |
| | | | 95% CI <sup>b</sup> | | | |
| | | IFNγ or IL-2/EM | n | | | |

| Time Point | Peptide Pool | Cytokine | Statistic | 50 μg<br>mRNA-1273.351<br>(N=X) | 25 μg<br>mRNA -1273 +<br>25 μg<br>mRNA -1273.351<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|---|---|
| | | | Mean | | | |
| | | | 95% CI <sup>2</sup> | | | |
| | | | Response Rate | | | |
| | | | 95% CI <sup>b</sup> | | | |
| | | IFNγ or IL-2/N | n | | | |
| | | | Mean | | | |
| | | | 95% CI <sup>a</sup> | | | |
| | | | Response Rate | | | |
| | | | 95% CI <sup>b</sup> | | | |
| | | IFNγ or IL-2/TD | n | | | |
| | | | Mean | | | |
| | | | 95% CI <sup>a</sup> | | | |
| | | | Response Rate | | | |
| | | | 95% CI <sup>b</sup> | | | |
| | Original S | IFNγ or IL-2 | n | | | |
| | | | Mean | | | |
| | | | 95% CI <sup>a</sup> | | | |
| | | | Response Rate | | | |
| | | | 95% CI <sup>b</sup> | | | |
| | | IFNγ or IL-2/CM | n | | | |
| | | | Mean | | | |
| | | | 95% CI <sup>a</sup> | | | |
| | | | Response Rate | | | |

| Time Point | Peptide Pool | Cytokine | Statistic | 50 μg<br>mRNA-1273.351<br>(N=X) | 25 μg<br>mRNA -1273 +<br>25 μg<br>mRNA -1273.351<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|---|---|
| | | | 95% CI <sup>b</sup> | | | |
| | | IFNγ or IL-2/EM | n | | | |
| | | | Mean | | | |
| | | | 95% CI <sup>a</sup> | | | |
| | | | Response Rate | | | |
| | | | 95% CI <sup>b</sup> | | | |
| | | IFNγ or IL-2/N | n | | | |
| | | | Mean | | | |
| | | | 95% CI <sup>a</sup> | | | |
| | | | Response Rate | | | |
| | | | 95% CI <sup>b</sup> | | | |
| | | IFNγ or IL-2/TD | n | | | |
| | | | Mean | | | |
| | | | 95% CI <sup>a</sup> | | | |
| | | | Response Rate | | | |
| | | | 95% CI <sup>b</sup> | | | |

Repeat for all study days

Note: N=Number of Subjects.

n=Number of subjects with results available at time point.

NE=Not Estimable

<sup>a</sup> Confidence interval calculated based on the Student's t-distribution

Table 77: Mean Percentages of CD8 T Cells Expressing Cytokines with 95% CI – Per Protocol Population

Table 78: Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIA Geometric Mean Fold Rise and 4-Fold Rise Results by Time Point and Treatment Group, S-2P-Wa-1 – mITT Population

| Planned Time Point | Statistic | 50 μg<br>mRNA-1273.351<br>(N=X) | 25 μg<br>mRNA -1273 +<br>25 μg<br>mRNA -1273.351<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|
| Day 15 | n | | | |
| | GMFR (95% CI) <sup>a</sup> | | | |
| | 4-Fold Rise - % (95% CI) <sup>b</sup> | | | |
| Day 29 | n | | | |
| | GMFR (95% CI) <sup>a</sup> | | | |
| | 4-Fold Rise - % (95% CI) <sup>b</sup> | | | |
| Day 91 | n | | | |
| | GMFR (95% CI) <sup>a</sup> | | | |
| | 4-Fold Rise - % (95% CI) <sup>b</sup> | | | |
| Day 181 | n | | | |
| | GMFR (95% CI) <sup>a</sup> | | | |
| | 4-Fold Rise - % (95% CI) <sup>b</sup> | | | |
| Day 366 | n | | | |
| | GMFR (95% CI) <sup>a</sup> | | | |
| | 4-Fold Rise - % (95% CI) <sup>b</sup> | | | |

Notes: N=Number of subjects in the mITT population.

n=Number of subjects with results available at time point.

GMFR=Geometric Mean Fold Rise, NE=Not Estimable.

<sup>a</sup> Confidence interval calculated based on the Student's t-distribution

## Implementation notes:

- For tables using the PP population, update footnote to read: "Notes: N=Number of subjects in the Per Protocol population."
- For all AUC tables, add footnote reading: "AUC results reported as 0 were imputed to the lowest non-zero reported value for the purposes of fold-rise calculations."
- Table 79: Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIA Geometric Mean Fold Rise and 4-Fold Rise Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-Wa-1 Per Protocol Population
- Table 80: Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIA Geometric Mean Fold Rise and 4-Fold Rise Results with 95% Confidence Intervals by Time Point and Treatment Group, RBD-Wa-1 mITT Population
- Table 81: Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIA Geometric Mean Fold Rise and 4-Fold Rise Results with 95% Confidence Intervals by Time Point and Treatment Group, RBD-Wa-1 Per Protocol Population
- Table 82: Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIAv2 (4-plex) Geometric Mean Fold Rise and 4-Fold Rise Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-Wa-1 mITT Population
- Table 83: Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIAv2 (4-plex) Geometric Mean Fold Rise and 4-Fold Rise Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-Wa-1 Per Protocol Population
- Table 84: Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIAv2 (4-plex) Geometric Mean Fold Rise and 4-Fold Rise Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-B.1.351 mITT Population
- Table 85: Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIAv2 (4-plex) Geometric Mean Fold Rise and 4-Fold Rise Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-B.1.351 Per Protocol Population
- Table 86: Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIAv2 (4-plex) Geometric Mean Fold Rise and 4-Fold Rise Results with 95% Confidence Intervals by Time Point and Treatment Group, RBD-B.1.351 mITT Population
- Table 87: Serum IgG Binding Assay Arbitrary Units/mL Measured by ECLIAv2 (4-plex) Geometric Mean Fold Rise and 4-Fold Rise Results with 95% Confidence Intervals by Time Point and Treatment Group, RBD–B.1.351 Per Protocol Population
- Table 88: Serum IgG Binding Assay Binding Antibody Units/mL Measured by ECLIAv2 (4-plex) Geometric Mean Fold Rise and 4-Fold Rise Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-Wa-1 mITT Population

- Table 89: Serum IgG Binding Assay Binding Antibody Units/mL Measured by ECLIAv2 (4-plex) Geometric Mean Fold Rise and 4-Fold Rise Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-Wa-1 Per Protocol Population
- Table 90: Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Fold Rise and 4-Fold Rise Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-Wa-1 mITT Population
- Table 91: Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Fold Rise and 4-Fold Rise Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-Wa-1 Per Protocol Population
- Table 92: Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Fold Rise and 4-Fold Rise Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-B.1.351 mITT Population
- Table 93: Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Fold Rise and 4-Fold Rise Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-B.1.351 Per Protocol Population
- Table 94: Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Fold Rise and 4-Fold Rise Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-B.1.617.2 mITT Population
- Table 95: Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Fold Rise and 4-Fold Rise Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-B.1.617.2 Per Protocol Population
- Table 96: Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Fold Rise and 4-Fold Rise Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-P.1 mITT Population
- Table 97: Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Fold Rise and 4-Fold Rise Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-P.1 Per Protocol Population
- Table 98: Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Fold Rise and 4-Fold Rise Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-B.1.1.7 mITT Population
- Table 99: Serum IgG Binding Assay Area Under the Curve Measured by ECLIAv2 (10-plex) Geometric Mean Fold Rise and 4-Fold Rise Results with 95% Confidence Intervals by Time Point and Treatment Group, S-2P-B.1.1.7 Per Protocol Population

Table 100: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean Fold Rise and 4-Fold Rise Results by Time Point and Treatment Group, S-2P-Wa-1, mITT Population

| Planned Time Point | Statistic | 50 μg<br>mRNA-1273.351<br>(N=X) | 25 μg<br>mRNA -1273 +<br>25 μg<br>mRNA -1273.351<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|
| Day 15 | n | | | |
| | GMFR (95% CI) <sup>a</sup> | | | |
| | 4-Fold Rise - % (95% CI) <sup>b</sup> | | | |
| Day 29 | n | | | |
| | GMFR (95% CI) <sup>a</sup> | | | |
| | 4-Fold Rise - % (95% CI) <sup>b</sup> | | | |
| Day 91 | n | | | |
| | GMFR (95% CI) <sup>a</sup> | | | |
| | 4-Fold Rise - % (95% CI) <sup>b</sup> | | | |
| Day 181 | n | | | |
| | GMFR (95% CI) <sup>a</sup> | | | |
| | 4-Fold Rise - % (95% CI) <sup>b</sup> | | | |
| Day 366 | n | | | |
| | GMFR (95% CI) <sup>a</sup> | | | |
| | 4-Fold Rise - % (95% CI) <sup>b</sup> | | | |

Notes: N=Number of subjects in the mITT population.

n=Number of subjects with results available at time point.

GMFR=Geometric Mean Fold Rise, NE=Not Estimable.

<sup>a</sup> Confidence interval calculated based on the Student's t-distribution

## Implementation notes:

For tables using the PP population, update footnote to read: "Notes: N=Number of subjects in the Per Protocol population."

- Table 101: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean Fold Rise and 4-Fold Rise Results by Time Point and Treatment Group, D614G Per Protocol Population
- Table 102: Pseudovirus Neutralization Assay ID<sub>80</sub> Geometric Mean Fold Rise and 4-Fold Rise Results by Time Point and Treatment Group,1 D614G mITT Population
- Table 103: Pseudovirus Neutralization Assay ID<sub>80</sub> Geometric Mean Fold Rise and 4-Fold Rise Results by Time Point and Treatment Group, D614G Per Protocol Population
- Table 104: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean Fold Rise and 4-Fold Rise Results by Time Point and Treatment Group, B.1.351 mITT Population
- Table 105: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean Fold Rise and 4-Fold Rise Results by Time Point and Treatment Group, B.1.351 Per Protocol Population
- Table 106: Pseudovirus Neutralization Assay ID<sub>80</sub> Geometric Mean Fold Rise and 4-Fold Rise Results by Time Point and Treatment Group, B.1.351 mITT Population
- Table 107: Pseudovirus Neutralization Assay ID<sub>80</sub> Geometric Mean Fold Rise and 4-Fold Rise Results by Time Point and Treatment Group, B.1.351 Per Protocol Population
- Table 108: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean Fold Rise and 4-Fold Rise Results by Time Point and Treatment Group, B.1.617.2 mITT Population
- Table 109: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean Fold Rise and 4-Fold Rise Results by Time Point and Treatment Group, B.1.617.2 Per Protocol Population
- Table 110: Pseudovirus Neutralization Assay ID<sub>80</sub> Geometric Mean Fold Rise and 4-Fold Rise Results by Time Point and Treatment Group, B.1.617.2 mITT Population
- Table 111: Pseudovirus Neutralization Assay ID<sub>80</sub> Geometric Mean Fold Rise and 4-Fold Rise Results by Time Point and Treatment Group, B.1.617.2 Per Protocol Population
- Table 112: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean Fold Rise and 4-Fold Rise Results by Time Point and Treatment Group, P.1 mITT Population

- Table 113: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean Fold Rise and 4-Fold Rise Results by Time Point and Treatment Group, P.1 Per Protocol Population
- Table 114: Pseudovirus Neutralization Assay ID<sub>80</sub> Geometric Mean Fold Rise and 4-Fold Rise Results by Time Point and Treatment Group, P.1 mITT Population
- Table 115: Pseudovirus Neutralization Assay ID<sub>80</sub> Geometric Mean Fold Rise and 4-Fold Rise Results by Time Point and Treatment Group, P.1 Per Protocol Population
- Table 116: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean Fold Rise and 4-Fold Rise Results by Time Point and Treatment Group, B.1.1.7 mITT Population
- Table 117: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean Fold Rise and 4-Fold Rise Results by Time Point and Treatment Group, B.1.1.7 Per Protocol Population
- Table 118: Pseudovirus Neutralization Assay ID<sub>80</sub> Geometric Mean Fold Rise and 4-Fold Rise Results by Time Point and Treatment Group, B.1.1.7 mITT Population
- Table 119: Pseudovirus Neutralization Assay ID<sub>80</sub> Geometric Mean Fold Rise and 4-Fold Rise Results by Time Point and Treatment Group, B.1.1.7 Per Protocol Population

Table 120: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean Fold Rise and 4-Fold Rise Results by Time Point and Treatment Group, S-2P-Wa-1 – mITT Population

| Planned Time Point | Statistic | 50 μg<br>mRNA-1273.351<br>(N=X) | 25 μg<br>mRNA -1273 +<br>25 μg<br>mRNA -1273.351<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|
| Day 15 | n | | | |
| | GMFR (95% CI) <sup>a</sup> | | | |
| | 4-Fold Rise - % (95% CI) <sup>b</sup> | | | |
| Day 29 | n | | | |
| | GMFR (95% CI) <sup>a</sup> | | | |
| | 4-Fold Rise - % (95% CI) <sup>b</sup> | | | |
| Day 91 | n | | | |
| | GMFR (95% CI) <sup>a</sup> | | | |
| | 4-Fold Rise - % (95% CI) <sup>b</sup> | | | |
| Day 181 | n | | | |
| | GMFR (95% CI) <sup>a</sup> | | | |
| | 4-Fold Rise - % (95% CI) <sup>b</sup> | | | |
| Day 366 | n | | | |
| | GMFR (95% CI) <sup>a</sup> | | | |
| | 4-Fold Rise - % (95% CI) <sup>b</sup> | | | |

Notes: N=Number of subjects in the mITT population.

n=Number of subjects with results available at time point.

GMFR=Geometric Mean Fold Rise, NE=Not Estimable.

<sup>a</sup> Confidence interval calculated based on the Student's t-distribution

## Implementation notes:

For tables using the PP population, update footnote to read: "Notes: N=Number of subjects in the Per Protocol population."

- Table 121: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean Fold Rise and 4-Fold Rise Results by Time Point and Treatment Group, D614G Per Protocol Population
- Table 122: Focus Reduction Neutralization Test ID<sub>80</sub> Geometric Mean Fold Rise and 4-Fold Rise Results by Time Point and Treatment Group, D614G mITT Population
- Table 123: Focus Reduction Neutralization Test ID<sub>80</sub> Geometric Mean Fold Rise and 4-Fold Rise Results by Time Point and Treatment Group, D614G Per Protocol Population
- Table 124: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean Fold Rise and 4-Fold Rise Results by Time Point and Treatment Group, B.1.351 mITT Population
- Table 125: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean Fold Rise and 4-Fold Rise Results by Time Point and Treatment Group, B.1.351 Per Protocol Population
- Table 126: Focus Reduction Neutralization Test ID<sub>80</sub> Geometric Mean Fold Rise and 4-Fold Rise Results by Time Point and Treatment Group, B.1.351 mITT Population
- Table 127: Focus Reduction Neutralization Test ID<sub>80</sub> Geometric Mean Fold Rise and 4-Fold Rise Results by Time Point and Treatment Group, B.1.351 Per Protocol Population
- Table 128: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean Fold Rise and 4-Fold Rise Results by Time Point and Treatment Group, B.1.617.2 mITT Population
- Table 129: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean Fold Rise and 4-Fold Rise Results by Time Point and Treatment Group, B.1.617.2 Per Protocol Population
- Table 130: Focus Reduction Neutralization Test ID<sub>80</sub> Geometric Mean Fold Rise and 4-Fold Rise Results by Time Point and Treatment Group, B.1.617.2 mITT Population
- Table 131: Focus Reduction Neutralization Test ID<sub>80</sub> Geometric Mean Fold Rise and 4-Fold Rise Results by Time Point and Treatment Group, B.1.617.2 Per Protocol Population
- Table 132: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean Fold Rise and 4-Fold Rise Results by Time Point and Treatment Group, P.1 mITT Population

- Table 133: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean Fold Rise and 4-Fold Rise Results by Time Point and Treatment Group, P.1 Per Protocol Population
- Table 134: Focus Reduction Neutralization Test ID<sub>80</sub> Geometric Mean Fold Rise and 4-Fold Rise Results by Time Point and Treatment Group, P.1 mITT Population
- Table 135: Focus Reduction Neutralization Test ID<sub>80</sub> Geometric Mean Fold Rise and 4-Fold Rise Results by Time Point and Treatment Group, P.1 Per Protocol Population
- Table 136: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean Fold Rise and 4-Fold Rise Results by Time Point and Treatment Group, B.1.1.7 mITT Population
- Table 137: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean Fold Rise and 4-Fold Rise Results by Time Point and Treatment Group, B.1.1.7 Per Protocol Population
- Table 138: Focus Reduction Neutralization Test ID<sub>80</sub> Geometric Mean Fold Rise and 4-Fold Rise Results by Time Point and Treatment Group, B.1.1.7 mITT Population
- Table 139: Focus Reduction Neutralization Test ID<sub>80</sub> Geometric Mean Fold Rise and 4-Fold Rise Results by Time Point and Treatment Group, B.1.1.7 Per Protocol Population

Table 140: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean Ratio to D614G Variant with 95% Confidence Intervals by Variant, Time Point, and Treatment Group – mITT Population

| Variant | Planned Time<br>Point | Statistic | 50 μg<br>mRNA-1273.351<br>(N=X) | 25 μg<br>mRNA -1273 +<br>25 μg<br>mRNA -1273.351<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|---|
| B.1.351 | Day 1, Pre-Booster | n | | | |
| | Dose | GMR | | | |
| | | 95% CI | | | |
| | Day 8 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 15 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 29 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | <b>Day 91</b> | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 181 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 366 | n | | | |

| Variant | Planned Time<br>Point | Statistic | 50 μg<br>mRNA-1273.351<br>(N=X) | 25 μg<br>mRNA -1273 +<br>25 μg<br>mRNA -1273.351<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|---|
| | | GMR | | | |
| | | 95% CI | | | |
| B.1.617.2 | Day 1, Pre-Booster | n | | | |
| | Dose | GMR | | | |
| | | 95% CI | | | |
| | Day 15 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 29 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 91 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 181 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 366 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| P.1 | | n | | | |

| Variant | Planned Time<br>Point | Statistic | 50 μg<br>mRNA-1273.351<br>(N=X) | 25 μg<br>mRNA -1273 +<br>25 μg<br>mRNA -1273.351<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|---|
| | Day 1, Pre-Booster | GMR | | | |
| | Dose | 95% CI | | | |
| | Day 15 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 29 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | <b>Day 91</b> | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 181 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | <b>Day 366</b> | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| B.1.1.7 | Day 1, Pre-Booster | n | | | |
| | Dose | GMR | | | |
| | | 95% CI | | | |
| | Day 15 | n | | | |

| Variant | Planned Time<br>Point | Statistic | 50 μg<br>mRNA-1273.351<br>(N=X) | 25 μg<br>mRNA -1273 +<br>25 μg<br>mRNA -1273.351<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|---|
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 29 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 91 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 181 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 366 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |

Notes: N=Number of subjects in the mITT population. n=Number of subjects with results available at time point.

GMR=Geometric Mean Ratio, NE=Not Estimable.

Geometric Mean Ratio was calculated by taking the ratio of the result for each variant divided by the result of the D614G variant for each subject and calculating the geometric

Confidence interval calculated based on the Student's t-distribution

- Table 141: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean Ratio to D614G Variant with 95% Confidence Intervals by Variant, Time Point, and Treatment Group Per Protocol Population
- Table 142: Pseudovirus Neutralization Assay ID<sub>80</sub> Geometric Mean Ratio to D614G Variant with 95% Confidence Intervals by Variant, Time Point, and Treatment Group mITT Population
- Table 143: Pseudovirus Neutralization Assay ID<sub>80</sub> Geometric Mean Ratio to D614G Variant with 95% Confidence Intervals by Variant, Time Point, and Treatment Group Per Protocol Population

Table 144: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean Ratio to D614G Variant with 95% Confidence Intervals by Variant, Time Point, and Treatment Group – mITT Population

| Variant | Planned Time<br>Point | Statistic | 50 μg<br>mRNA-1273.351<br>(N=X) | 25 μg<br>mRNA -1273 +<br>25 μg<br>mRNA -1273.351<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|---|
| B.1.351 | Day 1, Pre-Booster | n | | | |
| | Dose | GMR | | | |
| | | 95% CI | | | |
| | Day 8 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 15 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 29 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 91 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 181 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 366 | n | | | |

| Variant | Planned Time<br>Point | Statistic | 50 μg<br>mRNA-1273.351<br>(N=X) | 25 μg<br>mRNA -1273 +<br>25 μg<br>mRNA -1273.351<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|---|
| | | GMR | | | |
| | | 95% CI | | | |
| B.1.617.2 | Day 1, Pre-Booster | n | | | |
| | Dose | GMR | | | |
| | | 95% CI | | | |
| | Day 15 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 29 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 91 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 181 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 366 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| P.1 | | n | | | |

| Variant | Planned Time<br>Point | Statistic | 50 μg<br>mRNA-1273.351<br>(N=X) | 25 μg<br>mRNA -1273 +<br>25 μg<br>mRNA -1273.351<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|---|
| | Day 1, Pre-Booster | GMR | | | |
| | Dose | 95% CI | | | |
| | Day 15 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 29 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | <b>Day 91</b> | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 181 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | <b>Day 366</b> | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| B.1.1.7 | Day 1, Pre-Booster<br>Dose | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 15 | n | | | |

| Variant | Planned Time<br>Point | Statistic | 50 μg<br>mRNA-1273.351<br>(N=X) | 25 μg<br>mRNA -1273 +<br>25 μg<br>mRNA -1273.351<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|---|
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 29 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 91 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 181 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |
| | Day 366 | n | | | |
| | | GMR | | | |
| | | 95% CI | | | |

Notes: N=Number of subjects in the mITT population. n=Number of subjects with results available at time point.

GMR=Geometric Mean Ratio, NE=Not Estimable.

Geometric Mean Ratio was calculated by taking the ratio of the result for each variant divided by the result of the D614G variant for each subject and calculating the geometric

Confidence interval calculated based on the Student's t-distribution

- Table 145: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean Ratio to D614G Variant with 95% Confidence Intervals by Variant, Time Point, and Treatment Group Per Protocol Population
- Table 146: Focus Reduction Neutralization Test ID<sub>80</sub> Geometric Mean Ratio to D614G Variant with 95% Confidence Intervals by Variant, Time Point, and Treatment Group mITT Population
- Table 147: Focus Reduction Neutralization Test ID<sub>80</sub> Geometric Mean Ratio to D614G Variant with 95% Confidence Intervals by Variant, Time Point, and Treatment Group Per Protocol Population
### 14.3 Safety Data

## 14.3.1 Displays of Adverse Events

**Table 148:** Overall Summary of Adverse Events by Treatment Group - All Subjects

| Subjects <sup>a</sup> with | | mRNA- | μg<br>1273.351<br>=X) | 25<br>mRNA<br>25<br>mRNA -<br>(N= | -1273 +<br>μg | | lbjects<br>=X) |
|---|---|---|---|---|---|---|---|
| Category 1 | Category 2 | n | % | n | % | n | % |
| At least one local solicited adverse event | NA | | | | | | |
| At least one systemic solicited adverse event | NA | | | | | | |
| At least one unsolicited adverse event | NA | | | | | | |
| At least one related unsolicited adverse event | Any Grade | | | | | | |
| | Mild (Grade 1) | | | | | | |
| | Moderate (Grade 2) | | | | | | |
| | Severe (Grade 3) | | | | | | |
| At least one severe (Grade 3) unsolicited adverse event | Any relationship | | | | | | |
| | Related | | | | | | |
| | Unrelated | | | | | | |
| At least one serious adverse event <sup>b</sup> | Any relationship | | | | | | |
| | Related | | | | | | |
| | Unrelated | | | | | | |
| At least one adverse event leading to early termination <sup>c</sup> | NA | | | | | | |

| Subjects <sup>a</sup> with | Subjects <sup>a</sup> with | | | | μg<br>-1273 +<br>μg<br>.1273.351<br>=X) | All Subjects<br>(N=X) | |
|---|---|---|---|---|---|---|---|
| Category 1 | Category 2 | n | % | n | % | n | % |
| Any Vitals Signs Adverse Event | NA | | | | | | |
| At least one medically attended adverse event | NA | | | | | | |
| At least one new onset chronic medical NA condition | | | | | | | |

N = Number of subjects in the Safety Population

<sup>a</sup>Subjects are counted once for each category regardless of the number of events.

<sup>b</sup>A listing of Serious Adverse Events is included in Table 157.

<sup>c</sup>As reported on the Adverse Event eCRF.

Table 149: Serious Adverse Events and Non-Serious Adverse Events Occurring in 5% of Subjects in Any Treatment Group by MedDRA System Organ Class and Preferred Term, and Treatment Group - All Subjects

| Preferred Term | MedDRA System Organ Class | 1 | 50 μg<br>mRNA-127<br>(N=X) | 3.351 | | 25 μg<br>nRNA -127<br>25 μg<br>RNA -1273<br>(N=X) | | All Subjects<br>(N=X) | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | n | % | Events | n | % | Events | n | % | Events |
| Serious Adverse Events | <u> </u> | | | | | | | | | |
| All | All | X | х | X | х | х | х | x | x | x |
| PT1 | SOC1 | X | х | X | х | х | х | х | X | х |
| Etc. | Etc. | | | | | | | | | |
| Other (Non-serious) Adverse Events | | | | | | | | | | |
| All | All | X | x | X | х | x | x | x | x | x |
| PT1 | SOC1 | X | х | X | х | х | х | х | х | х |
| Etc | Etc | | | | | | | | | |

N = number of subjects in the Safety Population (number of subjects at risk).

n= number of subjects reporting event.

Events= total frequency of events reported.

#### 14.3.1.1 Solicited Adverse Events

Table 150: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Maximum Severity, and Treatment Group

| | | mRNA- | μg<br>1273.351<br>=X) | 25 <br>mRNA -<br>25 <br>mRNA -1<br>(N= | -1273 +<br>µg<br> 273.351 | All S | ubjects<br>i=X) |
|---|---|---|---|---|---|---|---|
| Symptom | Severity | n | % | n | % | n | % |
| Any Symptom | None | | | | | | |
| | Mild | | | | | | |
| | Moderate | | | | | | |
| | Severe | | | | | | |
| Any Systemic Symptom | None | | | | | | |
| | Mild | | | | | | |
| | Moderate | | | | | | |
| | Severe | | | | | | |
| Arthralgia | None | | | | | | |
| | Mild | | | | | | |
| | Moderate | | | | | | |
| | Severe | | | | | | |
| Fatigue | None | | | | | | |
| | Mild | | | | | | |
| | Moderate | | | | | | |
| | Severe | | | | | | |
| Fever <sup>a</sup> | None | | | | | | |
| | Mild | | | | | | |

| | | mRNA- | μg<br>1273.351<br>=X) | 25 µ<br>mRNA -<br>25 µ<br>mRNA -1<br>(N=2 | 1273 +<br>1g<br>273.351 | All Subjects<br>(N=X) | |
|---|---|---|---|---|---|---|---|
| Symptom | Severity | n | % | n | % | n | % |
| | Moderate | | | | | | |
| | Severe | | | | | | |
| Feverishness | None | | | | | | |
| | Mild | | | | | | |
| | Moderate | | | | | | |
| | Severe | | | | | | |
| Headache | None | | | | | | |
| | Mild | | | | | | |
| | Moderate | | | | | | |
| | Severe | | | | | | |
| Myalgia | None | | | | | | |
| | Mild | | | | | | |
| | Moderate | | | | | | |
| | Severe | | | | | | |
| Nausea | None | | | | | | |
| | Mild | | | | | | |
| | Moderate | | | | | | |
| | Severe | | | | | | |
| Any Local Symptom | None | | | | | | |
| | Mild | | | | | | |

| | | mRNA- | ) μg<br>.1273.351<br>=X) | 25 µ<br>mRNA -1<br>25 µ<br>mRNA -12<br>(N=2 | 1273 +<br>.g<br>273.351 | All Subjects<br>(N=X) | |
|---|---|---|---|---|---|---|---|
| Symptom | Severity | n | % | n | % | n | % |
| | Moderate | | | | | | |
| | Severe | | | | | | |
| Erythema/Redness | None | | | | | | |
| | Mild | | | | | | |
| | Moderate | | | | | | |
| | Severe | | | | | | |
| Erythema/Redness | None | | | | | | |
| Measurement (mm) | Mild | | | | | | |
| | Moderate | | | | | | |
| | Severe | | | | | | |
| Induration/Swelling | None | | | | | | |
| | Mild | | | | | | |
| | Moderate | | | | | | |
| | Severe | | | | | | |
| Induration/Swelling | None | | | | | | |
| Measurement (mm) | Mild | | | | | | |
| | Moderate | | | | | | |
| | Severe | | | | | | |
| Pain | None | | | | | | |
| | Mild | | | | | | |

| | | 50<br>mRNA-:<br>(N= | | mRNA<br>25<br>mRNA - | μg | All Subjects (N=X) | |
|---|---|---|---|---|---|---|---|
| Symptom | Severity | n | % | n | % | n | % |
| | Moderate | | | | | | |
| | Severe | | | | | | |

Severity is the maximum severity reported over all solicited symptoms post dosing for each subject. N=All subjects receiving vaccination with any solicited event data recorded in the database.

Table 151: Summary of Solicited Events by Days Post Treatment, Symptom, and Treatment Group – 50 μg mRNA-1273.351

| | | | -Dose<br>N=X) | | -Dose<br>=X) | Da<br>(N | ay 1<br>=X) | Da<br>(N: | ny 2<br>=X) | Da<br>(N: | ny 3<br>=X) | Da<br>(N | ay 4<br>=X) | Da<br>(N: | ny 5<br>=X) | Da<br>(N | ıy 6<br>=X) | Da<br>(N | ay 7<br>=X) | Day<br>(N | 8+ 1<br>=X) | A<br>Post- | ny<br>-Dose <sup>2</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Symptom | Severity | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| Any | None | | | | | | | | | | | | | | | | | | | | | | |
| Symptom | Mild | | | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | | | |
| Any | None | | | | | | | | | | | | | | | | | | | | | | |
| Systemic<br>Symptom | Mild | | | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | | | |
| Arthralgia | None | | | | | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | | | |
| Fatigue | None | | | | | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | | | |
| Fever | None | | | | | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | | | |
| Feverishness | None | | | | | | | | | | | | | | | | | | | | | | |

| | | | -Dose<br>N=X) | | -Dose<br>=X) | Da<br>(N | ay 1<br>=X) | | ny 2<br>=X) | Da<br>(N: | ny 3<br>=X) | Da<br>(N | ay 4<br>=X) | Da<br>(N: | ıy 5<br>=X) | Da<br>(N | ıy 6<br>=X) | Da<br>(N | ay 7<br>=X) | Day<br>(N | 8+ 1<br>=X) | A<br>Post- | ny<br>-Dose <sup>2</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Symptom | Severity | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| | Mild | | | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | | | |
| Headache | None | | | | | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | | | |
| Myalgia | None | | | | | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | | | |
| Nausea | None | | | | | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | | | |
| Any Local | None | | | | | | | | | | | | | | | | | | | | | | |
| Symptom | Mild | | | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | | | |
| Erythema/Redness | None | | | | | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | | | |

| | | | Dose =X) | | -Dose<br>=X) | Da<br>(N | ay 1<br>=X) | Da<br>(N: | ny 2<br>=X) | Da<br>(N: | ny 3<br>=X) | Da<br>(N | ay 4<br>=X) | Da<br>(N: | y 5<br>=X) | Da<br>(N | ıy 6<br>=X) | Da<br>(N | ay 7<br>=X) | Day<br>(N: | 8+ 1<br>=X) | A<br>Post- | ny<br>-Dose <sup>2</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Symptom | Severity | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| | Severe | | | | | | | | | | | | | | | | | | | | | | |
| Erythema/Redness | None | | | | | | | | | | | | | | | | | | | | | | |
| Measurement (mm) | Mild | | | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | | | |
| Induration/Swelling | None | | | | | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | | | |
| Induration/Swelling | None | | | | | | | | | | | | | | | | | | | | | | |
| Measurement (mm) | Mild | | | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | | | |
| Pain | None | | | | | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | | | |

Notes: N=Number of subjects in the Safety Population.
Severity is the maximum severity reported post dosing for each subject for each day.

<sup>&</sup>lt;sup>1</sup> Day 8+ includes the maximum severity of each symptom reported on or after Day 8 (includes ongoing symptoms)
<sup>2</sup> Indicates how many subjects had "None", "Mild", "Moderate", or "Severe" as their maximum severity for any day. A subject may be counted in more than one of these categories.

Table with Similar Format:

Implementation note: For any symptoms or days with missing data, add a "Not Reported" row.

Table 152: Summary of Solicited Events by Days Post Treatment, Symptom, and Treatment Group – 25 μg mRNA-1273 + 25 μg mRNA-1273.351

Table 153: Summary of Duration of Solicited Symptoms by Treatment Group - All Subjects

| Variable | Statistic | 50 μg<br>mRNA-1273.351<br>(N=X) | 25 μg<br>mRNA -1273 +<br>25 μg<br>mRNA -1273.351<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|
| Any Symptom | n | | ( | |
| | Mean | | | |
| | Standard Deviation | | | |
| | Median | | | |
| | Minimum | | | |
| | Maximum | | | |
| Any Systemic Symptom | n | | | |
| | Mean | | | |
| | Standard Deviation | | | |
| | Median | | | |
| | Minimum | | | |
| | Maximum | | | |
| Arthralgia | n | | | |
| | Mean | | | |
| | Standard Deviation | | | |
| | Median | | | |
| | Minimum | | | |
| | Maximum | | | |
| Fatigue | n | | | |
| | Mean | | | |

| | Standard Deviation |
|--------------|--------------------|
| | Median |
| | Minimum |
| | Maximum |
| Fever | n |
| | Mean |
| | Standard Deviation |
| | Median |
| | Minimum |
| | Maximum |
| Feverishness | n |
| | Mean |
| | Standard Deviation |
| | Median |
| | Minimum |
| | Maximum |
| Headache | n |
| | Mean |
| | Standard Deviation |
| | Median |
| | Minimum |
| | Maximum |
| Myalgia | n |
| | Mean |
| | Standard Deviation |

| | Median |
|---------------------|--------------------|
| | Minimum |
| | Maximum |
| Nausea | n |
| | Mean |
| | Standard Deviation |
| | Median |
| | Minimum |
| | Maximum |
| Any Local Symptom | n |
| | Mean |
| | Standard Deviation |
| | Median |
| | Minimum |
| | Maximum |
| Erythema/redness | n |
| | Mean |
| | Standard Deviation |
| | Median |
| | Minimum |
| | Maximum |
| Induration/swelling | n |
| | Mean |
| | Standard Deviation |
| | Median |

| | Minimum |
|------------------------------------|-----------------------------------------|
| | Maximum |
| Pain | n e e e e e e e e e e e e e e e e e e e |
| | Mean |
| | Standard Deviation |
| | Median |
| | Minimum |
| | Maximum |
| Notes: N=Number of subjects in the | Safety Population |

Notes: N=Number of subjects in the Safety Population.

n=Number of solicited adverse events.

#### 14.3.1.2 Unsolicited Adverse Events

Table 154: All Adverse Events Cross-Classified by MedDRA System Organ Class, Severity, Relationship to Study Treatment, and Treatment Group

| | | | Rela | ationship to | Vaccination |
|---|---|---|---|---|---|
| Treatment Group | MedDRA System Organ Class | Severity | Not Related (n) | Related (n) | Not Yet Determined (n) |
| 50 μg mRNA-1273.351 | Any SOC | Mild | | | |
| (N=X) | | Moderate | | | |
| | | Severe | | | |
| | [Repeat for all reported SOC] | Mild | | | |
| | | Moderate | | | |
| | | Severe | | | |
| 25 μg mRNA-1273 + 25 μg mRNA-1273.351 | Any SOC | Mild | | | |
| (N=X) | | Moderate | | | |
| | | Severe | | | |
| | [Repeat for all reported SOC] | Mild | | | |
| | | Moderate | | | |
| | | Severe | | | |
| All Subjects | Any SOC | Mild | | | |
| (N=X) | | Moderate | | | |
| | | Severe | | | |
| | [Repeat for all reported SOC] | Mild | | | |
| | | Moderate | | | |
| | | Severe | | | |

| | | | Rela | ationship to | Vaccination |
|---|---|---|---|---|---|
| Treatment Group | MedDRA System Organ Class | Severity | Not Related (n) | Related (n) | Not Yet Determined (n) |
| Notes: N=Number of subjects in the Safety Population. | | | | | |

n=Number of events.

Table 155: Summary of All Unsolicited Adverse Events by MedDRA System Organ Class and Preferred Term, Severity, Relationship, and Treatment Group

| | | | | | Severity | | Relatio | onship to Stud | y Vaccination |
|---|---|---|---|---|---|---|---|---|---|
| Treatment Group | System Organ Class (SOC) | Preferred Term (PT) | Total<br>Events<br>(n) | Mild (n) | Moderate (n) | Severe (n) | Not<br>Related<br>(n) | Related (n) | Not Yet<br>Determined<br>(n) |
| 50 μg mRNA-1273 | Any SOC | Any PT | | | | | | | |
| (N=X) | Gastrointestinal disorders | Any PT | | | | | | | |
| | | Flatulence | | | | | | | |
| | | Vomiting | | | | | | | |
| | [Repeat for all reported | Any PT | | | | | | | |
| | SOC] | [Repeat for all reported PT] | | | | | | | |
| 25 μg mRNA-1273 + | Any SOC | Any PT | | | | | | | |
| 25 μg mRNA-1273.351<br>(N=X) | [Repeat for all reported | Any PT | | | | | | | |
| | SOC] | [Repeat for all reported PT] | | | | | | | |
| All Subjects | Any SOC | Any PT | | | | | | | |
| (N=X) | [Repeat for all reported | Any PT | | | | | | | |
| | SOC] | [Repeat for all reported PT] | | | | | | | |

Notes: N=Number of subjects in the Safety Population.

n=Number of events.

Table 156: Number and Percentage of Subjects Experiencing Unsolicited Adverse Events by MedDRA® System Organ Class and Preferred Term, Severity, Relationship, and Treatment Group

| | | | | | | | Sev | erity | | | Rela | ationsh<br>Vacci | ip to St<br>nation | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | ny<br>lence | M | ild | Mod | erate | Sev | ere | | ot<br>ated | Rel | ated |
| Treatment Group | MedDRA System Organ Class | MedDRA Preferred<br>Term | n | % | n | % | n | % | n | % | n | % | n | % |
| 50 μg mRNA-1273.351 | Any SOC | Any PT | | | | | | | | | | | | |
| (N=X) | [Repeat for all reported SOC] | Any PT | | | | | | | | | | | | |
| | | [Repeat for all reported PT] | | | | | | | | | | | | |
| 25 μg mRNA-1273 + | Any SOC | Any PT | | | | | | | | | | | | |
| 25 μg mRNA-1273.351<br>(N=X) | [Repeat for all reported SOC] | Any PT | | | | | | | | | | | | |
| | | [Repeat for all reported PT] | | | | | | | | | | | | |
| All Subjects | Any SOC | Any PT | | | | | | | | | | | | |
| (N=X) | [Repeat for all reported SOC] | Any PT | | | | | | | | | | | | |
| | | [Repeat for all reported PT] | | | | | | | | | | | | |

Note: N=Number of subjects in the Safety Population.

n=Number of subjects reporting event with the specified SOC.

This table presents number and percentage of subjects. A subject is only counted once per PT and is summarized according to their highest severity and closest relationship.

## 14.3.2 Listing of Deaths, Other Serious and Significant Adverse Events

**Table 157:** Listing of Serious Adverse Events

| Adverse<br>Event | No. of Days Post Associated Dose (Duration) | No. of Days<br>Post Dose<br>the Event<br>Became<br>Serious | Reason<br>Reported<br>as an SAE | Severity | Relationship<br>to Study<br>Treatment | If Not<br>Related,<br>Alternative<br>Etiology | Action<br>Taken with<br>Study<br>Treatment | Subject<br>Discontinued<br>Due to AE | Outcome | MedDRA<br>System<br>Organ<br>Class | MedDRA<br>Preferred<br>Term |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject ID | :, Treatment | Group: , AE N | umber: , 20-00 | 03 Cohort: | | | | | | | |
| Comments: | | | | | | 1 | | | | | |
| Subject ID | :, Treatment ( | Group: , AE N | umber: , 20-00 | 03 Cohort: | | | | | | | |
| Comments: | | <u>'</u> | ı | 1 | | 1 | | | ı | | |

Table 158: Listing of Non-Serious, Unsolicited, Moderate or Severe Adverse Events

| Adverse<br>Event | No. of Days<br>Post<br>Vaccination<br>(Duration) | Severity | Relationship to Vaccination | If Not<br>Related,<br>Alternative<br>Etiology | Action Taken<br>with Study<br>Vaccination | Subject<br>Discontinued<br>Due to AE | Outcome | MedDRA®<br>Sytem Organ<br>Class | MedDRA®<br>Preferred<br>Term | Adverse<br>Event |
|---|---|---|---|---|---|---|---|---|---|---|
| Treatment Grou | ıp: , Dose #: :, Sub | oject ID, AE Num | ber: , 20-0003 Co | hort: | | | | | | |
| | | | Γ | | Γ | | Γ | | | |
| Comments: | | | | | | | | | | |
| Treatment Grou | ip: , Dose #: :, Sub | oject ID, AE Num | ber: , 20-0003 Co | hort: | | | | | | |
| | | | Г | | T | | Г | | | |
| Comments: | | | <u> </u> | | <u> </u> | | <u> </u> | | | <u> </u> |

# Table 159: Listing of MAAEs and NOCMCs

| Subject ID | Treatment<br>Group | Event<br>Description | Date of Product<br>Administration <sup>a</sup> | <br>Date of Onset | MedDRA®<br>Sytem Organ<br>Class | MAAEs | NOCMCs | Relationship <sup>b</sup> | Outcome |
|---|---|---|---|---|---|---|---|---|---|

### 14.3.3 Narratives of Deaths, Other Serious and Significant Adverse Events

(not included in SAP, but this is a placeholder for the CSR)

### 14.3.6 Displays of Vital Signs

Table 160: Vital Signs by Assessment, Maximum Severity, Time Point, and Treatment Group, Any Assessment – All Subjects

| | | 50<br>mRNA-<br>(N | 50 μg<br>mRNA-1273.351 | | All Si<br>(N | ıbjects<br>=X) | |
|---|---|---|---|---|---|---|---|
| Time Point | Severity | n | % | n | % | n | % |
| Baseline | None | | | | | | |
| | Mild | | | | | | |
| | Moderate | | | | | | |
| | Severe | | | | | | |
| Day 15 | None | | | | | | |
| | Mild | | | | | | |
| | Moderate | | | | | | |
| | Severe | | | | | | |
| Day 29 | None | | | | | | |
| | Mild | | | | | | |
| | Moderate | | | | | | |
| | Severe | | | | | | |
| Day 91 | None | | | | | | |
| | Mild | | | | | | |
| | Moderate | | | | | | |
| | Severe | | | | | | |
| Day 181 | None | | | | | | |
| | Mild | | | | | | |

| | | 50 μg<br>mRNA-1273.351<br>(N=X) | | mRNA<br>25<br>mRNA | 5 μg<br>3 -1273 +<br>5 μg<br>-1273.351<br>==X) | All Su<br>(N: | ubjects<br>=X) |
|---|---|---|---|---|---|---|---|
| Time Point | Severity | n | % | n | % | n | % |
| | Moderate | | | | | | |
| | Severe | | | | | | |
| Day 366 | None | | | | | | |
| | Mild | | | | | | |
| | Moderate | | | | | | |
| | Severe | | | | | | |
| Max Severity Post | None | | | | | | |
| Baseline | Mild | | | | | | |
| | Moderate | | | | | | |
| | Severe | | | | | | |

Note: The "Max Post Baseline" rows indicate the maximum severity experienced by each subject at any time point post baseline, including unscheduled assessments. N = Number of subjects in the Safety Population.

#### Tables with Similar Format:

- Table 161: Vital Signs by Assessment, Maximum Severity, Time Point, and Treatment Group, Systolic Blood Pressure All Subjects
- Table 162: Vital Signs by Assessment, Maximum Severity, Time Point, and Treatment Group, Diastolic Blood Pressure All Subjects
- Table 163: Vital Signs by Assessment, Maximum Severity, Time Point, and Treatment Group, Pulse Rate All Subjects
- Table 164: Vital Signs by Assessment, Maximum Severity, Time Point, and Treatment Group, Temperature All Subjects

#### 14.4 Summary of Concomitant Medications

Table 165: Number and Percentage of Subjects with Prior and Concurrent Medications by WHO Drug Classification and Treatment Group – All Subjects

[Implementation Note: Table below contains example medications.]

| | | 50<br>mRNA-1<br>(N= | 273.351 | mRNA<br>25<br>mRNA | i μg<br>-1273 +<br>i μg<br>-1273.351<br>=X) | | Subjects<br>N=X) |
|---|---|---|---|---|---|---|---|
| WHO Drug Code Level 1, Anatomic<br>Group | WHO Drug Code Level 2,<br>Therapeutic Group | n | % | n | % | n | % |
| Any Level 1 Codes | Any Level 2 Codes | | | | | | |
| Alimentary Tract And | Any Level 2 Codes | | | | | | |
| Metabolism | Antidiarrheals,<br>Intestinal<br>Antiinflammatory<br>/Antiinfective Agents | | | | | | |
| | Antiemetics And<br>Antinauseants | | | | | | |
| | Digestives, Incl.<br>Enzymes | | | | | | |
| | Drugs For Acid Related<br>Disorders | | | | | | |
| | Drugs For Constipation | | | | | | |
| | Drugs Used In Diabetes | | | | | | |
| | Mineral Supplements | | | | | | |
| | Other Alimentary<br>Tract And Metabolism<br>Products | | | | | | |
| | Stomatological<br>Preparations | | | | | | |

| | | 50 μg<br>mRNA-1273.351<br>(N=X) | | 25 μg<br>mRNA -1273 +<br>25 μg<br>mRNA -1273.351<br>(N=X) | | All Subjects<br>(N=X) | |
|---|---|---|---|---|---|---|---|
| WHO Drug Code Level 1, Anatomic<br>Group | WHO Drug Code Level 2,<br>Therapeutic Group | n | % | n | % | n | % |
| | Vitamins | | | | | | |
| Antiinfectives For | Any Level 2 Codes | | | | | | |
| Systemic Use | Antibacterials For<br>Systemic Use | | | | | | |
| | Antimycotics For<br>Systemic Use | | | | | | |
| | Antivirals For Systemic<br>Use | | | | | | |
| | Vaccines | | | | | | |
| Antineoplastic And | Any Level 2 Codes | | | | | | |
| Immunomodulating<br>Agents | Antineoplastic Agents | | | | | | |
| | Endocrine Therapy | | | | | | |
| Blood And Blood | Any Level 2 Codes | | | | | | |
| Forming Organs | Antianemic<br>Preparations | | | | | | |
| | Antithrombotic Agents | | | | | | |
| Cardiovascular System | Any Level 2 Codes | | | | | | |
| | Agents Acting On The<br>Renin-Angiotensin<br>System | | | | | | |
| | Beta Blocking Agents | | | | | | |
| | Calcium Channel<br>Blockers | | | | | | |

| | | 50 μg<br>mRNA-1273.351<br>(N=X) | | 25 μg<br>mRNA -1273 +<br>25 μg<br>mRNA -1273.351<br>(N=X) | | | Subjects<br>N=X) |
|---|---|---|---|---|---|---|---|
| WHO Drug Code Level 1, Anatomic<br>Group | WHO Drug Code Level 2,<br>Therapeutic Group | n | % | n | % | n | % |
| | Cardiac Therapy | | | | | | |
| | Diuretics | | | | | | |
| | <b>Lipid Modifying Agents</b> | | | | | | |
| | Vasoprotectives | | | | | | |
| Dermatologicals | Any Level 2 Codes | | | | | | |
| | Anti-Acne Preparations | | | | | | |
| | Antibiotics And<br>Chemotherapeutics For<br>Dermatological Use | | | | | | |
| | Antifungals For<br>Dermatological Use | | | | | | |
| | Antipruritics, Incl.<br>Antihistamines,<br>Anesthetics, Etc. | | | | | | |
| | Antiseptics And<br>Disinfectants | | | | | | |
| | Corticosteroids,<br>Dermatological<br>Preparations | | | | | | |
| | Emollients And<br>Protectives | | | | | | |
| | Other Dermatological<br>Preparations | | | | | | |
| | Preparations For<br>Treatment Of Wounds<br>And Ulcers | | | | | | |

| | | 50 μg<br>mRNA-1273.351<br>(N=X) | | 25 μg<br>mRNA -1273 +<br>25 μg<br>mRNA -1273.351<br>(N=X) | | | Subjects<br>N=X) |
|---|---|---|---|---|---|---|---|
| WHO Drug Code Level 1, Anatomic<br>Group | WHO Drug Code Level 2,<br>Therapeutic Group | n | % | n | % | n | % |
| Genito Urinary System | Any Level 2 Codes | | | | | | |
| And Sex Hormones | Gynecological<br>Antiinfectives And<br>Antiseptics | | | | | | |
| | Other Gynecologicals | | | | | | |
| | Sex Hormones And<br>Modulators Of The<br>Genital System | | | | | | |
| | Urologicals | | | | | | |
| Musculo-Skeletal | Any Level 2 Codes | | | | | | |
| System | Antiinflammatory And<br>Antirheumatic<br>Products | | | | | | |
| | Drugs For Treatment<br>Of Bone Diseases | | | | | | |
| | Muscle Relaxants | | | | | | |
| | Other Drugs For<br>Disorders Of The<br>Musculo-Skeletal<br>System | | | | | | |
| Nervous System | Any Level 2 Codes | | | | | | |
| | Analgesics | | | | | | |
| | Anesthetics | | | | | | |
| | Other Nervous System<br>Drugs | | | | | | |

| | | 50 μg<br>mRNA-1273.351<br>(N=X) | | 25 μg<br>mRNA -1273 +<br>25 μg<br>mRNA -1273.351<br>(N=X) | | All Subjects<br>(N=X) | |
|---|---|---|---|---|---|---|---|
| WHO Drug Code Level 1, Anatomic<br>Group | WHO Drug Code Level 2,<br>Therapeutic Group | n | % | n | % | n | % |
| | Psychoanaleptics | | | | | | |
| | Psycholeptics | | | | | | |
| Respiratory System | Any Level 2 Codes | | | | | | |
| | Antihistamines For<br>Systemic Use | | | | | | |
| | Cough And Cold<br>Preparations | | | | | | |
| | Drugs For Obstructive<br>Airway Diseases | | | | | | |
| | Nasal Preparations | | | | | | |
| Sensory Organs | Any Level 2 Codes | | | | | | |
| | Ophthalmologicals | | | | | | |
| Systemic Hormonal | Any Level 2 Codes | | | | | | |
| Preparations, Excl. Sex<br>Hormones And Insulins | Corticosteroids For<br>Systemic Use | | | | | | |
| | Thyroid Therapy | | | | | | |
| Various | Any Level 2 Codes | | | | | | |
| | General Nutrients | | | | | | |
| | Unspecified Herbal<br>And Traditional Medicine | | | | | | |

Notes: N=Number of subjects in the Safety Population.
n=Number of subjects reporting taking at least one medication in the specific WHO Drug Class.

# **APPENDIX 2. FIGURE MOCK-UPS**

# LIST OF FIGURES

| Figure 1: | CONSORT Flow Diagram | 155 |
|---|---|---|
| Figure 2: | Reverse Cumulative Distribution of Serum IgG ECLIA Arbitrary Units/mL by Time Point and Treatment Group - S-2P-Wa-1, mITT Population | 156 |
| Figure 3: | Reverse Cumulative Distribution of Serum IgG ECLIA Arbitrary Units/mL by Time Point and Treatment Group – S-2P–Wa-1, Per Protocol Population | 157 |
| Figure 4: | Reverse Cumulative Distribution of Serum IgG ECLIA Arbitrary Units/mL by Time Point and Treatment Group – RBD–Wa-1, mITT Population | 157 |
| Figure 5: | Reverse Cumulative Distribution of Serum IgG ECLIA Arbitrary Units/mL by Time Point and Treatment Group – RBD–Wa-1, Per Protocol Population | 157 |
| Figure 6: | Reverse Cumulative Distribution of Serum IgG ECLIAv2 Arbitrary Units/mL by Time Point and Treatment Group – S-2P–Wa-1, mITT Population | 157 |
| Figure 7: | Reverse Cumulative Distribution of Serum IgG ECLIAv2 Arbitrary Units/mL by Time Point and Treatment Group – S-2P–Wa-1, Per Protocol Population | 157 |
| Figure 8: | Reverse Cumulative Distribution of Serum IgG ECLIAv2 Arbitrary Units/mL by Time Point and Treatment Group – S-2P– B.1.351, mITT Population | 157 |
| Figure 9: | Reverse Cumulative Distribution of Serum IgG ECLIAv2 Arbitrary Units/mL by Time Point and Treatment Group – RBD– B.1.351, Per Protocol Population | 157 |
| Figure 10: | Reverse Cumulative Distribution of Serum IgG ECLIAv2 Arbitrary Units/mL by Time Point and Treatment Group – RBD– B.1.351, mITT Population | 157 |
| Figure 11: | Reverse Cumulative Distribution of Serum IgG ECLIAv2 Arbitrary Units/mL by Time Point and Treatment Group – S-2P– B.1.351, Per Protocol Population | 157 |
| Figure 12: | Reverse Cumulative Distribution of Serum IgG ECLIAv2 International Units by Time Point and Treatment Group – S-2P–Wa-1, mITT Population | 157 |
| Figure 13: | Reverse Cumulative Distribution of Serum IgG ECLIAv2 International Units by Time Point and Treatment Group – S-2P–Wa-1, Per Protocol Population | 157 |
| Figure 14: | Reverse Cumulative Distribution of Serum IgG ECLIAv2 Area Under the Curve by Time Point and Treatment Group – S-2P–Wa-1, mITT Population | 157 |

| Figure 15: | Reverse Cumulative Distribution of Serum IgG ECLIAv2 Area Under the Curve by Time Point and Treatment Group – S-2P–Wa-1, Per Protocol Population | 157 |
|---|---|---|
| Figure 16: | Reverse Cumulative Distribution of Serum IgG ECLIAv2 Area Under the Curve by Time Point and Treatment Group – S-2P–B.1.351, mITT Population | 157 |
| Figure 17: | Reverse Cumulative Distribution of Serum IgG ECLIAv2 Area Under the Curve by Time Point and Treatment Group – S-2P–B.1.351, Per Protocol Population | 157 |
| Figure 18: | Reverse Cumulative Distribution of Serum IgG ECLIAv2 Area Under the Curve by Time Point and Treatment Group – S-2P–B.1.617.2, mITT Population | 157 |
| Figure 19: | Reverse Cumulative Distribution of Serum IgG ECLIAv2 Area Under the Curve by Time Point and Treatment Group – S-2P–B.1.617.2, Per Protocol Population | 157 |
| Figure 20: | Reverse Cumulative Distribution of Serum IgG ECLIAv2 Area Under the Curve by Time Point and Treatment Group – S-2P–P.1, mITT Population | 157 |
| Figure 21: | Reverse Cumulative Distribution of Serum IgG ECLIAv2 Area Under the Curve by Time Point and Treatment Group – S-2P–P.1, Per Protocol Population | 158 |
| Figure 22: | Reverse Cumulative Distribution of Serum IgG ECLIAv2 Area Under the Curve by Time Point and Treatment Group – S-2P–B.1.1.7, mITT Population | 158 |
| Figure 23: | Reverse Cumulative Distribution of Serum IgG ECLIAv2 Area Under the Curve by Time Point and Treatment Group – S-2P–B.1.1.7, Per Protocol Population | 158 |
| Figure 24: | Serum IgG ECLIA Arbitrary Units/mL by Time Point and Treatment Group — S-2P–Wa-1, mITT Population | 159 |
| Figure 25: | Serum IgG ECLIA Arbitrary Units/mL by Time Point and Treatment Group - S-2P-Wa-1, Per Protocol Population | 160 |
| Figure 26: | Serum IgG ECLIA Arbitrary Units/mL by Time Point and Treatment Group - RBD-Wa-1, mITT Population | 160 |
| Figure 27: | Serum IgG ECLIA Arbitrary Units/mL by Time Point and Treatment Group - RBD-Wa-1, Per Protocol Population | 160 |
| Figure 28: | Serum IgG ECLIAv2 Arbitrary Units/mL by Time Point and Treatment<br>Group – S-2P–Wa-1, mITT Population | 160 |
| Figure 29: | Serum IgG ECLIAv2 Arbitrary Units/mL by Time Point and Treatment Group – S-2P–Wa-1, Per Protocol Population | 160 |

| Figure 30: | Serum IgG ECLIAv2 Arbitrary Units/mL by Time Point and Treatment<br>Group – S-2P– B.1.351, mITT Population |
|---|---|
| Figure 31: | Serum IgG ECLIAv2 Arbitrary Units/mL by Time Point and Treatment<br>Group – S-2P– B.1.351, Per Protocol Population |
| Figure 32: | Serum IgG ECLIAv2 Arbitrary Units/mL by Time Point and Treatment<br>Group – RBD– B.1.351, mITT Population |
| Figure 33: | Serum IgG ECLIAv2 Arbitrary Units/mL by Time Point and Treatment<br>Group – RBD– B.1.351, Per Protocol Population |
| Figure 34: | Serum IgG ECLIAv2 International Units by Time Point and Treatment Group – S-2P–Wa-1, mITT Population |
| Figure 35: | Serum IgG ECLIAv2 International Units by Time Point and Treatment<br>Group – S-2P–Wa-1, Per Protocol Population |
| Figure 36: | Serum IgG ECLIAv2 Area Under the Curve by Time Point and Treatment Group – S-2P–Wa-1, mITT Population |
| Figure 37: | Serum IgG ECLIAv2 Area Under the Curve by Time Point and Treatment Group – S-2P–Wa-1, Per Protocol Population |
| Figure 38: | Serum IgG ECLIAv2 Area Under the Curve by Time Point and Treatment<br>Group – S-2P– B.1.351, mITT Population |
| Figure 39: | Serum IgG ECLIAv2 Area Under the Curve by Time Point and Treatment<br>Group – S-2P– B.1.351, Per Protocol Population |
| Figure 40: | Serum IgG ECLIAv2 Area Under the Curve by Time Point and Treatment Group – S-2P– B.1.617.2, mITT Population |
| Figure 41: | Serum IgG ECLIAv2 Area Under the Curve by Time Point and Treatment<br>Group – S-2P– B.1.617.2, Per Protocol Population |
| Figure 42: | Serum IgG ECLIAv2 Area Under the Curve by Time Point and Treatment Group – S-2P– P.1, mITT Population |
| Figure 43: | Serum IgG ECLIAv2 Area Under the Curve by Time Point and Treatment Group – S-2P– P.1, Per Protocol Population |
| Figure 44: | Serum IgG ECLIAv2 Area Under the Curve by Time Point and Treatment Group – S-2P– B.1.1.7, mITT Population |
| Figure 45: | Serum IgG ECLIAv2 Area Under the Curve by Time Point and Treatment Group – S-2P– B.1.1.7, Per Protocol Population |
| Figure 46: | Geometric Mean Serum IgG ECLIA Arbitrary Units/mL by Time Point and Treatment Group – S-2P–Wa-1, mITT Population |
| Figure 47: | Geometric Mean Serum IgG ECLIA Arbitrary Units/mL by Time Point and Treatment Group – S-2P–Wa-1, Per Protocol Population |
| Figure 48: | Geometric Mean Serum IgG ECLIA Arbitrary Units/mL by Time Point and Treatment Group – RBD–Wa-1, mITT Population |

| Figure 49: | Geometric Mean Serum IgG ECLIA Arbitrary Units/mL by Time Point and Treatment Group – RBD–Wa-1, Per Protocol Population | 163 |
|---|---|---|
| Figure 50: | Geometric Mean Serum IgG ECLIAv2 Arbitrary Units/mL by Time Point and Treatment Group – S-2P–Wa-1, mITT Population | 163 |
| Figure 51: | Geometric Mean Serum IgG ECLIAv2 Arbitrary Units/mL by Time Point and Treatment Group – S-2P–Wa-1, Per Protocol Population | 163 |
| Figure 52: | Geometric Mean Serum IgG ECLIAv2 Arbitrary Units/mL by Time Point and Treatment Group – S-2P– B.1.351, mITT Population | 163 |
| Figure 53: | Geometric Mean Serum IgG ECLIAv2 Arbitrary Units/mL by Time Point and Treatment Group – S-2P– B.1.351, Per Protocol Population | 163 |
| Figure 54: | Geometric Mean Serum IgG ECLIAv2 Arbitrary Units/mL by Time Point and Treatment Group – RBD– B.1.351, mITT Population | 163 |
| Figure 55: | Geometric Mean Serum IgG ECLIAv2 Arbitrary Units/mL by Time Point and Treatment Group – RBD– B.1.351, Per Protocol Population | 163 |
| Figure 56: | Geometric Mean Serum IgG ECLIAv2 International Units by Time Point and Treatment Group – S-2P–Wa-1, mITT Population | 163 |
| Figure 57: | Geometric Mean Serum IgG ECLIAv2 International Units by Time Point and Treatment Group – S-2P–Wa-1, Per Protocol Population | 163 |
| Figure 58: | Geometric Mean Serum IgG ECLIAv2 Area Under the Curve by Time Point and Treatment Group – S-2P–Wa-1, mITT Population | 163 |
| Figure 59: | Geometric Mean Serum IgG ECLIAv2 Area Under the Curve by Time Point and Treatment Group – S-2P–Wa-1, Per Protocol Population | 163 |
| Figure 60: | Geometric Mean Serum IgG ECLIAv2 Area Under the Curve by Time Point and Treatment Group – S-2P– B.1.351, mITT Population | 163 |
| Figure 61: | Geometric Mean Serum IgG ECLIAv2 Area Under the Curve by Time Point and Treatment Group – S-2P–B.1.351, Per Protocol Population | 163 |
| Figure 62: | Geometric Mean Serum IgG ECLIAv2 Area Under the Curve by Time Point and Treatment Group – S-2P– B.1.617.2, mITT Population | 163 |
| Figure 63: | Geometric Mean Serum IgG ECLIAv2 Area Under the Curve by Time Point and Treatment Group – S-2P– B.1.617.2, Per Protocol Population | 163 |
| Figure 64: | Geometric Mean Serum IgG ECLIAv2 Area Under the Curve by Time Point and Treatment Group – S-2P– P.1, mITT Population | 163 |
| Figure 65: | Geometric Mean Serum IgG ECLIAv2 Area Under the Curve by Time Point and Treatment Group – S-2P– P.1, Per Protocol Population | 164 |
| Figure 66: | Geometric Mean Serum IgG ECLIAv2 Area Under the Curve by Time Point and Treatment Group – S-2P–B.1.1.7, mITT Population | 164 |
| Figure 67: | Geometric Mean Serum IgG ECLIAv2 Area Under the Curve by Time Point and Treatment Group – S-2P–B.1.1.7, Per Protocol Population | 164 |

| Figure 68: | Geometric Mean Pseudovirus Neutralization Assay ID <sub>50</sub> Titers by Time Point and Treatment Group – D614G, mITT Population | .164 |
|---|---|---|
| Figure 69: | Geometric Mean Pseudovirus Neutralization Assay ID <sub>50</sub> Titers by Time Point and Treatment Group – D614G, Per Protocol Population | .164 |
| Figure 70: | Geometric Mean Pseudovirus Neutralization Assay ID <sub>80</sub> Titers by Time Point and Treatment Group – D614G, mITT Population | .164 |
| Figure 71: | Geometric Mean Pseudovirus Neutralization Assay ID <sub>80</sub> Titers by Time Point and Treatment Group – D614G, Per Protocol Population | .164 |
| Figure 72: | Geometric Mean Pseudovirus Neutralization Assay ID <sub>50</sub> Titers by Time Point and Treatment Group – B.1.351, mITT Population | .164 |
| Figure 73: | Geometric Mean Pseudovirus Neutralization Assay ID <sub>50</sub> Titers by Time Point and Treatment Group – B.1.351, Per Protocol Population | .164 |
| Figure 74: | Geometric Mean Pseudovirus Neutralization Assay ID <sub>80</sub> Titers by Time Point and Treatment Group – B.1.351, mITT Population | .164 |
| Figure 75: | Geometric Mean Pseudovirus Neutralization Assay ID <sub>80</sub> Titers by Time Point and Treatment Group – B.1.351, Per Protocol Population | .164 |
| Figure 76: | Geometric Mean Pseudovirus Neutralization Assay ID <sub>50</sub> Titers by Time Point and Treatment Group – B.1.617.2, mITT Population | .164 |
| Figure 77: | Geometric Mean Pseudovirus Neutralization Assay ID <sub>50</sub> Titers by Time Point and Treatment Group – B.1.617.2, Per Protocol Population | .164 |
| Figure 78: | Geometric Mean Pseudovirus Neutralization Assay ID <sub>80</sub> Titers by Time Point and Treatment Group – B.1.617.2, mITT Population | .164 |
| Figure 79: | Geometric Mean Pseudovirus Neutralization Assay ID <sub>80</sub> Titers by Time Point and Treatment Group – B.1.617.2, Per Protocol Population | .164 |
| Figure 80: | Geometric Mean Pseudovirus Neutralization Assay ID <sub>50</sub> Titers by Time Point and Treatment Group – P.1, mITT Population | .164 |
| Figure 81: | Geometric Mean Pseudovirus Neutralization Assay ID <sub>50</sub> Titers by Time Point and Treatment Group – P.1, Per Protocol Population | .164 |
| Figure 82: | Geometric Mean Pseudovirus Neutralization Assay ID <sub>80</sub> Titers by Time Point and Treatment Group – P.1, mITT Population | .164 |
| Figure 83: | Geometric Mean Pseudovirus Neutralization Assay ID <sub>80</sub> Titers by Time Point and Treatment Group – P.1, Per Protocol Population | .164 |
| Figure 84: | Geometric Mean Pseudovirus Neutralization Assay ID <sub>50</sub> Titers by Time Point and Treatment Group – B.1.1.7, mITT Population | .165 |
| Figure 85: | Geometric Mean Pseudovirus Neutralization Assay ID <sub>50</sub> Titers by Time Point and Treatment Group – B.1.1.7, Per Protocol Population | .165 |
| Figure 86: | Geometric Mean Pseudovirus Neutralization Assay ID <sub>80</sub> Titers by Time Point and Treatment Group – B.1.1.7, mITT Population | .165 |
| Figure 87: | Geometric Mean Pseudovirus Neutralization Assay ID <sub>80</sub> Titers by Time Point and Treatment Group – B.1.1.7, Per Protocol Population | 165 |
|---|---|---|
| Figure 88: | Geometric Mean Focus Reduction Neutralization Test ID <sub>50</sub> Titers by Time Point and Treatment Group – D614G, mITT Population | 165 |
| Figure 89: | Geometric Mean Focus Reduction Neutralization Test ID <sub>50</sub> Titers by Time Point and Treatment Group – D614G, Per Protocol Population | 165 |
| Figure 90: | Geometric Mean Focus Reduction Neutralization Test ID <sub>80</sub> Titers by Time Point and Treatment Group – D614G, mITT Population | 165 |
| Figure 91: | Geometric Mean Focus Reduction Neutralization Test ID <sub>80</sub> Titers by Time Point and Treatment Group – D614G, Per Protocol Population | 165 |
| Figure 92: | Geometric Mean Focus Reduction Neutralization Test ID <sub>50</sub> Titers by Time Point and Treatment Group – B.1.351, mITT Population | 165 |
| Figure 93: | Geometric Mean Focus Reduction Neutralization Test ID <sub>50</sub> Titers by Time Point and Treatment Group – B.1.351, Per Protocol Population | 165 |
| Figure 94: | Geometric Mean Focus Reduction Neutralization Test ID <sub>80</sub> Titers by Time Point and Treatment Group – B.1.351, mITT Population | 165 |
| Figure 95: | Geometric Mean Focus Reduction Neutralization Test ID <sub>80</sub> Titers by Time Point and Treatment Group – B.1.351, Per Protocol Population | 165 |
| Figure 96: | Geometric Mean Focus Reduction Neutralization Test ID <sub>50</sub> Titers by Time Point and Treatment Group – B.1.617.2, mITT Population | 165 |
| Figure 97: | Geometric Mean Focus Reduction Neutralization Test ID <sub>50</sub> Titers by Time Point and Treatment Group – B.1.617.2, Per Protocol Population | 165 |
| Figure 98: | Geometric Mean Focus Reduction Neutralization Test ID <sub>80</sub> Titers by Time Point and Treatment Group – B.1.617.2, mITT Population | 165 |
| Figure 99: | Geometric Mean Focus Reduction Neutralization Test ID <sub>80</sub> Titers by Time Point and Treatment Group – B.1.617.2, Per Protocol Population | 165 |
| Figure 100: | : Geometric Mean Focus Reduction Neutralization Test ID <sub>50</sub> Titers by Time<br>Point and Treatment Group – P.1, mITT Population | 165 |
| Figure 101: | : Geometric Mean Focus Reduction Neutralization Test ID <sub>50</sub> Titers by Time<br>Point and Treatment Group – P.1, Per Protocol Population | 165 |
| Figure 102: | : Geometric Mean Focus Reduction Neutralization Test ID <sub>80</sub> Titers by Time<br>Point and Treatment Group – P.1, mITT Population | 165 |
| Figure 103: | : Geometric Mean Focus Reduction Neutralization Test ID <sub>80</sub> Titers by Time<br>Point and Treatment Group – P.1, Per Protocol Population | 166 |
| Figure 104: | : Geometric Mean Focus Reduction Neutralization Test ID <sub>50</sub> Titers by Time<br>Point and Treatment Group – B.1.1.7, mITT Population | 166 |
| Figure 105: | : Geometric Mean Focus Reduction Neutralization Test ID <sub>50</sub> Titers by Time<br>Point and Treatment Group – B.1.1.7, Per Protocol Population | 166 |

| Figure | 6: Geometric Mean Focus Reduction Neutralization Test ID <sub>80</sub> Titers by Time<br>Point and Treatment Group – B.1.1.7, mITT Population | .166 |
|---|---|---|
| Figure | 7: Geometric Mean Focus Reduction Neutralization Test ID <sub>80</sub> Titers by Time<br>Point and Treatment Group – B.1.1.7, Per Protocol Population | .166 |
| Figure | 3: Distribution of Serum IgG ECLIA Arbitrary Units/mL by Time Point and Treatment Group – S-2P–Wa-1, mITT Population | .167 |
| Figure | 2: Distribution of Serum IgG ECLIA Arbitrary Units/mL by Time Point and<br>Treatment Group – S-2P–Wa-1, Per Protocol Population | .168 |
| Figure | Distribution of Serum IgG ECLIA Arbitrary Units/mL by Time Point and Treatment Group – RBD–Wa-1, mITT Population | .168 |
| Figure | : Distribution of Serum IgG ECLIA Arbitrary Units/mL by Time Point and<br>Treatment Group – RBD–Wa-1, Per Protocol Population | .168 |
| Figure | 2: Distribution of Serum IgG ECLIAv2 Arbitrary Units/mL by Time Point and Treatment Group – S-2P–Wa-1, mITT Population | .168 |
| Figure | 3: Distribution of Serum IgG ECLIAv2 Arbitrary Units/mL by Time Point and Treatment Group – S-2P–Wa-1, Per Protocol Population | .168 |
| Figure | : Distribution of Serum IgG ECLIAv2 Arbitrary Units/mL by Time Point and Treatment Group – S-2P–B.1.351, mITT Population | .168 |
| Figure | 5: Distribution of Serum IgG ECLIAv2 Arbitrary Units/mL by Time Point and Treatment Group – S-2P–Wa-1, Per Protocol Population | .168 |
| Figure | b: Distribution of Serum IgG ECLIAv2 Arbitrary Units/mL by Time Point and Treatment Group – RBD– B.1.351, mITT Population | .168 |
| Figure | 7: Distribution of Serum IgG ECLIAv2 Arbitrary Units/mL by Time Point and Treatment Group – RBD– B.1.351, Per Protocol Population | .168 |
| Figure | 8: Distribution of Serum IgG ECLIAv2 International Units by Time Point and Treatment Group – S-2P–Wa-1, mITT Population | .168 |
| Figure | 2: Distribution of Serum IgG ECLIAv2 International Units by Time Point and Treatment Group – S-2P–Wa-1, Per Protocol Population | .168 |
| Figure | 2: Distribution of Serum IgG ECLIAv2 Area Under the Curve by Time Point and Treatment Group – S-2P–Wa-1, mITT Population | .168 |
| Figure | : Distribution of Serum IgG ECLIAv2 Area Under the Curve by Time Point and Treatment Group – S-2P–Wa-1, Per Protocol Population | .168 |
| Figure | 2: Distribution of Serum IgG ECLIAv2 Area Under the Curve by Time Point and Treatment Group – S-2P– B.1.351, mITT Population | .168 |
| Figure | B: Distribution of Serum IgG ECLIAv2 Area Under the Curve by Time Point and Treatment Group – S-2P– B.1.351, Per Protocol Population | |
| Figure | H: Distribution of Serum IgG ECLIAv2 Area Under the Curve by Time Point and Treatment Group – S-2P– B.1.617.2, mITT Population | |

| Figure 125 | : Distribution of Serum IgG ECLIAv2 Area Under the Curve by Time Point and Treatment Group – S-2P– B.1.617.2, Per Protocol Population | 168 |
|---|---|---|
| Figure 126 | b: Distribution of Serum IgG ECLIAv2 Area Under the Curve by Time Point and Treatment Group – S-2P– P.1, mITT Population | 168 |
| Figure 127 | : Distribution of Serum IgG ECLIAv2 Area Under the Curve by Time Point and Treatment Group – S-2P–P.1, Per Protocol Population | 169 |
| Figure 128 | : Distribution of Serum IgG ECLIAv2 Area Under the Curve by Time Point and Treatment Group – S-2P– B.1.1.7, mITT Population | 169 |
| Figure 129 | 2: Distribution of Serum IgG ECLIAv2 Area Under the Curve by Time Point and Treatment Group – S-2P– B.1.1.7, Per Protocol Population | 169 |
| Figure 130 | 2: Distribution of Pseudovirus Neutralization Assay ID <sub>50</sub> Titers by Time Point and Treatment Group – D614G, mITT Population | 169 |
| Figure 131 | : Distribution of Pseudovirus Neutralization Assay ID <sub>50</sub> Titers by Time Point and Treatment Group – D614G, Per Protocol Population | 169 |
| Figure 132 | : Distribution of Pseudovirus Neutralization Assay ID <sub>80</sub> Titers by Time Point and Treatment Group – D614G, mITT Population | 169 |
| Figure 133 | : Distribution of Pseudovirus Neutralization Assay ID <sub>80</sub> Titers by Time Point and Treatment Group – D614G, Per Protocol Population | 169 |
| Figure 134 | : Distribution of Pseudovirus Neutralization Assay ID <sub>50</sub> Titers by Time Point and Treatment Group – B.1.351, mITT Population | 169 |
| Figure 135 | : Distribution of Pseudovirus Neutralization Assay ID <sub>50</sub> Titers by Time Point and Treatment Group – B.1.351, Per Protocol Population | 169 |
| Figure 136 | b: Distribution of Pseudovirus Neutralization Assay ID <sub>80</sub> Titers by Time Point and Treatment Group – B.1.351, mITT Population | 169 |
| Figure 137 | 2: Distribution of Pseudovirus Neutralization Assay ID <sub>80</sub> Titers by Time Point and Treatment Group – B.1.351, Per Protocol Population | 169 |
| Figure 138 | : Distribution of Pseudovirus Neutralization Assay ID <sub>50</sub> Titers by Time Point and Treatment Group – B.1.617.2, mITT Population | 169 |
| Figure 139 | 2: Distribution of Pseudovirus Neutralization Assay ID <sub>50</sub> Titers by Time Point and Treatment Group – B.1.617.2, Per Protocol Population | 169 |
| Figure 140 | 2: Distribution of Pseudovirus Neutralization Assay ID <sub>80</sub> Titers by Time Point and Treatment Group – B.1.617.2, mITT Population | 169 |
| Figure 141 | : Distribution of Pseudovirus Neutralization Assay ID <sub>80</sub> Titers by Time Point and Treatment Group – B.1.617.2, Per Protocol Population | 169 |
| Figure 142 | 2: Distribution of Pseudovirus Neutralization Assay ID <sub>50</sub> Titers by Time Point and Treatment Group – P.1, mITT Population | 169 |
| Figure 143 | : Distribution of Pseudovirus Neutralization Assay ID <sub>50</sub> Titers by Time Point and Treatment Group – P.1, Per Protocol Population | 169 |

| Figure 144: | Distribution of Pseudovirus Neutralization Assay ID <sub>80</sub> Titers by Time Point and Treatment Group – P.1, mITT Population |
|---|---|
| Figure 145: | Distribution of Pseudovirus Neutralization Assay ID <sub>80</sub> Titers by Time Point and Treatment Group – P.1, Per Protocol Population |
| Figure 146: | $\begin{array}{lll} Distribution \ of \ Pseudovirus \ Neutralization \ Assay \ ID_{50} \ Titers \ by \ Time \ Point \\ and \ Treatment \ Group - B.1.1.7, mITT \ Population$ |
| Figure 147: | $\begin{array}{lll} Distribution \ of \ Pseudovirus \ Neutralization \ Assay \ ID_{50} \ Titers \ by \ Time \ Point \\ and \ Treatment \ Group - B.1.1.7, Per \ Protocol \ Population$ |
| Figure 148: | $\begin{array}{c} Distribution \ of \ Pseudovirus \ Neutralization \ Assay \ ID_{80} \ Titers \ by \ Time \ Point \\ and \ Treatment \ Group - B.1.1.7, mITT \ Population$ |
| Figure 149: | $\begin{array}{lll} Distribution \ of \ Pseudovirus \ Neutralization \ Assay \ ID_{80} \ Titers \ by \ Time \ Point \\ and \ Treatment \ Group - B.1.1.7, Per \ Protocol \ Population$ |
| Figure 150: | $\begin{array}{lll} Distribution \ of \ Focus \ Reduction \ Neutralization \ Test \ ID_{50} \ Titers \ by \ Time \\ Point \ and \ Treatment \ Group - D614G, mITT \ Population$ |
| Figure 151: | $\begin{array}{ll} Distribution \ of \ Focus \ Reduction \ Neutralization \ Test \ ID_{50} \ Titers \ by \ Time \\ Point \ and \ Treatment \ Group - D614G, Per \ Protocol \ Population$ |
| Figure 152: | $\begin{array}{lll} Distribution \ of \ Focus \ Reduction \ Neutralization \ Test \ ID_{80} \ Titers \ by \ Time \\ Point \ and \ Treatment \ Group - D614G, mITT \ Population. \end{array}$ |
| Figure 153: | $\begin{array}{lll} Distribution \ of \ Focus \ Reduction \ Neutralization \ Test \ ID_{80} \ Titers \ by \ Time \\ Point \ and \ Treatment \ Group - D614G, Per \ Protocol \ Population$ |
| Figure 154: | $\begin{array}{ll} Distribution \ of \ Focus \ Reduction \ Neutralization \ Test \ ID_{50} \ Titers \ by \ Time \\ Point \ and \ Treatment \ Group - B.1.351, mITT \ Population. \end{array}$ |
| Figure 155: | Distribution of Focus Reduction Neutralization Test ID <sub>50</sub> Titers by Time Point and Treatment Group – B.1.351, Per Protocol Population |
| Figure 156: | Distribution of Focus Reduction Neutralization Test ID <sub>80</sub> Titers by Time Point and Treatment Group – B.1.351, mITT Population |
| Figure 157: | Distribution of Focus Reduction Neutralization Test $ID_{80}$ Titers by Time Point and Treatment Group $-$ B.1.351, Per Protocol Population |
| Figure 158: | Distribution of Focus Reduction Neutralization Test ID <sub>50</sub> Titers by Time Point and Treatment Group – B.1.617.2, mITT Population170 |
| Figure 159: | Distribution of Focus Reduction Neutralization Test ID <sub>50</sub> Titers by Time Point and Treatment Group – B.1.617.2, Per Protocol Population170 |
| Figure 160: | Distribution of Focus Reduction Neutralization Test $ID_{80}$ Titers by Time Point and Treatment Group $-$ B.1.617.2, mITT Population170 |
| Figure 161: | Distribution of Focus Reduction Neutralization Test ID <sub>80</sub> Titers by Time Point and Treatment Group – B.1.617.2, Per Protocol Population170 |
| Figure 162: | Distribution of Focus Reduction Neutralization Test ID <sub>50</sub> Titers by Time Point and Treatment Group – P.1, mITT Population |

| Figure 163: Distribution of Focus Reduction Neutralization Test ID <sub>50</sub> Titers by Time Point and Treatment Group – P.1, Per Protocol Population | 170 |
|---|---|
| Figure 164: Distribution of Focus Reduction Neutralization Test ID <sub>80</sub> Titers by Time Point and Treatment Group – P.1, mITT Population | 170 |
| Figure 165: Distribution of Focus Reduction Neutralization Test ID <sub>80</sub> Titers by Time Point and Treatment Group – P.1, Per Protocol Population | 171 |
| Figure 166: Distribution of Focus Reduction Neutralization Test ID <sub>50</sub> Titers by Time Point and Treatment Group – B.1.1.7, mITT Population | 171 |
| Figure 167: Distribution of Focus Reduction Neutralization Test ID <sub>50</sub> Titers by Time Point and Treatment Group – B.1.1.7, Per Protocol Population | 171 |
| Figure 168: Distribution of Focus Reduction Neutralization Test ID <sub>80</sub> Titers by Time Point and Treatment Group – B.1.1.7, mITT Population | 171 |
| Figure 169: Distribution of Focus Reduction Neutralization Test ID <sub>80</sub> Titers by Time Point and Treatment Group – B.1.1.7, Per Protocol Population | 171 |
| Figure 170: Correlation Heatmap, D614G – mITT Population | 172 |
| Figure 171: Correlation Heatmap, D614G – Per Protocol Population | 173 |
| Figure 172: Correlation Heatmap, B.1.351 – mITT Population | 173 |
| Figure 173: Correlation Heatmap, B.1.351 – Per Protocol Population | 173 |
| Figure 174: Correlation Heatmap, B.1.617.2 – mITT Population | 173 |
| Figure 175: Correlation Heatmap, B.1.617.2 – Per Protocol Population | 173 |
| Figure 176: Correlation Heatmap, P.1 – mITT Population | 173 |
| Figure 177: Correlation Heatmap, P.1 – Per Protocol Population | 173 |
| Figure 178: Correlation Heatmap, B.1.1.7 – mITT Population | 173 |
| Figure 179: Correlation Heatmap, B.1.1.7 – Per Protocol Population | 173 |
| Figure 180: Percentages of CD4 T Cells Expressing IFNγ or IL-2, Beta Mutations | 174 |
| Figure 181: Percentages of CD4 T Cells Expressing IFNγ or IL-2/CM, Beta Mutations | 175 |
| Figure 182: Percentages of CD4 T Cells Expressing IFNγ or IL-2/EM, Beta Mutations | 175 |
| Figure 183: Percentages of CD4 T Cells Expressing IFNγ or IL-2/N, Beta Mutations | 175 |
| Figure 184: Percentages of CD4 T Cells Expressing IFNγ or IL-2/TD, Beta Mutations | 175 |
| Figure 185: Percentages of CD4 T Cells Expressing IFNγ or IL-2 and 154, Beta Mutations | 175 |
| Figure 186: Percentages of CD4 T Cells Expressing IFNy or IL-2 or 154, Beta Mutations | |
| Figure 187: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/C, Beta | |
| Mutations | 175 |

| Figure 188: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/E, Beta Mutations | 175 |
|---|---|
| Figure 189: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/N, Beta Mutations | 175 |
| Figure 190: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/T, Beta Mutations | 175 |
| Figure 191: Percentages of CD4 T Cells Expressing IFNγ, Beta Mutations | 175 |
| Figure 192: Percentages of CD4 T Cells Expressing IL-17, Beta Mutations | 175 |
| Figure 193: Percentages of CD4 T Cells Expressing IL-2, Beta Mutations | 175 |
| Figure 194: Percentages of CD4 T Cells Expressing IL-4 and 154, Beta Mutations | 175 |
| Figure 195: Percentages of CD4 T Cells Expressing IL-4, IL-5, IL-13 and 154, Beta Mutations | 175 |
| Figure 196: Percentages of CD4 T Cells Expressing IL-5 or IL-13 and 154, Beta Mutations | 175 |
| Figure 197: Percentages of CD4 T Cells Expressing TNFα, Beta Mutations | 175 |
| Figure 198: Percentages of CD4 T Cells Expressing IFNγ or IL-2, Beta S | 175 |
| Figure 199: Percentages of CD4 T Cells Expressing IFNγ or IL-2/CM, Beta S | 175 |
| Figure 200: Percentages of CD4 T Cells Expressing IFNγ or IL-2/EM, Beta S | 175 |
| Figure 201: Percentages of CD4 T Cells Expressing IFNγ or IL-2/N, Beta S | 175 |
| Figure 202: Percentages of CD4 T Cells Expressing IFNγ or IL-2/TD, Beta S | 175 |
| Figure 203: Percentages of CD4 T Cells Expressing IFNγ or IL-2 and 154, Beta S | 176 |
| Figure 204: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154, Beta S | 176 |
| Figure 205: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/C, Beta S | 176 |
| Figure 206: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/E, Beta S | 176 |
| Figure 207: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/N, Beta S | 176 |
| Figure 208: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/T, Beta S | 176 |
| Figure 209: Percentages of CD4 T Cells Expressing IFNγ, Beta S | 176 |
| Figure 210: Percentages of CD4 T Cells Expressing IL-17, Beta S | 176 |
| Figure 211: Percentages of CD4 T Cells Expressing IL-2, Beta S | 176 |
| Figure 212: Percentages of CD4 T Cells Expressing IL-4 and 154, Beta S | 176 |
| Figure 213: Percentages of CD4 T Cells Expressing IL-4, IL-5, IL-13 and 154, Beta S | 176 |
| Figure 214: Percentages of CD4 T Cells Expressing IL-5 or IL-13 and 154, Beta S | 176 |
| Figure 215: Percentages of CD4 T Cells Expressing TNFα, Beta S | 176 |

| Figure 216: | : Percentages of CD4 T Cells Expressing IFNγ or IL-2, Conserved S1 | 176 |
|---|---|---|
| Figure 217: | : Percentages of CD4 T Cells Expressing IFNγ or IL-2/CM, Conserved S1 | 176 |
| Figure 218: | : Percentages of CD4 T Cells Expressing IFNγ or IL-2/EM, Conserved S1 | 176 |
| Figure 219: | : Percentages of CD4 T Cells Expressing IFNγ or IL-2/N, Conserved S1 | 176 |
| Figure 220: | : Percentages of CD4 T Cells Expressing IFNγ or IL-2/TD, Conserved S1 | 176 |
| Figure 221: | Percentages of CD4 T Cells Expressing IFNγ or IL-2 and 154, Conserved S1 | 176 |
| Figure 222: | Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154, Conserved S1 | 176 |
| Figure 223: | Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/C, Conserved S1 | 176 |
| Figure 224: | Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/E, Conserved S1 | 176 |
| Figure 225: | Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/N, Conserved S1 | 176 |
| Figure 226: | Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/T, Conserved S1 | 177 |
| Figure 227: | : Percentages of CD4 T Cells Expressing IFNγ, Conserved S1 | 177 |
| Figure 228: | : Percentages of CD4 T Cells Expressing IL-17, Conserved S1 | 177 |
| Figure 229: | : Percentages of CD4 T Cells Expressing IL-2, Conserved S1 | 177 |
| Figure 230: | Percentages of CD4 T Cells Expressing IL-4 and 154, Conserved S1 | 177 |
| Figure 231: | : Percentages of CD4 T Cells Expressing IL-4, IL-5, IL-13 and 154,<br>Conserved S1 | 177 |
| Figure 232: | Percentages of CD4 T Cells Expressing IL-5 or IL-13 and 154, Conserved S1 | 177 |
| Figure 233: | : Percentages of CD4 T Cells Expressing TNFα, Conserved S1 | 177 |
| Figure 234: | : Percentages of CD4 T Cells Expressing IFNγ or IL-2, Conserved S2 | 177 |
| Figure 235: | : Percentages of CD4 T Cells Expressing IFNγ or IL-2/CM, Conserved S2 | 177 |
| Figure 236: | : Percentages of CD4 T Cells Expressing IFNγ or IL-2/EM, Conserved S2 | 177 |
| Figure 237: | : Percentages of CD4 T Cells Expressing IFNγ or IL-2/N, Conserved S2 | 177 |
| Figure 238: | : Percentages of CD4 T Cells Expressing IFNγ or IL-2/TD, Conserved S2 | 177 |
| Figure 239: | Percentages of CD4 T Cells Expressing IFNγ or IL-2 and 154, Conserved S2 | 177 |
| Figure 240: | Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154, Conserved S2 | 177 |
| Figure 241: | Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/C, Conserved S2 | 177 |

| Figure 242 | : Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/E, Conserved S2 | 177 |
|---|---|---|
| Figure 243 | : Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/N, Conserved S2 | 177 |
| Figure 244 | : Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/T, Conserved S2 | 177 |
| Figure 245 | : Percentages of CD4 T Cells Expressing IFNγ, Conserved S2 | 177 |
| Figure 246 | : Percentages of CD4 T Cells Expressing IL-17, Conserved S2 | 177 |
| Figure 247 | : Percentages of CD4 T Cells Expressing IL-2, Conserved S2 | 177 |
| Figure 248 | : Percentages of CD4 T Cells Expressing IL-4 and 154, Conserved S2 | 177 |
| Figure 249 | : Percentages of CD4 T Cells Expressing IL-4, IL-5, IL-13 and 154,<br>Conserved S2 | 178 |
| Figure 250 | : Percentages of CD4 T Cells Expressing IL-5 or IL-13 and 154, Conserved S2 | 178 |
| Figure 251 | : Percentages of CD4 T Cells Expressing TNFα, Conserved S2 | 178 |
| Figure 252 | : Percentages of CD4 T Cells Expressing IFNγ or IL-2, Original Matched | 178 |
| Figure 253 | : Percentages of CD4 T Cells Expressing IFNγ or IL-2/CM, Original Matched | 178 |
| Figure 254 | : Percentages of CD4 T Cells Expressing IFNγ or IL-2/EM, Original Matched | 178 |
| Figure 255 | : Percentages of CD4 T Cells Expressing IFNγ or IL-2/N, Original Matched | 178 |
| Figure 256 | : Percentages of CD4 T Cells Expressing IFNγ or IL-2/TD, Original Matched | 178 |
| Figure 257 | : Percentages of CD4 T Cells Expressing IFNγ or IL-2 and 154, Original Matched | 178 |
| Figure 258 | : Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154, Original Matched | 178 |
| Figure 259 | : Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/C, Original Matched | 178 |
| Figure 260 | : Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/E, Original Matched | 178 |
| Figure 261 | : Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/N, Original Matched | 178 |
| Figure 262 | : Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/T, Original Matched | 178 |
| Figure 263 | : Percentages of CD4 T Cells Expressing IFNγ, Original Matched | 178 |
| Figure 264 | : Percentages of CD4 T Cells Expressing IL-17, Original Matched | 178 |
| Figure 265 | : Percentages of CD4 T Cells Expressing IL-2, Original Matched | 178 |

| Figure 266: Percentages of CD4 T Cells Expressing IL-4 and 154, Original Matched178 |
|---|
| Figure 267: Percentages of CD4 T Cells Expressing IL-4, IL-5, IL-13 and 154, Original Matched |
| Figure 268: Percentages of CD4 T Cells Expressing IL-5 or IL-13 and 154, Original Matched |
| Figure 269: Percentages of CD4 T Cells Expressing TNFα, Original Matched178 |
| Figure 270: Percentages of CD8 T Cells Expressing IFNγ or IL-2, Beta Mutations179 |
| Figure 271: Percentages of CD8 T Cells Expressing IFNγ or IL-2/CM, Beta Mutations180 |
| Figure 272: Percentages of CD8 T Cells Expressing IFNγ or IL-2/EM, Beta Mutations180 |
| Figure 273: Percentages of CD8 T Cells Expressing IFNγ or IL-2/N, Beta Mutations180 |
| Figure 274: Percentages of CD8 T Cells Expressing IFNγ or IL-2/TD, Beta Mutations180 |
| Figure 275: Percentages of CD8 T Cells Expressing IFNγ or IL-2, Beta S |
| Figure 276: Percentages of CD8 T Cells Expressing IFNγ or IL-2/CM, Beta S180 |
| Figure 277: Percentages of CD8 T Cells Expressing IFNγ or IL-2/EM, Beta S180 |
| Figure 278: Percentages of CD8 T Cells Expressing IFNγ or IL-2/N, Beta S180 |
| Figure 279: Percentages of CD8 T Cells Expressing IFNγ or IL-2/TD, Beta S180 |
| Figure 280: Percentages of CD8 T Cells Expressing IFNγ or IL-2, Conserved S1180 |
| Figure 281: Percentages of CD8 T Cells Expressing IFNγ or IL-2/CM, Conserved S1180 |
| Figure 282: Percentages of CD8 T Cells Expressing IFNγ or IL-2/EM, Conserved S1180 |
| Figure 283: Percentages of CD8 T Cells Expressing IFNγ or IL-2/N, Conserved S1180 |
| Figure 284: Percentages of CD8 T Cells Expressing IFNγ or IL-2/TD, Conserved S1180 |
| Figure 285: Percentages of CD8 T Cells Expressing IFNγ or IL-2, Conserved S2180 |
| Figure 286: Percentages of CD8 T Cells Expressing IFNγ or IL-2/CM, Conserved S2180 |
| Figure 287: Percentages of CD8 T Cells Expressing IFNγ or IL-2/EM, Conserved S2180 |
| Figure 288: Percentages of CD8 T Cells Expressing IFNγ or IL-2/N, Conserved S2180 |
| Figure 289: Percentages of CD8 T Cells Expressing IFNγ or IL-2/TD, Conserved S2180 |
| Figure 290: Percentages of CD8 T Cells Expressing IFNγ or IL-2, Original Matched180 |
| Figure 291: Percentages of CD8 T Cells Expressing IFNγ or IL-2/CM, Original Matched180 |
| Figure 292: Percentages of CD8 T Cells Expressing IFNγ or IL-2/EM, Original Matched180 |
| Figure 293: Percentages of CD8 T Cells Expressing IFNγ or IL-2/N, Original Matched181 |
| Figure 294: Percentages of CD8 T Cells Expressing IFN $\gamma$ or IL-2/TD, Original Matched181 |
| Figure 295: Percentages of CD8 T Cells Expressing IFNγ or IL-2, Original S181 |

| Figure 296: | Percentages of CD8 T Cells Expressing IFNγ or IL-2/CM, Original S13 | 81 |
|---|---|---|
| Figure 297: | Percentages of CD8 T Cells Expressing IFNγ or IL-2/EM, Original S13 | 81 |
| Figure 298: | Percentages of CD8 T Cells Expressing IFNγ or IL-2/N, Original S13 | 81 |
| Figure 299: | Percentages of CD8 T Cells Expressing IFNγ or IL-2/TD, Original13 | 81 |
| Figure 300: | Maximum Severity of Solicited Systemic Symptoms by Days Post Vaccination and Treatment Group | 82 |
| Figure 301: | Maximum Severity of Solicited Local Symptoms by Days Post Vaccination and Treatment Group | 83 |
| Figure 302: | Onset of Solicited Systemic Symptoms by Days Post Vaccination and Treatment Group | 84 |
| Figure 303: | Onset of Solicited Local Symptoms by Days Post Vaccination and Treatment Group | 85 |
| | Solicited Symptoms by Days Post Vaccination and Treatment Group— Arthralgia | 86 |
| Figure 305: | Solicited Symptoms by Days Post Vaccination and Treatment Group- Chills1 | 87 |
| | Solicited Symptoms by Days Post Vaccination and Treatment Group— Erythema | 87 |
| | Solicited Symptoms by Days Post Vaccination and Treatment Group— Erythema (mm) | 87 |
| | Solicited Symptoms by Days Post Vaccination and Treatment Group— Fatigue | 87 |
| Figure 309: | Solicited Symptoms by Days Post Vaccination and Treatment Group-Fever1 | 87 |
| | Solicited Symptoms by Days Post Vaccination and Treatment Group—Headache | 87 |
| | Solicited Symptoms by Days Post Vaccination and Treatment Group— Induration | 87 |
| Figure 312: | Solicited Symptoms by Days Post Vaccination and Treatment Group— Induration (mm) | 87 |
| Figure 313: | Solicited Symptoms by Days Post Vaccination and Treatment Group— Myalgia | 87 |
| | Solicited Symptoms by Days Post Vaccination and Treatment Group— Nausea | 87 |
| | Solicited Symptoms by Days Post Vaccination and Treatment Group- Pain | |
| Figure 316: | Frequency of Adverse Events by MedDRA System Organ Class and Severity | 88 |

| Statistical Ar | ıalysis Plan - | DMID F | Protocol: 21 | 1-0002 ( | Cohort 1 |
|---|---|---|---|---|---|

| 1 | ersic | n | 2.0 |
|----|-------|---|-----|
| 23 | May | 2 | 023 |

| Figure 317: Incidence of Adverse Events by MedDRA® System Organ Class and | | |
|---|---|---|
| Maximum Severity | 18 | c |

## 10.1 Disposition of Subjects

## Figure 1: CONSORT Flow Diagram

[Implementation Note: Below is an example CONSORT diagram. The final CONSORT will include the two cohort 1 groups.]



# 14.2.2 Immunogenicity Response Figures by Measure, Treatment/Vaccination, and Time Point

Figure 2: Reverse Cumulative Distribution of Serum IgG ECLIA Arbitrary Units/mL by Time Point and Treatment Group - S-2P-Wa-1, mITT Population

[Implementation Note: Below is an example figure. Lines will only be shown for the two cohort 1 groups.]



- Figure 3: Reverse Cumulative Distribution of Serum IgG ECLIA Arbitrary Units/mL by Time Point and Treatment Group S-2P–Wa-1, Per Protocol Population
- Figure 4: Reverse Cumulative Distribution of Serum IgG ECLIA Arbitrary Units/mL by Time Point and Treatment Group RBD–Wa-1, mITT Population
- Figure 5: Reverse Cumulative Distribution of Serum IgG ECLIA Arbitrary Units/mL by Time Point and Treatment Group RBD–Wa-1, Per Protocol Population
- Figure 6: Reverse Cumulative Distribution of Serum IgG ECLIAv2 Arbitrary Units/mL by Time Point and Treatment Group S-2P–Wa-1, mITT Population
- Figure 7: Reverse Cumulative Distribution of Serum IgG ECLIAv2 Arbitrary Units/mL by Time Point and Treatment Group S-2P–Wa-1, Per Protocol Population
- Figure 8: Reverse Cumulative Distribution of Serum IgG ECLIAv2 Arbitrary Units/mL by Time Point and Treatment Group S-2P–B.1.351, mITT Population
- Figure 9: Reverse Cumulative Distribution of Serum IgG ECLIAv2 Arbitrary Units/mL by Time Point and Treatment Group RBD– B.1.351, Per Protocol Population
- Figure 10: Reverse Cumulative Distribution of Serum IgG ECLIAv2 Arbitrary Units/mL by Time Point and Treatment Group RBD– B.1.351, mITT Population
- Figure 11: Reverse Cumulative Distribution of Serum IgG ECLIAv2 Arbitrary Units/mL by Time Point and Treatment Group S-2P– B.1.351, Per Protocol Population
- Figure 12: Reverse Cumulative Distribution of Serum IgG ECLIAv2 International Units by Time Point and Treatment Group S-2P–Wa-1, mITT Population
- Figure 13: Reverse Cumulative Distribution of Serum IgG ECLIAv2 International Units by Time Point and Treatment Group S-2P–Wa-1, Per Protocol Population
- Figure 14: Reverse Cumulative Distribution of Serum IgG ECLIAv2 Area Under the Curve by Time Point and Treatment Group S-2P–Wa-1, mITT Population
- Figure 15: Reverse Cumulative Distribution of Serum IgG ECLIAv2 Area Under the Curve by Time Point and Treatment Group S-2P–Wa-1, Per Protocol Population
- Figure 16: Reverse Cumulative Distribution of Serum IgG ECLIAv2 Area Under the Curve by Time Point and Treatment Group S-2P–B.1.351, mITT Population
- Figure 17: Reverse Cumulative Distribution of Serum IgG ECLIAv2 Area Under the Curve by Time Point and Treatment Group S-2P–B.1.351, Per Protocol Population
- Figure 18: Reverse Cumulative Distribution of Serum IgG ECLIAv2 Area Under the Curve by Time Point and Treatment Group S-2P–B.1.617.2, mITT Population
- Figure 19: Reverse Cumulative Distribution of Serum IgG ECLIAv2 Area Under the Curve by Time Point and Treatment Group S-2P–B.1.617.2, Per Protocol Population
- Figure 20: Reverse Cumulative Distribution of Serum IgG ECLIAv2 Area Under the Curve by Time Point and Treatment Group S-2P–P.1, mITT Population

- Figure 21: Reverse Cumulative Distribution of Serum IgG ECLIAv2 Area Under the Curve by Time Point and Treatment Group S-2P–P.1, Per Protocol Population
- Figure 22: Reverse Cumulative Distribution of Serum IgG ECLIAv2 Area Under the Curve by Time Point and Treatment Group S-2P–B.1.1.7, mITT Population
- Figure 23: Reverse Cumulative Distribution of Serum IgG ECLIAv2 Area Under the Curve by Time Point and Treatment Group S-2P–B.1.1.7, Per Protocol Population

Figure 24: Serum IgG ECLIA Arbitrary Units/mL by Time Point and Treatment Group – S-2P-Wa-1, mITT Population

[Implementation Note: Below is an example figure. Panels will only be shown for the two cohort 1 groups.]



Implementation note: y-axis label should read "Arbitrary Units/mL (S-2P-Wa-1) (log<sub>10</sub>)" and x-axis should read "Day Post Vaccination."

- Figure 25: Serum IgG ECLIA Arbitrary Units/mL by Time Point and Treatment Group S-2P–Wa-1, Per Protocol Population
- Figure 26: Serum IgG ECLIA Arbitrary Units/mL by Time Point and Treatment Group RBD–Wa-1, mITT Population
- Figure 27: Serum IgG ECLIA Arbitrary Units/mL by Time Point and Treatment Group RBD–Wa-1, Per Protocol Population
- Figure 28: Serum IgG ECLIAv2 Arbitrary Units/mL by Time Point and Treatment Group S-2P–Wa-1, mITT Population
- Figure 29: Serum IgG ECLIAv2 Arbitrary Units/mL by Time Point and Treatment Group S-2P–Wa-1, Per Protocol Population
- Figure 30: Serum IgG ECLIAv2 Arbitrary Units/mL by Time Point and Treatment Group S-2P–B.1.351, mITT Population
- Figure 31: Serum IgG ECLIAv2 Arbitrary Units/mL by Time Point and Treatment Group S-2P–B.1.351, Per Protocol Population
- Figure 32: Serum IgG ECLIAv2 Arbitrary Units/mL by Time Point and Treatment Group RBD–B.1.351, mITT Population
- Figure 33: Serum IgG ECLIAv2 Arbitrary Units/mL by Time Point and Treatment Group RBD–B.1.351, Per Protocol Population
- Figure 34: Serum IgG ECLIAv2 International Units by Time Point and Treatment Group S-2P–Wa-1, mITT Population
- Figure 35: Serum IgG ECLIAv2 International Units by Time Point and Treatment Group S-2P–Wa-1, Per Protocol Population
- Figure 36: Serum IgG ECLIAv2 Area Under the Curve by Time Point and Treatment Group S-2P–Wa-1, mITT Population
- Figure 37: Serum IgG ECLIAv2 Area Under the Curve by Time Point and Treatment Group S-2P–Wa-1, Per Protocol Population
- Figure 38: Serum IgG ECLIAv2 Area Under the Curve by Time Point and Treatment Group S-2P–B.1.351, mITT Population
- Figure 39: Serum IgG ECLIAv2 Area Under the Curve by Time Point and Treatment Group S-2P– B.1.351, Per Protocol Population
- Figure 40: Serum IgG ECLIAv2 Area Under the Curve by Time Point and Treatment Group S-2P–B.1.617.2, mITT Population
- Figure 41: Serum IgG ECLIAv2 Area Under the Curve by Time Point and Treatment Group S-2P–B.1.617.2, Per Protocol Population
- Figure 42: Serum IgG ECLIAv2 Area Under the Curve by Time Point and Treatment Group S-2P–P.1, mITT Population

- Figure 43: Serum IgG ECLIAv2 Area Under the Curve by Time Point and Treatment Group S-2P–P.1, Per Protocol Population
- Figure 44: Serum IgG ECLIAv2 Area Under the Curve by Time Point and Treatment Group S-2P–B.1.1.7, mITT Population
- Figure 45: Serum IgG ECLIAv2 Area Under the Curve by Time Point and Treatment Group S-2P–B.1.1.7, Per Protocol Population

Figure 46: Geometric Mean Serum IgG ECLIA Arbitrary Units/mL by Time Point and Treatment Group – S-2P–Wa-1, mITT Population

[Implementation Note: Below is an example figure. Lines will only be shown for the two cohort 1 groups.]



- Figure 47: Geometric Mean Serum IgG ECLIA Arbitrary Units/mL by Time Point and Treatment Group S-2P-Wa-1, Per Protocol Population
- Figure 48: Geometric Mean Serum IgG ECLIA Arbitrary Units/mL by Time Point and Treatment Group RBD–Wa-1, mITT Population
- Figure 49: Geometric Mean Serum IgG ECLIA Arbitrary Units/mL by Time Point and Treatment Group RBD–Wa-1, Per Protocol Population
- Figure 50: Geometric Mean Serum IgG ECLIAv2 Arbitrary Units/mL by Time Point and Treatment Group S-2P–Wa-1, mITT Population
- Figure 51: Geometric Mean Serum IgG ECLIAv2 Arbitrary Units/mL by Time Point and Treatment Group S-2P-Wa-1, Per Protocol Population
- Figure 52: Geometric Mean Serum IgG ECLIAv2 Arbitrary Units/mL by Time Point and Treatment Group S-2P–B.1.351, mITT Population
- Figure 53: Geometric Mean Serum IgG ECLIAv2 Arbitrary Units/mL by Time Point and Treatment Group S-2P–B.1.351, Per Protocol Population
- Figure 54: Geometric Mean Serum IgG ECLIAv2 Arbitrary Units/mL by Time Point and Treatment Group RBD– B.1.351, mITT Population
- Figure 55: Geometric Mean Serum IgG ECLIAv2 Arbitrary Units/mL by Time Point and Treatment Group RBD– B.1.351, Per Protocol Population
- Figure 56: Geometric Mean Serum IgG ECLIAv2 International Units by Time Point and Treatment Group S-2P–Wa-1, mITT Population
- Figure 57: Geometric Mean Serum IgG ECLIAv2 International Units by Time Point and Treatment Group S-2P–Wa-1, Per Protocol Population
- Figure 58: Geometric Mean Serum IgG ECLIAv2 Area Under the Curve by Time Point and Treatment Group S-2P–Wa-1, mITT Population
- Figure 59: Geometric Mean Serum IgG ECLIAv2 Area Under the Curve by Time Point and Treatment Group S-2P–Wa-1, Per Protocol Population
- Figure 60: Geometric Mean Serum IgG ECLIAv2 Area Under the Curve by Time Point and Treatment Group S-2P– B.1.351, mITT Population
- Figure 61: Geometric Mean Serum IgG ECLIAv2 Area Under the Curve by Time Point and Treatment Group S-2P– B.1.351, Per Protocol Population
- Figure 62: Geometric Mean Serum IgG ECLIAv2 Area Under the Curve by Time Point and Treatment Group S-2P– B.1.617.2, mITT Population
- Figure 63: Geometric Mean Serum IgG ECLIAv2 Area Under the Curve by Time Point and Treatment Group S-2P–B.1.617.2, Per Protocol Population
- Figure 64: Geometric Mean Serum IgG ECLIAv2 Area Under the Curve by Time Point and Treatment Group S-2P– P.1, mITT Population

- Figure 65: Geometric Mean Serum IgG ECLIAv2 Area Under the Curve by Time Point and Treatment Group S-2P– P.1, Per Protocol Population
- Figure 66: Geometric Mean Serum IgG ECLIAv2 Area Under the Curve by Time Point and Treatment Group S-2P–B.1.1.7, mITT Population
- Figure 67: Geometric Mean Serum IgG ECLIAv2 Area Under the Curve by Time Point and Treatment Group S-2P– B.1.1.7, Per Protocol Population
- Figure 68: Geometric Mean Pseudovirus Neutralization Assay ID<sub>50</sub> Titers by Time Point and Treatment Group D614G, mITT Population
- Figure 69: Geometric Mean Pseudovirus Neutralization Assay ID<sub>50</sub> Titers by Time Point and Treatment Group D614G, Per Protocol Population
- Figure 70: Geometric Mean Pseudovirus Neutralization Assay ID<sub>80</sub> Titers by Time Point and Treatment Group D614G, mITT Population
- Figure 71: Geometric Mean Pseudovirus Neutralization Assay ID<sub>80</sub> Titers by Time Point and Treatment Group D614G, Per Protocol Population
- Figure 72: Geometric Mean Pseudovirus Neutralization Assay ID<sub>50</sub> Titers by Time Point and Treatment Group B.1.351, mITT Population
- Figure 73: Geometric Mean Pseudovirus Neutralization Assay ID<sub>50</sub> Titers by Time Point and Treatment Group B.1.351, Per Protocol Population
- Figure 74: Geometric Mean Pseudovirus Neutralization Assay ID<sub>80</sub> Titers by Time Point and Treatment Group B.1.351, mITT Population
- Figure 75: Geometric Mean Pseudovirus Neutralization Assay ID<sub>80</sub> Titers by Time Point and Treatment Group B.1.351, Per Protocol Population
- Figure 76: Geometric Mean Pseudovirus Neutralization Assay ID<sub>50</sub> Titers by Time Point and Treatment Group B.1.617.2, mITT Population
- Figure 77: Geometric Mean Pseudovirus Neutralization Assay ID<sub>50</sub> Titers by Time Point and Treatment Group B.1.617.2, Per Protocol Population
- Figure 78: Geometric Mean Pseudovirus Neutralization Assay ID<sub>80</sub> Titers by Time Point and Treatment Group B.1.617.2, mITT Population
- Figure 79: Geometric Mean Pseudovirus Neutralization Assay ID<sub>80</sub> Titers by Time Point and Treatment Group B.1.617.2, Per Protocol Population
- Figure 80: Geometric Mean Pseudovirus Neutralization Assay ID<sub>50</sub> Titers by Time Point and Treatment Group P.1, mITT Population
- Figure 81: Geometric Mean Pseudovirus Neutralization Assay ID<sub>50</sub> Titers by Time Point and Treatment Group P.1, Per Protocol Population
- Figure 82: Geometric Mean Pseudovirus Neutralization Assay ID<sub>80</sub> Titers by Time Point and Treatment Group P.1, mITT Population
- Figure 83: Geometric Mean Pseudovirus Neutralization Assay ID<sub>80</sub> Titers by Time Point and Treatment Group P.1, Per Protocol Population

- Figure 84: Geometric Mean Pseudovirus Neutralization Assay ID<sub>50</sub> Titers by Time Point and Treatment Group B.1.1.7, mITT Population
- Figure 85: Geometric Mean Pseudovirus Neutralization Assay ID<sub>50</sub> Titers by Time Point and Treatment Group B.1.1.7, Per Protocol Population
- Figure 86: Geometric Mean Pseudovirus Neutralization Assay ID<sub>80</sub> Titers by Time Point and Treatment Group B.1.1.7, mITT Population
- Figure 87: Geometric Mean Pseudovirus Neutralization Assay ID<sub>80</sub> Titers by Time Point and Treatment Group B.1.1.7, Per Protocol Population
- Figure 88: Geometric Mean Focus Reduction Neutralization Test ID<sub>50</sub> Titers by Time Point and Treatment Group D614G, mITT Population
- Figure 89: Geometric Mean Focus Reduction Neutralization Test ID<sub>50</sub> Titers by Time Point and Treatment Group D614G, Per Protocol Population
- Figure 90: Geometric Mean Focus Reduction Neutralization Test ID<sub>80</sub> Titers by Time Point and Treatment Group D614G, mITT Population
- Figure 91: Geometric Mean Focus Reduction Neutralization Test ID<sub>80</sub> Titers by Time Point and Treatment Group D614G, Per Protocol Population
- Figure 92: Geometric Mean Focus Reduction Neutralization Test ID<sub>50</sub> Titers by Time Point and Treatment Group B.1.351, mITT Population
- Figure 93: Geometric Mean Focus Reduction Neutralization Test ID<sub>50</sub> Titers by Time Point and Treatment Group B.1.351, Per Protocol Population
- Figure 94: Geometric Mean Focus Reduction Neutralization Test ID<sub>80</sub> Titers by Time Point and Treatment Group B.1.351, mITT Population
- Figure 95: Geometric Mean Focus Reduction Neutralization Test ID<sub>80</sub> Titers by Time Point and Treatment Group B.1.351, Per Protocol Population
- Figure 96: Geometric Mean Focus Reduction Neutralization Test ID<sub>50</sub> Titers by Time Point and Treatment Group B.1.617.2, mITT Population
- Figure 97: Geometric Mean Focus Reduction Neutralization Test ID<sub>50</sub> Titers by Time Point and Treatment Group B.1.617.2, Per Protocol Population
- Figure 98: Geometric Mean Focus Reduction Neutralization Test ID<sub>80</sub> Titers by Time Point and Treatment Group B.1.617.2, mITT Population
- Figure 99: Geometric Mean Focus Reduction Neutralization Test ID<sub>80</sub> Titers by Time Point and Treatment Group B.1.617.2, Per Protocol Population
- Figure 100: Geometric Mean Focus Reduction Neutralization Test ID<sub>50</sub> Titers by Time Point and Treatment Group P.1, mITT Population
- Figure 101: Geometric Mean Focus Reduction Neutralization Test ID<sub>50</sub> Titers by Time Point and Treatment Group P.1, Per Protocol Population
- Figure 102: Geometric Mean Focus Reduction Neutralization Test ID<sub>80</sub> Titers by Time Point and Treatment Group P.1, mITT Population

- Figure 103: Geometric Mean Focus Reduction Neutralization Test ID<sub>80</sub> Titers by Time Point and Treatment Group P.1, Per Protocol Population
- Figure 104: Geometric Mean Focus Reduction Neutralization Test ID<sub>50</sub> Titers by Time Point and Treatment Group B.1.1.7, mITT Population
- Figure 105: Geometric Mean Focus Reduction Neutralization Test ID<sub>50</sub> Titers by Time Point and Treatment Group B.1.1.7, Per Protocol Population
- Figure 106: Geometric Mean Focus Reduction Neutralization Test ID<sub>80</sub> Titers by Time Point and Treatment Group B.1.1.7, mITT Population
- Figure 107: Geometric Mean Focus Reduction Neutralization Test ID<sub>80</sub> Titers by Time Point and Treatment Group B.1.1.7, Per Protocol Population

Figure 108: Distribution of Serum IgG ECLIA Arbitrary Units/mL by Time Point and Treatment Group – S-2P–Wa-1, mITT Population



- Figure 109: Distribution of Serum IgG ECLIA Arbitrary Units/mL by Time Point and Treatment Group S-2P–Wa-1, Per Protocol Population
- Figure 110: Distribution of Serum IgG ECLIA Arbitrary Units/mL by Time Point and Treatment Group RBD–Wa-1, mITT Population
- Figure 111: Distribution of Serum IgG ECLIA Arbitrary Units/mL by Time Point and Treatment Group RBD–Wa-1, Per Protocol Population
- Figure 112: Distribution of Serum IgG ECLIAv2 Arbitrary Units/mL by Time Point and Treatment Group S-2P–Wa-1, mITT Population
- Figure 113: Distribution of Serum IgG ECLIAv2 Arbitrary Units/mL by Time Point and Treatment Group S-2P–Wa-1, Per Protocol Population
- Figure 114: Distribution of Serum IgG ECLIAv2 Arbitrary Units/mL by Time Point and Treatment Group S-2P–B.1.351, mITT Population
- Figure 115: Distribution of Serum IgG ECLIAv2 Arbitrary Units/mL by Time Point and Treatment Group S-2P-Wa-1, Per Protocol Population
- Figure 116: Distribution of Serum IgG ECLIAv2 Arbitrary Units/mL by Time Point and Treatment Group RBD– B.1.351, mITT Population
- Figure 117: Distribution of Serum IgG ECLIAv2 Arbitrary Units/mL by Time Point and Treatment Group RBD– B.1.351, Per Protocol Population
- Figure 118: Distribution of Serum IgG ECLIAv2 International Units by Time Point and Treatment Group S-2P–Wa-1, mITT Population
- Figure 119: Distribution of Serum IgG ECLIAv2 International Units by Time Point and Treatment Group S-2P–Wa-1, Per Protocol Population
- Figure 120: Distribution of Serum IgG ECLIAv2 Area Under the Curve by Time Point and Treatment Group S-2P–Wa-1, mITT Population
- Figure 121: Distribution of Serum IgG ECLIAv2 Area Under the Curve by Time Point and Treatment Group S-2P–Wa-1, Per Protocol Population
- Figure 122: Distribution of Serum IgG ECLIAv2 Area Under the Curve by Time Point and Treatment Group S-2P– B.1.351, mITT Population
- Figure 123: Distribution of Serum IgG ECLIAv2 Area Under the Curve by Time Point and Treatment Group S-2P– B.1.351, Per Protocol Population
- Figure 124: Distribution of Serum IgG ECLIAv2 Area Under the Curve by Time Point and Treatment Group S-2P– B.1.617.2, mITT Population
- Figure 125: Distribution of Serum IgG ECLIAv2 Area Under the Curve by Time Point and Treatment Group S-2P–B.1.617.2, Per Protocol Population
- Figure 126: Distribution of Serum IgG ECLIAv2 Area Under the Curve by Time Point and Treatment Group S-2P–P.1, mITT Population

- Figure 127: Distribution of Serum IgG ECLIAv2 Area Under the Curve by Time Point and Treatment Group S-2P– P.1, Per Protocol Population
- Figure 128: Distribution of Serum IgG ECLIAv2 Area Under the Curve by Time Point and Treatment Group S-2P–B.1.1.7, mITT Population
- Figure 129: Distribution of Serum IgG ECLIAv2 Area Under the Curve by Time Point and Treatment Group S-2P–B.1.1.7, Per Protocol Population
- Figure 130: Distribution of Pseudovirus Neutralization Assay ID<sub>50</sub> Titers by Time Point and Treatment Group D614G, mITT Population
- Figure 131: Distribution of Pseudovirus Neutralization Assay ID<sub>50</sub> Titers by Time Point and Treatment Group D614G, Per Protocol Population
- Figure 132: Distribution of Pseudovirus Neutralization Assay ID<sub>80</sub> Titers by Time Point and Treatment Group D614G, mITT Population
- Figure 133: Distribution of Pseudovirus Neutralization Assay ID<sub>80</sub> Titers by Time Point and Treatment Group D614G, Per Protocol Population
- Figure 134: Distribution of Pseudovirus Neutralization Assay ID<sub>50</sub> Titers by Time Point and Treatment Group B.1.351, mITT Population
- Figure 135: Distribution of Pseudovirus Neutralization Assay ID<sub>50</sub> Titers by Time Point and Treatment Group B.1.351, Per Protocol Population
- Figure 136: Distribution of Pseudovirus Neutralization Assay ID<sub>80</sub> Titers by Time Point and Treatment Group B.1.351, mITT Population
- Figure 137: Distribution of Pseudovirus Neutralization Assay ID<sub>80</sub> Titers by Time Point and Treatment Group B.1.351, Per Protocol Population
- Figure 138: Distribution of Pseudovirus Neutralization Assay ID<sub>50</sub> Titers by Time Point and Treatment Group B.1.617.2, mITT Population
- Figure 139: Distribution of Pseudovirus Neutralization Assay ID<sub>50</sub> Titers by Time Point and Treatment Group B.1.617.2, Per Protocol Population
- Figure 140: Distribution of Pseudovirus Neutralization Assay ID<sub>80</sub> Titers by Time Point and Treatment Group B.1.617.2, mITT Population
- Figure 141: Distribution of Pseudovirus Neutralization Assay ID<sub>80</sub> Titers by Time Point and Treatment Group B.1.617.2, Per Protocol Population
- Figure 142: Distribution of Pseudovirus Neutralization Assay ID<sub>50</sub> Titers by Time Point and Treatment Group P.1, mITT Population
- Figure 143: Distribution of Pseudovirus Neutralization Assay ID<sub>50</sub> Titers by Time Point and Treatment Group P.1, Per Protocol Population
- Figure 144: Distribution of Pseudovirus Neutralization Assay ID<sub>80</sub> Titers by Time Point and Treatment Group P.1, mITT Population
- Figure 145: Distribution of Pseudovirus Neutralization Assay ID<sub>80</sub> Titers by Time Point and Treatment Group P.1, Per Protocol Population

- Figure 146: Distribution of Pseudovirus Neutralization Assay ID<sub>50</sub> Titers by Time Point and Treatment Group B.1.1.7, mITT Population
- Figure 147: Distribution of Pseudovirus Neutralization Assay ID<sub>50</sub> Titers by Time Point and Treatment Group B.1.1.7, Per Protocol Population
- Figure 148: Distribution of Pseudovirus Neutralization Assay ID<sub>80</sub> Titers by Time Point and Treatment Group B.1.1.7, mITT Population
- Figure 149: Distribution of Pseudovirus Neutralization Assay ID<sub>80</sub> Titers by Time Point and Treatment Group B.1.1.7, Per Protocol Population
- Figure 150: Distribution of Focus Reduction Neutralization Test ID<sub>50</sub> Titers by Time Point and Treatment Group D614G, mITT Population
- Figure 151: Distribution of Focus Reduction Neutralization Test ID<sub>50</sub> Titers by Time Point and Treatment Group D614G, Per Protocol Population
- Figure 152: Distribution of Focus Reduction Neutralization Test ID<sub>80</sub> Titers by Time Point and Treatment Group D614G, mITT Population
- Figure 153: Distribution of Focus Reduction Neutralization Test ID<sub>80</sub> Titers by Time Point and Treatment Group D614G, Per Protocol Population
- Figure 154: Distribution of Focus Reduction Neutralization Test ID<sub>50</sub> Titers by Time Point and Treatment Group B.1.351, mITT Population
- Figure 155: Distribution of Focus Reduction Neutralization Test ID<sub>50</sub> Titers by Time Point and Treatment Group B.1.351, Per Protocol Population
- Figure 156: Distribution of Focus Reduction Neutralization Test ID<sub>80</sub> Titers by Time Point and Treatment Group B.1.351, mITT Population
- Figure 157: Distribution of Focus Reduction Neutralization Test ID<sub>80</sub> Titers by Time Point and Treatment Group B.1.351, Per Protocol Population
- Figure 158: Distribution of Focus Reduction Neutralization Test ID<sub>50</sub> Titers by Time Point and Treatment Group B.1.617.2, mITT Population
- Figure 159: Distribution of Focus Reduction Neutralization Test ID<sub>50</sub> Titers by Time Point and Treatment Group B.1.617.2, Per Protocol Population
- Figure 160: Distribution of Focus Reduction Neutralization Test ID<sub>80</sub> Titers by Time Point and Treatment Group B.1.617.2, mITT Population
- Figure 161: Distribution of Focus Reduction Neutralization Test ID<sub>80</sub> Titers by Time Point and Treatment Group B.1.617.2, Per Protocol Population
- Figure 162: Distribution of Focus Reduction Neutralization Test ID<sub>50</sub> Titers by Time Point and Treatment Group P.1, mITT Population
- Figure 163: Distribution of Focus Reduction Neutralization Test ID<sub>50</sub> Titers by Time Point and Treatment Group P.1, Per Protocol Population
- Figure 164: Distribution of Focus Reduction Neutralization Test ID<sub>80</sub> Titers by Time Point and Treatment Group P.1, mITT Population

- Figure 165: Distribution of Focus Reduction Neutralization Test ID<sub>80</sub> Titers by Time Point and Treatment Group P.1, Per Protocol Population
- Figure 166: Distribution of Focus Reduction Neutralization Test ID<sub>50</sub> Titers by Time Point and Treatment Group B.1.1.7, mITT Population
- Figure 167: Distribution of Focus Reduction Neutralization Test ID<sub>50</sub> Titers by Time Point and Treatment Group B.1.1.7, Per Protocol Population
- Figure 168: Distribution of Focus Reduction Neutralization Test ID<sub>80</sub> Titers by Time Point and Treatment Group B.1.1.7, mITT Population
- Figure 169: Distribution of Focus Reduction Neutralization Test ID<sub>80</sub> Titers by Time Point and Treatment Group B.1.1.7, Per Protocol Population

Figure 170: Correlation Heatmap, D614G – mITT Population

| ELISA AUC<br>RBD | N=707<br>0.962<br>(0.956, 0.967) | N=707<br>0.975<br>(0.971, 0.978) | N=706<br>0.921<br>(0.909, 0.931) | N=245<br>0.930<br>(0.910, 0.945) | N=665<br>0.900<br>(0.884, 0.913) | N=80<br>0.656<br>(0.509, 0.765) |
|---|---|---|---|---|---|---|
| | ELISA AUC<br>S-2P | N=707<br>0.936<br>(0.926, 0.944) | N=706<br>0.968<br>(0.963, 0.972) | N=245<br>0.895<br>(0.867, 0.917) | N=665<br>0.871<br>(0.852, 0.889) | N=80<br>0.584<br>(0.418, 0.713) |
| | | Endpoint Titer<br>RBD | N=706<br>0.903<br>(0.889, 0.916) | N=245<br>0.879<br>(0.847, 0.905) | N=665<br>0.867<br>(0.847, 0.885) | N=80<br>0.568<br>(0.398, 0.701) |
| | | | Endpoint Titer<br>S-2P | N=245<br>0.846<br>(0.806, 0.878) | N=664<br>0.842<br>(0.819, 0.863) | N=80<br>0.529<br>(0.350, 0.671) |
| | | | | FRNT-mNG<br>ID <sub>50</sub> | N=245<br>0.930<br>(0.910, 0.945) | N=80<br>0.781<br>(0.678, 0.854) |
| | | | | | PsVNA (614D)<br>ID <sub>50</sub> | N=80<br>0.611<br>(0.452, 0.733) |
| | | | | | | Live-Virus Neut<br>PRNT <sub>80</sub> |

- Figure 171: Correlation Heatmap, D614G Per Protocol Population
- Figure 172: Correlation Heatmap, B.1.351 mITT Population
- Figure 173: Correlation Heatmap, B.1.351 Per Protocol Population
- Figure 174: Correlation Heatmap, B.1.617.2 mITT Population
- Figure 175: Correlation Heatmap, B.1.617.2 Per Protocol Population
- Figure 176: Correlation Heatmap, P.1 mITT Population
- Figure 177: Correlation Heatmap, P.1 Per Protocol Population
- Figure 178: Correlation Heatmap, B.1.1.7 mITT Population
- Figure 179: Correlation Heatmap, B.1.1.7 Per Protocol Population

Figure 180: Percentages of CD4 T Cells Expressing IFNγ or IL-2, Beta Mutations



Note: Open symbols represent Non-responders and closed symbols represent responders. Plots are annotated with Responder Rate.

Implementation note: Please include all study groups and study time points.

- Figure 181: Percentages of CD4 T Cells Expressing IFNγ or IL-2/CM, Beta Mutations
- Figure 182: Percentages of CD4 T Cells Expressing IFNγ or IL-2/EM, Beta Mutations
- Figure 183: Percentages of CD4 T Cells Expressing IFNy or IL-2/N, Beta Mutations
- Figure 184: Percentages of CD4 T Cells Expressing IFNy or IL-2/TD, Beta Mutations
- Figure 185: Percentages of CD4 T Cells Expressing IFNy or IL-2 and 154, Beta Mutations
- Figure 186: Percentages of CD4 T Cells Expressing IFNy or IL-2 or 154, Beta Mutations
- Figure 187: Percentages of CD4 T Cells Expressing IFNy or IL-2 or 154/C, Beta Mutations
- Figure 188: Percentages of CD4 T Cells Expressing IFNy or IL-2 or 154/E, Beta Mutations
- Figure 189: Percentages of CD4 T Cells Expressing IFNy or IL-2 or 154/N, Beta Mutations
- Figure 190: Percentages of CD4 T Cells Expressing IFNy or IL-2 or 154/T, Beta Mutations
- Figure 191: Percentages of CD4 T Cells Expressing IFNy, Beta Mutations
- Figure 192: Percentages of CD4 T Cells Expressing IL-17, Beta Mutations
- Figure 193: Percentages of CD4 T Cells Expressing IL-2, Beta Mutations
- Figure 194: Percentages of CD4 T Cells Expressing IL-4 and 154, Beta Mutations
- Figure 195: Percentages of CD4 T Cells Expressing IL-4, IL-5, IL-13 and 154, Beta Mutations
- Figure 196: Percentages of CD4 T Cells Expressing IL-5 or IL-13 and 154, Beta Mutations
- Figure 197: Percentages of CD4 T Cells Expressing TNFa, Beta Mutations
- Figure 198: Percentages of CD4 T Cells Expressing IFNγ or IL-2, Beta S
- Figure 199: Percentages of CD4 T Cells Expressing IFNy or IL-2/CM, Beta S
- Figure 200: Percentages of CD4 T Cells Expressing IFNγ or IL-2/EM, Beta S
- Figure 201: Percentages of CD4 T Cells Expressing IFNγ or IL-2/N, Beta S
- Figure 202: Percentages of CD4 T Cells Expressing IFNy or IL-2/TD, Beta S

Figure 224:

Figure 225:

Figure 203: Percentages of CD4 T Cells Expressing IFNy or IL-2 and 154, Beta S **Figure 204:** Percentages of CD4 T Cells Expressing IFNy or IL-2 or 154, Beta S Figure 205: Percentages of CD4 T Cells Expressing IFNy or IL-2 or 154/C, Beta S Figure 206: Percentages of CD4 T Cells Expressing IFNy or IL-2 or 154/E, Beta S Figure 207: Percentages of CD4 T Cells Expressing IFNy or IL-2 or 154/N, Beta S Figure 208: Percentages of CD4 T Cells Expressing IFNy or IL-2 or 154/T, Beta S Figure 209: Percentages of CD4 T Cells Expressing IFNy, Beta S Figure 210: Percentages of CD4 T Cells Expressing IL-17, Beta S Figure 211: Percentages of CD4 T Cells Expressing IL-2, Beta S Figure 212: Percentages of CD4 T Cells Expressing IL-4 and 154, Beta S Figure 213: Percentages of CD4 T Cells Expressing IL-4, IL-5, IL-13 and 154, Beta S Percentages of CD4 T Cells Expressing IL-5 or IL-13 and 154, Beta S Figure 214: **Figure 215:** Percentages of CD4 T Cells Expressing TNFα, Beta S Figure 216: Percentages of CD4 T Cells Expressing IFNy or IL-2, Conserved S1 Figure 217: Percentages of CD4 T Cells Expressing IFNy or IL-2/CM, Conserved S1 Figure 218: Percentages of CD4 T Cells Expressing IFNy or IL-2/EM, Conserved S1 **Figure 219:** Percentages of CD4 T Cells Expressing IFNy or IL-2/N, Conserved S1 Figure 220: Percentages of CD4 T Cells Expressing IFNy or IL-2/TD, Conserved S1 Figure 221: Percentages of CD4 T Cells Expressing IFNy or IL-2 and 154, Conserved S1 Figure 222: Percentages of CD4 T Cells Expressing IFNy or IL-2 or 154, Conserved S1 Percentages of CD4 T Cells Expressing IFNy or IL-2 or 154/C, Conserved S1 Figure 223:

Percentages of CD4 T Cells Expressing IFNy or IL-2 or 154/E, Conserved S1

Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/N, Conserved S1

- Figure 226: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/T, Conserved S1
- Figure 227: Percentages of CD4 T Cells Expressing IFNγ, Conserved S1
- Figure 228: Percentages of CD4 T Cells Expressing IL-17, Conserved S1
- Figure 229: Percentages of CD4 T Cells Expressing IL-2, Conserved S1
- Figure 230: Percentages of CD4 T Cells Expressing IL-4 and 154, Conserved S1
- Figure 231: Percentages of CD4 T Cells Expressing IL-4, IL-5, IL-13 and 154, Conserved S1
- Figure 232: Percentages of CD4 T Cells Expressing IL-5 or IL-13 and 154, Conserved S1
- Figure 233: Percentages of CD4 T Cells Expressing TNFα, Conserved S1
- Figure 234: Percentages of CD4 T Cells Expressing IFNy or IL-2, Conserved S2
- Figure 235: Percentages of CD4 T Cells Expressing IFNy or IL-2/CM, Conserved S2
- Figure 236: Percentages of CD4 T Cells Expressing IFNy or IL-2/EM, Conserved S2
- Figure 237: Percentages of CD4 T Cells Expressing IFNy or IL-2/N, Conserved S2
- Figure 238: Percentages of CD4 T Cells Expressing IFNγ or IL-2/TD, Conserved S2
- Figure 239: Percentages of CD4 T Cells Expressing IFNγ or IL-2 and 154, Conserved S2
- Figure 240: Percentages of CD4 T Cells Expressing IFNy or IL-2 or 154, Conserved S2
- Figure 241: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/C, Conserved S2
- Figure 242: Percentages of CD4 T Cells Expressing IFNy or IL-2 or 154/E, Conserved S2
- Figure 243: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/N, Conserved S2
- Figure 244: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/T, Conserved S2
- Figure 245: Percentages of CD4 T Cells Expressing IFNy, Conserved S2
- Figure 246: Percentages of CD4 T Cells Expressing IL-17, Conserved S2
- Figure 247: Percentages of CD4 T Cells Expressing IL-2, Conserved S2
- Figure 248: Percentages of CD4 T Cells Expressing IL-4 and 154, Conserved S2

- Figure 249: Percentages of CD4 T Cells Expressing IL-4, IL-5, IL-13 and 154, Conserved S2
- Figure 250: Percentages of CD4 T Cells Expressing IL-5 or IL-13 and 154, Conserved S2
- Figure 251: Percentages of CD4 T Cells Expressing TNFα, Conserved S2
- Figure 252: Percentages of CD4 T Cells Expressing IFNy or IL-2, Original Matched
- Figure 253: Percentages of CD4 T Cells Expressing IFNγ or IL-2/CM, Original Matched
- Figure 254: Percentages of CD4 T Cells Expressing IFNy or IL-2/EM, Original Matched
- Figure 255: Percentages of CD4 T Cells Expressing IFNy or IL-2/N, Original Matched
- Figure 256: Percentages of CD4 T Cells Expressing IFNγ or IL-2/TD, Original Matched
- Figure 257: Percentages of CD4 T Cells Expressing IFNy or IL-2 and 154, Original Matched
- Figure 258: Percentages of CD4 T Cells Expressing IFNy or IL-2 or 154, Original Matched
- Figure 259: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/C, Original Matched
- Figure 260: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/E, Original Matched
- Figure 261: Percentages of CD4 T Cells Expressing IFNy or IL-2 or 154/N, Original Matched
- Figure 262: Percentages of CD4 T Cells Expressing IFNγ or IL-2 or 154/T, Original Matched
- Figure 263: Percentages of CD4 T Cells Expressing IFNy, Original Matched
- Figure 264: Percentages of CD4 T Cells Expressing IL-17, Original Matched
- Figure 265: Percentages of CD4 T Cells Expressing IL-2, Original Matched
- Figure 266: Percentages of CD4 T Cells Expressing IL-4 and 154, Original Matched
- Figure 267: Percentages of CD4 T Cells Expressing IL-4, IL-5, IL-13 and 154, Original Matched
- Figure 268: Percentages of CD4 T Cells Expressing IL-5 or IL-13 and 154, Original Matched
- Figure 269: Percentages of CD4 T Cells Expressing TNFα, Original Matched

Figure 270: Percentages of CD8 T Cells Expressing IFNγ or IL-2, Beta Mutations



Note: Open symbols represent Non-responders and closed symbols represent responders. Plots are annotated with Responder Rate.

Implementation note: Do not include a graph for "Responder Rate" and please include all study groups and study time points.
#### Figures with Similar Format:

Figure 292:

Figure 271: Percentages of CD8 T Cells Expressing IFNy or IL-2/CM, Beta Mutations Percentages of CD8 T Cells Expressing IFNy or IL-2/EM, Beta Mutations Figure 272: **Figure 273:** Percentages of CD8 T Cells Expressing IFNy or IL-2/N, Beta Mutations **Figure 274:** Percentages of CD8 T Cells Expressing IFNy or IL-2/TD, Beta Mutations **Figure 275:** Percentages of CD8 T Cells Expressing IFNy or IL-2, Beta S **Figure 276:** Percentages of CD8 T Cells Expressing IFNy or IL-2/CM, Beta S **Figure 277:** Percentages of CD8 T Cells Expressing IFNy or IL-2/EM, Beta S **Figure 278:** Percentages of CD8 T Cells Expressing IFNy or IL-2/N, Beta S Figure 279: Percentages of CD8 T Cells Expressing IFNy or IL-2/TD, Beta S Figure 280: Percentages of CD8 T Cells Expressing IFNy or IL-2, Conserved S1 Percentages of CD8 T Cells Expressing IFNy or IL-2/CM, Conserved S1 Figure 281: Figure 282: Percentages of CD8 T Cells Expressing IFNy or IL-2/EM, Conserved S1 Figure 283: Percentages of CD8 T Cells Expressing IFNy or IL-2/N, Conserved S1 Figure 284: Percentages of CD8 T Cells Expressing IFNy or IL-2/TD, Conserved S1 **Figure 285:** Percentages of CD8 T Cells Expressing IFNy or IL-2, Conserved S2 **Figure 286:** Percentages of CD8 T Cells Expressing IFNy or IL-2/CM, Conserved S2 **Figure 287:** Percentages of CD8 T Cells Expressing IFNy or IL-2/EM, Conserved S2 Figure 288: Percentages of CD8 T Cells Expressing IFNy or IL-2/N, Conserved S2 Figure 289: Percentages of CD8 T Cells Expressing IFNy or IL-2/TD, Conserved S2 Figure 290: Percentages of CD8 T Cells Expressing IFNy or IL-2, Original Matched Percentages of CD8 T Cells Expressing IFNy or IL-2/CM, Original Matched Figure 291:

Percentages of CD8 T Cells Expressing IFNy or IL-2/EM, Original Matched

- Figure 293: Percentages of CD8 T Cells Expressing IFNγ or IL-2/N, Original Matched
- Figure 294: Percentages of CD8 T Cells Expressing IFNy or IL-2/TD, Original Matched
- Figure 295: Percentages of CD8 T Cells Expressing IFNγ or IL-2, Original S
- Figure 296: Percentages of CD8 T Cells Expressing IFNγ or IL-2/CM, Original S
- Figure 297: Percentages of CD8 T Cells Expressing IFNγ or IL-2/EM, Original S
- Figure 298: Percentages of CD8 T Cells Expressing IFNγ or IL-2/N, Original S
- Figure 299: Percentages of CD8 T Cells Expressing IFNγ or IL-2/TD, Original

#### 14.3.1.1 Solicited Adverse Events

Figure 300: Maximum Severity of Solicited Systemic Symptoms by Days Post Vaccination and Treatment Group

[Implementation Note: Panels will only be shown for the two Cohort 1 groups.]



Figure 301: Maximum Severity of Solicited Local Symptoms by Days Post Vaccination and Treatment Group

[Implementation Note: Panels will only be shown for the two Cohort 1 groups.]



Figure 302: Onset of Solicited Systemic Symptoms by Days Post Vaccination and Treatment Group

[Implementation Note: Panels will only be shown for the two Cohort 1 groups.]



Figure with Similar Format:

Figure 303: Onset of Solicited Local Symptoms by Days Post Vaccination and Treatment Group

Figure 304: Solicited Symptoms by Days Post Vaccination and Treatment Group–Arthralgia



Implementation Note: Figure should be a single column with results from the third dose only.

# Figures with Similar Format:

| Figure 305: | Solicited Symptoms by Days Post Vaccination and Treatment Group-Chills |
|---|---|
| Figure 306: | Solicited Symptoms by Days Post Vaccination and Treatment Group- Erythema |
| Figure 307: | Solicited Symptoms by Days Post Vaccination and Treatment Group–Erythema (mm) |
| Figure 308: | Solicited Symptoms by Days Post Vaccination and Treatment Group-Fatigue |
| Figure 309: | Solicited Symptoms by Days Post Vaccination and Treatment Group-Fever |
| Figure 310: | Solicited Symptoms by Days Post Vaccination and Treatment Group-Headache |
| Figure 311: | Solicited Symptoms by Days Post Vaccination and Treatment Group-Induration |
| Figure 312: | Solicited Symptoms by Days Post Vaccination and Treatment Group-Induration (mm) |
| Figure 313: | Solicited Symptoms by Days Post Vaccination and Treatment Group-Myalgia |
| Figure 314: | Solicited Symptoms by Days Post Vaccination and Treatment Group-Nausea |
| Figure 315: | Solicited Symptoms by Days Post Vaccination and Treatment Group-Pain |

#### 14.3.1.2 Unsolicited Adverse Events

Figure 316: Frequency of Adverse Events by MedDRA System Organ Class and Severity



Figure 317: Incidence of Adverse Events by MedDRA® System Organ Class and Maximum Severity



# 14.3.5 Displays of Laboratory Results

Not Applicable.

# APPENDIX 3. LISTINGS MOCK-UPS

# **LISTINGS**

| Listing 1: | 16.1.6: Listing of Subjects Receiving Investigational Product | 192 |
|---|---|---|
| Listing 2: | 16.2.1: Early Terminations or Discontinued Subjects | 193 |
| Listing 3: | 16.2.2.1: Subject-Specific Protocol Deviations | 194 |
| Listing 4: | 16.2.2.2: Non-Subject-Specific Protocol Deviations | 195 |
| Listing 5: | 16.2.3: Subjects Excluded from Analysis Populations | 196 |
| Listing 6: | 16.2.4.1: Demographic Data | 197 |
| Listing 7: | 16.2.4.2: Pre-Existing and Concurrent Medical Conditions | 198 |
| Listing 8: | 16.2.6: Individual Immunogenicity Response Data | 200 |
| Listing 9: | 16.2.6: Individual T-cell Response Data | 200 |
| Listing 10: | 16.2.7.1: Solicited Events – Systemic Symptoms | 201 |
| Listing 11: | 16.2.7.2: Solicited Events – Local Symptoms | 202 |
| Listing 12: | 16.2.7.3: Unsolicited Adverse Events. | 203 |
| Listing 13: | 16.2.9.1: Vital Signs | 205 |
| Listing 14: | 16.2.9.2: Physical Exam Findings | 206 |
| Listing 15: | 16.2.10: Concomitant Medications | 207 |
| Listing 16: | 16.2.11.1: Pregnancy Reports – Maternal Information | 208 |
| Listing 17: | 16.2.11.2: Pregnancy Reports – Gravida and Para | 208 |
| Listing 18: | 16.2.11.3: Pregnancy Reports – Live Birth Outcomes | 209 |
| Listing 19: | 16.2.11.4: Pregnancy Reports – Still Birth Outcomes | 209 |
| Listing 20: | 16.2.11.5: Pregnancy Reports – Spontaneous, Elective, or Therapeutic Abortion Outcomes | 209 |

## Listing 1: 16.1.6: Listing of Subjects Receiving Investigational Product

(not included in SAP, but this is a placeholder for the CSR)

## 16.2 Database Listings by Subject

# **16.2.1 Discontinued Subjects**

# **Listing 2:** 16.2.1: Early Terminations or Discontinued Subjects

| Treatment Group | Subject ID | Category | Reason for Early Termination or Treatment Discontinuation | Study Day |
|---|---|---|---|---|

## **16.2.2 Protocol Deviations**

# **Listing 3:** 16.2.2.1: Subject-Specific Protocol Deviations

| Treatment<br>Group | Subject<br>ID | DV<br>Number | Deviation | Deviation<br>Category | Deviation<br>Severity | Study<br>Day | Reason<br>for<br>Deviation | Deviation<br>Resulted<br>in AE? | Deviation Resulted in Subject Termination? | Deviation<br>Affected<br>Product<br>Stability? | Deviation<br>Resolution | Comments |
|---|---|---|---|---|---|---|---|---|---|---|---|---|

# Listing 4: 16.2.2.2: Non-Subject-Specific Protocol Deviations

| \$<br>Site | Deviation<br>Number | Deviation | Deviation Severity | Reason for<br>Deviation | Deviation<br>Resulted in<br>Subject<br>Termination? | Deviation<br>Affected<br>Product<br>Stability? | Deviation<br>Category | Deviation<br>Resolution | Comments |
|---|---|---|---|---|---|---|---|---|---|

## 16.2.3 Subjects Excluded from the Efficacy Analysis

## **Listing 5:** 16.2.3: Subjects Excluded from Analysis Populations

| Treatment Group | Subject ID | Analyses in which<br>Subject is Included | Analyses from which<br>Subject is Excluded | Results Available? | Reason Subject Excluded |
|---|---|---|---|---|---|
| | | [e.g., Safety, ITT, PP] | [e.g., Safety, ITT, PP, Day x] | | |

Note: "Yes" in the "Results available" column indicates that available data were removed from the analysis. "No" indicates that no data were available for inclusion in the analysis.

## 16.2.4 Demographic Data

**Listing 6:** 16.2.4.1: Demographic Data

| Treatment<br>Group | Subject ID | Sex | Age at Enrollment (years) | Ethnicity | Race | ВМІ | Time Between<br>Dose 2 and Dose 3<br>(Days) |
|---|---|---|---|---|---|---|---|

# Listing 7: 16.2.4.2: Pre-Existing and Concurrent Medical Conditions

| Treatment<br>Group | Subject ID | MH Number | Medical History Term | Condition Start Day | Condition End Day | MedDRA System Organ Class | MedDRA Preferred Term |
|---|---|---|---|---|---|---|---|

# 16.2.5 Compliance and/or Drug Concentration Data (if available)

Not Applicable.

# 16.2.6 Individual Immunogenicity Response Data

16.2.6: Individual Immunogenicity Response Data **Listing 8:** 

| Treatment<br>Group | Subject ID | Planned Time Point | Actual Study Day | Assay | Units | Results |
|---|---|---|---|---|---|---|

#### **Listing 9:** 16.2.6: Individual T-cell Response Data

| Treatment<br>Group | Subject ID | Planned Time Point | Actual Study Day | T-Cell | Peptide Pool | Cytokine | Adjusted Percent | Responder (Y/N) |
|---|---|---|---|---|---|---|---|---|

#### 16.2.7 Adverse Events

**Listing 10:** 16.2.7.1: Solicited Events – Systemic Symptoms

| Treatment<br>Group | Subject ID | Post Dose Day | Assessment <sup>a</sup> | Symptom | Severity | Attributed to<br>Alternate<br>Etiology? <sup>b</sup> | Alternate Etiology |
|---|---|---|---|---|---|---|---|
| | | | MA | | | | |
| | | | Clinic | | | | |

<sup>&</sup>lt;sup>a</sup> MA = Data reported by subject on the Memory Aid and reviewed by clinic staff and reported in Solicited Events eCRF.

Note: Clinic = Data collected by clinic staff during physical exam or symptom assessment (treatment administration record, in-clinic assessment, etc.)

<sup>&</sup>lt;sup>b</sup> Grade 3 events only.

**Listing 11:** 16.2.7.2: Solicited Events – Local Symptoms

| Treatment<br>Group | Subject ID | Post Dose Day | Assessmenta | Symptom | Severity |
|---|---|---|---|---|---|
| | | | MA | | |
| | | | Clinic | | |

<sup>&</sup>lt;sup>a</sup> MA = Data reported by subject on the Memory Aid and reviewed by clinic staff and reported in Solicited Events eCRF.

Note: Clinic = Data collected by clinic staff during physical exam or symptom assessment (treatment administration record, in-clinic assessment, etc.)

# Listing 12: 16.2.7.3: Unsolicited Adverse Events

| Adverse<br>Event | Associated with Dose No. | No. of Days Post Associated Dose (Duration) | Severity | SAE? | Relationship<br>to Study<br>Treatment | In Not<br>Related,<br>Alternative<br>Etiology | Action<br>Taken with<br>Study<br>Treatment | Subject<br>Discontinued<br>Due to AE | Outcome | MedDRA<br>System<br>Organ Class | MedDRA<br>Preferred<br>Term |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Treatment ( | Group: , Subject | ID: , AE Numbe | er: | | <u>'</u> | | | | | | |
| Comments: | | • | • | • | | | | • | | | |
| Treatment ( | Group: , Subject | ID: , AE Numbe | er: | | | | | | | | |
| Comments: | | | | | | | | | | | |
| Note: For ac | dditional details | s about SAEs, se | ee Table: xx. | | | | | | | | |

# **16.2.8 Individual Laboratory Measurements**

Not Applicable.

# 16.2.9 Vital Signs and Physical Exam Findings

Listing 13: 16.2.9.1: Vital Signs

| Treatment<br>Group | Subject ID | Planned Time<br>Point | Actual Study<br>Day | Temperature<br>(°C) | Systolic Blood<br>Pressure<br>(mmHg) | Diastolic Blood<br>Pressure<br>(mmHg) | Heart Rate<br>(beats/min) | Weight<br>(kg) | Height (cm) |
|---|---|---|---|---|---|---|---|---|---|

# Listing 14: 16.2.9.2: Physical Exam Findings

| Treatment<br>Group | Subject ID | Visit<br>Number | Body System | Interpretation | If Abnormal,<br>Findings | If Abnormal,<br>Reported as an AE? |
|---|---|---|---|---|---|---|

## **16.2.10** Concomitant Medications

# **Listing 15:** 16.2.10: Concomitant Medications

| Treatment<br>Group | Subject<br>ID | CM<br>Number | Medication | Medication Start<br>Day | Medication End<br>Day | Indication | Taken for an AE? (AE Description; Number) | Taken for a condition<br>on Medical History?<br>(MH Description;<br>Number) | ATC Level 1<br>(ATC Level 2) |
|---|---|---|---|---|---|---|---|---|---|

## 16.2.11 Pregnancy Reports

**Listing 16:** 16.2.11.1: Pregnancy Reports – Maternal Information

| Treatment<br>Group | Subject<br>ID | Pregnancy<br>Number | Study Day Corresponding to Estimated Date of Conception | Source of<br>Maternal<br>Information | Pregnancy<br>Status | Mother's<br>Pre-<br>Pregnancy<br>BMI | Mother's<br>Weight<br>Gain<br>During<br>Pregnancy | Tobacco, Alcohol, or Drug Use During Pregnancy? | Medications<br>During<br>Pregnancy? | Maternal<br>Complications<br>During<br>Pregnancy? | Maternal<br>Complications<br>During Labor,<br>Delivery, or<br>Post-Partum? |
|---|---|---|---|---|---|---|---|---|---|---|---|

Note: Maternal Complications are included in the Adverse Event listing. Medications taken during pregnancy are included in the Concomitant Medications Listing.

Listing 17: 16.2.11.2: Pregnancy Reports – Gravida and Para

| | | | | Live Births | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject<br>ID | Pregnancy<br>Number | Gravida | Extremely<br>PB <sup>a</sup> | Very<br>Early<br>PB <sup>a</sup> | Early<br>PB <sup>a</sup> | Late<br>PB <sup>a</sup> | Early<br>TB <sup>b</sup> | Full<br>TB <sup>b</sup> | Late<br>TB <sup>b</sup> | Post<br>TB <sup>b</sup> | Still<br>Births | Spontaneous<br>Abortion/<br>Miscarriage | Elective<br>Abortions | Therapeutic<br>Abortions | Major<br>Congenital<br>Anomaly<br>with<br>Previous<br>Pregnancy? |

Note: Gravida includes the current pregnancy, para events do not.

<sup>&</sup>lt;sup>a</sup> Preterm Birth

<sup>&</sup>lt;sup>b</sup> Term Birth

## **Listing 18:** 16.2.11.3: Pregnancy Reports – Live Birth Outcomes

| Subject<br>ID | Pregnancy<br>Number | Fetus<br>Number | Pregnancy<br>Outcome<br>(for this<br>Fetus) | Fetal Distress During Labor and Delivery? | Delivery<br>Method | Gestational<br>Age at Live<br>Birth | Size for<br>Gestational<br>Age | Apgar<br>Score, 1<br>minute | Apgar<br>Score, 5<br>minutes | Cord pH | Congenital<br>Anomalies? | Illnesses/<br>Hospitalizations<br>within 1 Month of<br>Birth? |
|---|---|---|---|---|---|---|---|---|---|---|---|---|

Note: Congenital Anomalies are included in the Adverse Event listing.

## **Listing 19:** 16.2.11.4: Pregnancy Reports – Still Birth Outcomes

| Subject<br>ID | Date of<br>Initial<br>Report | Fetus<br>Number | Pregnancy<br>Outcome<br>(for this<br>Fetus) | Fetal Distress During Labor and Delivery? | Delivery<br>Method | Gestational<br>Age at Still<br>Birth | Size for<br>Gestational<br>Age | Cord pH | Congenital<br>Anomalies? | Autopsy<br>Performed? | If Autopsy, Etiology<br>for Still Birth<br>Identified? |
|---|---|---|---|---|---|---|---|---|---|---|---|

## **Listing 20:** 16.2.11.5: Pregnancy Reports – Spontaneous, Elective, or Therapeutic Abortion Outcomes

| Subject<br>ID | Date of Initial<br>Report | Fetus Number | Pregnancy Outcome<br>(for this Fetus) | Gestational Age at<br>Termination | Abnormality in Product of Conception? | Reason for Therapeutic<br>Abortion |
|---|---|---|---|---|---|---|